

# Statistical Analysis Plan for Interventional Studies Text Only

SAP Text Version Number: 3.0
SAP Text Date: (DD-Mmm-YYYY): 04-Feb-2022

**Sponsor Name: Zogenix International Limited** 

Protocol Number: ZX008-1601

Protocol Title: A Two-Part Study of ZX008 in Children and Adults with Lennox-Gastaut Syndrome (LGS); Part 1: A Randomized, Double-blind, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as Adjunctive Therapy for Seizures in Children and Adults with LGS, Followed by Part 2: An Open-label Extension to Assess Long-Term Safety of ZX008 in Children and Adults with LGS

Protocol Version and Date: (DD-Mmm-YYYY):

13-Jan-2017 Version 1.1

10-Jan-2018 (Amendment 1 Rest of World)

20-Jun-2019 (Amendment 2.0)

29 July 2019 (Amendment 2.1)

02-Jul-2020 (Amendment 3.1)

29-Jul-2020 (Amendment 3.2\_Japan)

Syneos Health Project Code: 1009529A

Authors: Principal Biostatistician

### Notice of Confidential and Proprietary Information:

The information contained in this document is confidential belonging to Zogenix International Limited. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Zogenix International Limited. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, Syneos Health should be notified promptly.

### **Revision History**

| | Version<br># | Date<br>(dd-mmm-<br>yyyy) | Document<br>Owner | Revision Summary |
|---|---|---|---|---|
| | 0.1 | 08-Feb-2019 | | Initial Release Version (unsigned) |
| | 0.2 | 24-May-2019 | | Proposed Updates: Separating Part 1 SAP from Part 2 SAP. Requested revisions from Draft 1. |
| , | 0.3 | 20-Jun-2019 | | Proposed Updates: Separation of Part 1 analyses into Cohort A and Cohort B. |
| • | 0.4 | 08-Jul-2019 | | Proposed Updates: 4th Draft. |
| | 0.5 | 29-Jul-2019 | | Proposed Updates prior to Finalization<br>Version 1.0 |
| | 1.0 | 05-Aug-2019 | | Finalization Version 1.0 |
| | 1.1 | 20-Dec-2019 | | Proposed Updates: Updates to the<br>Additional Secondary Objectives<br>specified for Part 1, Cohort A in the<br>protocol, and to the associated<br>Additional Secondary Efficacy<br>Endpoints |
| | 2.0 | 06-Jan-2020 | | Proposed Updates and Finalization of SAP shells |
| • | 2.0 | 08-Jan-2020 | | Signoff |
| This of | ochines | Phication | | |
| | | | This document is | confidential. |

| Version<br># | Date<br>(dd-mmm-<br>yyyy) | Document<br>Owner | Revision Summary |
|---|---|---|---|
| 2.1 | 10-Dec-2021 | | Proposed Updates: Incorporating changes from Part 1 Note to File dated 31-Jun-2021 that described changes in the SAP after Version 2.0. |
| | | | Incorporated changes to indicate the Part 1 analysis of Cohort B will now occur after all subjects have completed Part 1 instead of after all have completed Part 2. |
| | | | Incorporated changes for analysis of Cohort B results after dry run. |
| | | | Made corrections and added clarifying text in several places throughout the document. |
| 3.0 | 28-Jan-2022 | | Proposed Updates: Removal of selected per protocol outputs for Cohort B Editorial changes to text and shell document. |
| | | | Preparation for Signoff |
| 3.0 | 04-Feb-2022 | - | Final Edits |
| | X | | Signoff |
| ocumes | on 3.0 04-Feb-2022 | | |

I confirm that I have reviewed this document and agree with the content.



### **TABLE OF CONTENTS**

| 1. | GLOSSARY OF ABBREVIATIONS | 9 |
|-----------|------------------------------------|-----|
| | | 100 |
| 2. | PURPOSE | 12 |
| 2.1. | Responsibilities | 12 |
| 2.2. | Timing of Analyses | 12 |
| 2.3. | Unblinding Plan | 13 |
| 3. | PART 1 OBJECTIVES | 13 |
| 3.1. | | 13 |
| 3.2. | Key Secondary Objective | 13 |
| 3.3. | Additional Secondary Objectives | 14 |
| 3.4. | Safety Objectives | 15 |
| 3.5. | Pharmacokinetic Objectives | 15 |
| 3.6. | | 15 |
| 4. | BRIEF DESCRIPTION | 16 |
| 4. | | 10 |
| 4.1. | Subject Selection | 17 |
| 4.2. | Determination of Sample Size | 17 |
| 4.3. | Treatment Assignment & Blinding | 18 |
| 4.4. | Administration of Study Medication | 18 |
| <b>50</b> | | 00 |
| 30 | ENDPOINTS | 26 |
| 5.1. | Primary Efficacy Endpoint | 26 |
| 5.2. | Key Secondary Efficacy Endpoints | 26 |

| 5.3. | Additional Secondary Efficacy Endpoints | . 27 |
|---|---|---|
| 5.4. | Safety Endpoints | . <b>2</b> 8 |
| 5.5. | Exploratory Endpoints | <b>28</b> |
| 6. | ANALYSIS SETS | 28 |
| 6.1. | Enrolled Population | . 29 |
| 6.2. | Safety (SAF) Population | . 29 |
| 6.3. | Modified Intent-to-Treat (mITT) Population | 29 |
| 6.4. | Per Protocol (PP) Population | . 29 |
| 6.5. | Protocol Deviations | . 29 |
| <b>6.6.</b> 6.6 6.6 | .2. Definitions | 30<br>30 |
| 6.7. | Visit Windows | . 32 |
| 6.8. | Pooling of Centers | . 34 |
| 6.9. | Subgroups | . 34 |
| | DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION | . 34 |
| 7.1. | Subject Disposition and Withdrawals | . 34 |
| 7.2. | Demographic and Other Baseline Characteristics | . 35 |
| 7.3. | Medical History, Neurologic History, and Concomitant Diseases | . 36 |
| <b>7.4.</b> 7.4 | Medication | |
| 80 | EFFICACY | . 38 |
| 8.1. | Multiplicity Strategy and Testing Hierarchy | . 38 |
| <b>8.2.</b> 8.2 | Primary Efficacy Endpoint and Analysis | |

| Sensit | ivity Analysis of Cluster Imputation | |
|---|---|---|
| 8.2.2 | 2. Part 1 Primary Efficacy Endpoint Analyses | 42 |
| 8.2.3 | 3. Sensitivity Analyses of Part 1 Primary Efficacy Endpoint | |
| 8.3. | Key Secondary Efficacy Endpoints and Analyses | |
| 8.3. | | 48 |
| 8.3.2 | | |
| Prin | cipal Investigator | 49 |
| | | 10 |
| 8.4. | Additional Efficacy Endpoints and Analyses | |
| 8.4. | , | |
| 8.4.2 | | 50 |
| 8.4.3 | | 52 |
| 8.4.4 | | 53 |
| 8.4. | | 54 |
| 8.4.0 | | |
| 8.4. | 6. Incidence of Status Epilepticus | 54 |
| 8.4.8 | | 50 |
| 8.4.9 | Vineland Adaptive Rehavior Scale (VARS) | 50 |
| 8.4. | | 50<br>57 |
| 8.4. | 11. Zarit Caregiver Burden Inventory | 51 |
| 8.4. | | 50 |
| 8.4. | 13. New Seizure Types | 60 |
| 0.4. | 10. New Ocizaro Types | 00 |
| | 0,076 | |
| 9. <b>S</b> | AFETY | 61 |
| | (6) | |
| 9.1. | Extent of Exposure | 61 |
| 9.2. | Treatment Compliance (Diary) | 61 |
| | Soci | |
| 9.3. | Adverse Events | |
| 9.3. | | |
| 9.3. | | |
| 9.3. | 3. Adverse Events of Special Interest (AESI) | 64 |
| 9.4. | Physical Examination | 65 |
| ٥. | | |
| 9.5. | Neurologic Examination | 65 |
| 0.0 | Vital Signs, Weight, and BMI | |
| 9.6. | vital Signs, weight, and Billings and Billin | bt |
| 9.7. | Electrocardiogram | |
| 9.7. | Electrocardiogram | 66 |
| 9,8. | Doppler Echocardiography | 66 |
| <b>3.</b> 0. | Depple: Lenocardiography | 00 |
| 9.9. | Tanner Staging | 66 |
| J.J. | rainier otaying | 00 |
| 9.10. | Laboratory Parameters | 67 |
| J. 1U. | Euroratory i didinetera | 01 |

| | 9.11. Columbia-Suicide Severity Rating Scale | 69 |
|---|---|---|
| | 9.12. Brief Rating Inventory of Executive Function (BRIEF) | 70 |
| | 10. INTERIM ANALYSES | 71 |
| | 11. CHANGE FROM PLANNED ANALYSES | <b>72</b> |
| | 12. PROGRAMMING CONSIDERATIONS | 76 |
| | 12.1. General Considerations | |
| | 12.2.2. Headers 12.2.3. Display Titles 12.2.4. Column Headers 12.2.5. Body of the Data Display 12.2.6. Footnotes 13. QUALITY CONTROL 14. INDEX OF TABLES, FIGURES, AND LISTINGS 15. REFERENCES 16. APPENDICES 16.1. Appendix 1 – Seizure Types 16.2. Seizure Classification – Primary Endpoint | 8082158159 |
| (his | This document is confidential. | |
| | SAP Text Version 3.0 04-Feb-2022 | |

# 1. GLOSSARY OF ABBREVIATIONS

| Abbreviation | Description |
|--------------|-------------------------------------------------|
| AE | adverse events |
| AED | antiepileptic drugs |
| AESI | adverse event of special interest |
| ALB | albumin |
| ALT; SGPT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AP | alkaline phosphatase |
| AS | atonic seizures |
| AST; SGOT | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | body mass index |
| BRI | Behavioral Regulation Index |
| BRIEF | Behavior Rating Inventory of Executive Function |
| BUN | blood urea nitrogen |
| Ca | calcium |
| CBD | cannabidio |
| CDSF | change in drop seizure frequency |
| CGI-I | Clinical Global Impression – Improvement |
| CI | confidence interval |
| CL | chloride |
| CMH | Cochran-Mantel-Haenszel |
| CO2 | carbon dioxide |
| CS | clonic seizures |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| DCR | Data Change Request |
| DSD X | Daily Seizure Diary |
| DSF | drop seizure frequency |
| ECG | electrocardiogram |
| ЕСНО | echocardiogram |
| eCRF | electronic Case Report Form |
| EMI | Emergent Metacognition Index |
| ESC | Epilepsy Study Consortium |
| ET | Early Termination |

| Abbreviation | Description |
|----------------|----------------------------------------------|
| FI | Flexibility Index |
| FS | focal seizures |
| FSH | Follicle Stimulating Hormone |
| GEC | Global Executive Composite |
| GGT | gamma-glutamyl transferase |
| GH | Growth hormone |
| GTC | generalized tonic-clonic seizures |
| HS | hemiclonic seizures |
| ICH | International Conference on Harmonisation |
| IGF-1 | insulin-like growth factor-1 |
| ILAE | International League Against Epilepsy |
| IMP | Investigational Medicinal Product |
| INR | International normalized ratio |
| ISCI | Inhibitory Self-Control Index |
| IWR | Interactive Web Response system |
| K | potassium |
| kg | kilogram |
| LDH | lactate dehydrogenase |
| LGS | Lennox-Gastaut syndrome |
| LH | Luteinizing Hormone |
| M | Maintenance Period |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| MI | Metacognition Index |
| mITT | Modified Intent-to-Treat Population |
| MS | myoclonic seizures |
| Na | sodium |
| NTF | Note to File |
| PBPK | physiologically-based pharmacokinetic |
| PCDSF | percent change in drop seizure frequency |
| PK | pharmacokinetics |
| PP | Per Protocol Population |
| PT O | Preferred Term |
| PTT | partial thromboplastin time |
| $Q_1$ | 25th Percentile / 1st Quartile |
| Q <sub>3</sub> | 75th Percentile / 3rd Quartile |

| Abbreviation | Description |
|---|---|
| QoL | Quality of Life |
| QOLCE | Quality of Life in Childhood Epilepsy |
| SAF | Safety Population |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SE | status epilepticus |
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| STC | secondarily tonic-clonic |
| T+M | Titration and Maintenance Periods |
| TA | tonic/atonic seizures |
| TEAE | Treatment-emergent adverse events |
| TLF | tables, data listings, figures |
| TS | tonic seizures |
| TSH | thyroid stimulating hormone |
| VABS | Vineland Adaptive Behavior Scale |
| WHO-DD | World Health Organization Drug Dictionary |
| rhis document can | tonic seizures thyroid stimulating hormone Vineland Adaptive Behavior Scale World Health Organization Drug Dictionary This document is confidential. 2022 3A.02, Effective Date 31-Aug-2020 |
| SAP Text Version 3.0 04-Feb<br>Controlled Document ID: <b>390</b><br>Filing requirements: TMF | This document is confidential2022 3A.02, Effective Date 31-Aug-2020 Page 11 of 160 |
| Timing requirements. TWF | 1 age 11 01 100 |

### 2. PURPOSE

The purpose of this statistical analysis plan (SAP) is to ensure that the summary tables, figures, and data listings that will be produced for Part 1 of the trial, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives.

### 2.1. RESPONSIBILITIES

Syneos Health will perform the statistical analyses and are responsible for the production and quality control of all tables, figures and listings with the exception of pharmacokinetics (PK), electrocardiogram (ECG), and echocardiogram (ECHO).

Separate analysis plans for PK and for ECG/ECHO will be produced.

BioMedical Systems, a division of Biomedical System/ERT, will provide analyses of ECG and ECHO data.

### 2.2. TIMING OF ANALYSES

Study 1601 is an international multicenter study being conducted in 2 parts. Up to approximately 80 study sites in North America, Europe, Australia, and Japan are planned to participate. Part 1 is a double-blind, parallel-group, placebo-controlled, study to assess the efficacy and safety of two doses of ZX008 when used as adjunctive therapy for seizures in children and adult subjects with LGS. Part 1 will include 2 cohorts: Cohort A will include randomized subjects from North America, Europe, and Australia; Cohort B will include randomized subjects from Japan.

All objectives will be evaluated in Cohort A and B independently. Data from Part 1, Cohort A will constitute the primary analyses of the study. The primary analyses for Part 1, Cohort A of the study, to include safety, efficacy, and PK, will be conducted once all Cohort A subjects have completed Part 1 of the study and the Per-Protocol (PP) Population and other populations have been defined, and approval for unblinding has been granted by Zogenix International Limited. This analysis will be completed by the primary unblinded statistical team of Syneos Health.

Data from Part 1, Cohort B will be analyzed independently after the last subject in Cohort B completes Part 1 and the PP Population and other populations have been defined, and approval for unblinding of Cohort B has been granted by Zogenix International Limited.

Analysis results for Part 1 from Cohort A and B will be compared through descriptive statistics; that is, the results from Cohort A and B will be compared by reviewing the descriptive statistics calculated from each cohort. Some analyses may be performed using data from Cohorts A and B combined.

Additional analyses for long-term safety and effectiveness data from Part 2 will be completed independently by cohort. The description of the analysis methodology for Part 2 of the study will be provided in a separate SAP.

Cohort A is expected to finish Part 1 before Cohort B. In order to prevent any bias in the completion of Cohort B, whether intentional or unintentional, an unblinding plan will be unblinded and responsible facility. unblinded individuals will have no involvement in study decisions that would have the potential to affect data integrity for Cohort B.

### 3. PART 1 OBJECTIVES

Cohorts A and B will be analyzed independently. Cohort A will be analyzed after the last subject completes Part 1. These analyses will form the main analyses to establish safety and efficacy of ZX008 in patients with LGS. Cohort A Part 1 will be evaluated with formal statistical testing as described below. Cohort B Part 1 will be analyzed after the last subject completes Part 1. Inferential statistics for Cohort B will be evaluated using the same methodology stated for Cohort A, but the inferential statistics will be considered as descriptive.

### 3.1. **PRIMARY OBJECTIVE**

The primary objective of Part 1 is the primary objective of the entire study. The primary objective of Part 1 is:

To evaluate the effect of ZX008 0.8 mg/kg/day versus placebo as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with Lennox-Gastaut syndrome (LGS) based on the change in frequency of seizures that result in drops (DSF) between baseline and the combined Titration and Maintenance Periods (T+M).

Seizures that result in drops include seizures of the following types that have been reviewed and confirmed for each subject as a drop seizure by the Epilepsy Study Consortium (ESC): generalized tonic-clonic seizures (GTC), secondarily generalized tonic-clonic seizures (SGTC), tonic seizures (TS), atonic seizures (AS), tonic/atonic seizures (TA).

### KEY SECONDARY OBJECTIVE

The key secondary objectives of Part 1 are:

To evaluate the effect of ZX008 0.2 mg/kg/day versus placebo as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with LGS based on the change in DSF between baseline and T+M.

- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the proportion of subjects who achieve a  $\geq$  50% reduction from baseline in the frequency of seizures that result in drops.
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the Clinical Global Impression - Improvement (CGI-I) rating, as assessed by the Principal Investigator.

### 3.3. ADDITIONAL SECONDARY OBJECTIVES

The additional secondary objectives specified in this section have been modified from those given in the protocol. Those modifications are described in detail in Section 11. The additional secondary endpoints specified in Section 5.3, and their corresponding analyses, are based on the objectives as specified in this section.

Additional secondary objectives of Part 1 of the study are:

- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints:
  - Change in frequency of all seizures that (typically) result in drops (i.e., GTC, SGTC, TS, AS, TA) between baseline and T+M whether ESC confirmed as drop or not.
  - Change in the frequency of all countable motor seizures between baseline and T+M (countable seizures include: GTC, SGTC, TS, AS, TA, clonic seizures [CS], focal seizures with clear observable motor signs [FS], and hemiclonic seizures [HS]).
  - Change in the frequency of all countable non-motor seizures between baseline and T+M (countable non-motor seizures include: absence, myoclonic, focal without clear observable motor signs, infantile spasms, and epileptic spasms)
  - Change in the frequency of all countable seizures (i.e., motor and nonmotor) between baseline and T+M
  - Change in frequency of seizures that result in drops (ESC confirmed) between baseline and the Maintenance Period (M)
  - Change in frequency of seizures that (typically) result in drops between baseline and the Maintenance Period (M)
  - Change in the frequency of all countable motor seizures between baseline and M
  - Change in the frequency of all countable non-motor seizures between baseline and M
    - Change in the frequency of all countable seizures (i.e., motor and nonmotor) between baseline and M
  - The proportion of subjects who achieve a worsening, >0, ≥25%, ≥50%, ≥75%, 100% reduction, and "near seizure freedom" (i.e. 0 or 1 seizures) between baseline and T+M, and baseline and M, in seizures that result in drops (ESC confirmed), seizures that typically result in drops, all

- countable motor seizures, all countable non-motor seizures, and all countable seizures
- Number of seizure-free days, defined as 1) no seizures that result in drops (ESC confirmed), and 2) days with no countable motor seizures
- Longest interval between seizures that result in drops (ESC confirmed)
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the CGI-I rating, as assessed by the parent/caregiver.

### 3.4. SAFETY OBJECTIVES

The safety objectives of Part 1 are:

- To evaluate the safety and tolerability of ZX008 0.2 and 0.8 mg/kg/day versus
  placebo with regard to adverse events (AEs), laboratory parameters, physical
  examination, neurological examination, vital signs (blood pressure, heart rate,
  temperature, and respiratory rate), electrocardiograms (ECG), echocardiograms
  (ECHO), body weight, and body mass index (BMI)
- To evaluate the change from baseline in cognition using age-appropriate versions of the Behavior Rating Inventory of Executive Function (BRIEF)

### 3.5. PHARMACOKINETIC OBJECTIVES

The pharmacokinetic (PK) objective of the study is:

 To evaluate the PK of ZX008 0.2 and 0.8 mg/kg/day at steady state in subjects < 18 years and ≥18 years with LGS using a non-compartmental analysis and obtain exposure data that will be used in population pharmacokinetic (PopPK) analysis, the results of which will be reported separately.

### 3.6. EXPLORATORY OBJECTIVES

The exploratory objectives of the study are:

- To compare the ZX008 0.2 and 0.8 mg/kg/day doses on primary, secondary, and safety endpoints.
- To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints:
  - The change from baseline in behavior using the Vineland Adaptive Behavior Scale (VABS)
  - The change from baseline in quality of life (QoL) using the QOLCE
    The change from baseline in caregiver burden using the Zarit Caregiver
    Burden Inventory
  - The change from baseline in affective symptoms of the parent/caregiver using the Hospital Anxiety and Depression Scale (HADS)
  - The frequency of rescue medication usage
  - The incidence of medical services to treat seizures

- The incidence of status epilepticus (SE)

### 4. BRIEF DESCRIPTION

Study 1601 is an international multicenter study being conducted in two parts. Up to approximately 80 study sites in North America, Europe, Australia, and Japan are planned to participate. Part 1 is a double-blind, parallel-group, placebo-controlled, study to assess the efficacy and safety of two doses of ZX008 when used as adjunctive therapy for seizures in children and adult subjects with LGS. Part 1 will include 2 cohorts: Cohort A will include randomized subjects from North America, Europe, and Australia; Cohort B will include randomized subjects from Japan. The main analyses for the study, including the primary and key secondary study endpoints are assessed from Part 1, Cohort A data. The primary analysis will be conducted when the last subject in Cohort A has completed Part 1. Part 2 will be an open-label, flexible-dose extension for subjects completing Part 1 of the study.

Part 1 consists of a 4-week Baseline, 2-week Titration, 12-week Maintenance, and 2-week Taper or Transition Period. The 4-week Baseline Period consists of the establishment of initial eligibility during a screening visit to include an assessment of cardiac parameters (ECG and ECHO), followed by an observation period where subjects will be assessed for baseline seizure frequency based on recordings of daily seizure activity entered into a diary. Upon completion of the Baseline Period, subjects who qualify for the study are randomized (1:1:1) in a double-blind manner to receive 1 of 2 doses of ZX008 (0.2 mg/kg/day, 0.8 mg/kg/day; maximum dose: 30 mg/day [or 0.5] mg/kg/day, maximum 20 mg/day, for subjects taking concomitant STP]) or placebo. Randomization is stratified by weight (<37.5 kg, ≥37.5 kg) to ensure balance across treatment arms, and at least 25% of subjects will be in each weight group. All subjects are titrated to their blinded randomized dose over a 2-week Titration Period. Following titration, subjects continue treatment at their randomly assigned dose over a 12-week Maintenance Period. Total treatment time from the beginning of the Titration Period through the end of the Maintenance Period is 14 weeks. Subjects will have ECG and ECHO assessments at weeks 6 and 14 during the Maintenance Period. At the end of the Maintenance Period (or early discontinuation), all subjects undergo a blinded 2-week Taper or Transition Period depending on whether they exit the study or are enrolled in Part 2, the long-term open-label extension, respectively. Cardiac safety follow-up visits are performed after study drug discontinuation for early termination, or for those subjects who complete the study but do not enter the open-label extension part. All subjects are required to have follow-ups at 3 and 6 months. Subjects enrolled in Germany, France and Netherlands will have an additional follow-up at 24 months. If there are any findings at a post-dose follow-up, a follow-up visit will be scheduled every 3 months until resolved or stabilized.

Part 2 is an open-label, long-term safety study of ZX008 for subjects who have successfully completed 14 weeks of treatment (titration + maintenance) in Part 1 and are candidates for continuous treatment for an extended period of time; subjects who have not completed the entire 14 weeks of treatment in Part 1 may be eligible to

participate in Part 2 on a case-by-case basis and only following Sponsor approval. Part 2 consists of a 12-month Open-Label Extension (OLE) Treatment Period and a 2-week Post-Dosing Period. Thus, subjects who were randomized to ZX008 during Part 1 and

During Part 2, all subjects are treated initially with ZX008 0.2 mg/kg/day for 1 month to assess effectiveness of this dose in all study subjects. After 1 month at a dose of 7000 effectiveness and tolerability 2 ZX008 0.2 mg/kg/day, to a maximum of ZX008 0.8 mg/kg/day (or ZX008 0.5 mg/kg/day) for subjects taking concomitant STP) but not to exceed total dose of 30 mg/day (or. 20mg/kg/day for subjects taking concomitant STP). During the 12-month OLE subjects will have ECG and ECHO assessments at months 1, 3, 6, and 9, and at the end of study visit.

A follow-up ECG and ECHO will be performed at 3 and 6 months after study drug discontinuation for early termination and for those subjects who complete Part 2. Subjects enrolled in Germany, France and Netherlands will have an additional follow-up at 24 months. If there are any findings at a post-dose follow-up, another follow-up will be scheduled every 3 months until resolved or stabilized. In both Part 1 and Part 2, parents/caregivers will use a diary every day to record dosing of study drug, the number of seizures, type of seizures, time and duration of seizures, whether the seizure resulted in a drop, and use of rescue medication.

### SUBJECT SELECTION 4.1.

The inclusion and exclusion criteria are stated in full in Sections 4.1, 4.2, and 4.3 of the protocol document.

### 4.2. DETERMINATION OF SAMPLE SIZE

The sample size was estimated for Part 1 Cohort A under the assumption that adding ZX008 at 0.8 mg/kg/day to current therapy will lead to a mean decrease in drop seizures that is 30 percentage points greater than adding placebo to current therapy. For example, if adding placebo leads to a 10% decrease in seizures, then adding the ZX008 0.8 mg/kg/day dose would be expected to decrease seizures by at least 40%. The variability expected in the trial was estimated from a Phase 3 trial of clobazam for patients with Lennox-Gastaut syndrome (Ng 2011) leading to an assumption that the standard deviation (SD) is 50%. Other assumptions include an allowance for 20% dropouts between randomization and the start of the maintenance period. Under these assumptions, a sample size of 63 subjects per treatment group for a nonparametric analysis affords 90% power to detect a difference between the ZX008 0.8 mg/kg/day and placebo groups that is significant at the  $\alpha$ =0.05 level. Assuming a 20% drop-out rate prior to the start of the maintenance period yields a requirement for an additional 14

subjects per group for a total of 79 subjects per treatment group for a nonparametric analysis. Similar calculations for the ZX008 0.2 mg/kg/day group lead to a total required sample size of 237. The number of subjects randomized into Part 1 Cohort A is estimated to be approximately 250 due to the long baseline period.

The sample size of 10 to 15 subjects per treatment group in Cohort B is expected to provide a descriptive assessment of whether the treatment effect in Japanese subjects is similar to that observed in Cohort A subjects from the rest of the world.

### 4.3. TREATMENT ASSIGNMENT & BLINDING

Upon completion of the Baseline Period in Part 1, subjects who qualify for the study are randomized (1:1:1) in a double-blind manner to receive 1 of 2 doses of ZX008 (0.2 mg/kg/day, 0.8 mg/kg/day; 30mg/day maximum [0.2 mg/kg/day or 0.5 mg/kg/day; 20 mg/day maximum for subjects taking concomitant STP]) or placebo. The randomization is stratified by weight (< 37.5 kg,  $\geq$  37.5 kg) to ensure balance across treatment arms, with a target of at least 25% in each weight group. Subjects are assigned a randomization number by the Interactive Web Response (IWR) system upon confirmation that the subject qualifies for enrollment in the Titration Period.

The primary biostatistical team, data management team, and clinical team will remain blinded to Cohort A subject treatment assignments until approval is given for the unblinding of the Part 1, Cohort A database and finalization of subject inclusion in the study populations is made. Similarly, the primary biostatistical team, data management team, and clinical team will remain blinded to Cohort B subject treatment assignments until approval is given for the unblinding of the Part 1, Cohort B database and finalization of inclusion in the study populations is made.

The release of unblinded PK concentration, ECG, and ECHO data to facilitate external analyses will be completed only after the approval for unblinding of the Part 1 Cohort A and Part 1 Cohort B databases by Zogenix.

### 4.4. ADMINISTRATION OF STUDY MEDICATION

Each bottle of study medication contains the appropriate concentration and volume of liquid to administer the assigned treatment (ZX008 0.2 mg/kg/day, ZX008 0.8 mg/kg/day [or 0.5 mg/kg/day for subjects taking concomitant STP], or placebo). ZX008 and placebo are identical, thus rendering the study drug and placebo indistinguishable.

The blinding scheme instituted for this study ensures that the volume of study medication taken cannot be associated with the dose group, thus unblinding the study. This is achieved by random assignment of different concentrations of ZX008 or placebo (1.25 mg/mL, 2.5 mg/mL, and/or 5 mg/mL) by the IWR system. The IWR system instructs site personnel to the volume of oral solution to be administered based on that subject's weight. (Dose is recalculated by the system based on weight once at the midpoint of Part 1 of the study.) During the Titration, Maintenance, and

Taper/Transition Periods, the subjects and study personnel (investigators, clinical staff, personnel involved in data collection and analysis, the Medical Monitor, and the sponsor) are blinded to the treatment allocation and to the concentration of ZX008. If an investigator feels the blind should be broken, he/she can do so when necessary for treatment decisions. However, the investigator should endeavor to discuss with the Medical Monitor or Sponsor's Medical Representative, if available. The blind should only be broken in the event the knowledge of whether the subject is on active study medication versus placebo is needed to determine course of medical treatment for the event. The subject will be discontinued from the clinical trial upon breaking of the blind and the decision whether the subject can enter Part 2 will rest with the Sponsor if the subject exited Part 1 prior to completion.

Following randomization, subjects enter the Titration Period and are blindly titrated to their randomized dose as outlined in Table 1.

Table 1: Titration Algorithm for Part 1

| Tuble 1: The action Algorical for Fall C | | | |
|---|---|---|---|
| Randomized Group | Titration Step 1 | | Titration Step 3 |
| | Study Days 1-4 | Study Days 5-8 | Study Days 9-14 |
| ZX008 0.2 | ZX008 0.2 | ZX008 0.2 | ZX008 0.2 |
| mg/kg/day | mg/kg/day | mg/kg/day | mg/kg/day |
| ZX008 0.8 | ZX008 0.2 | ZX008 0.4 | ZX008 0.8 |
| mg/kg/day (0.5 | mg/kg/day | mg/kg/day | mg/kg/day |
| mg/kg/day for | | 04 6 | (0.5 mg/kg/day for |
| subjects taking | | 0,1 | subjects |
| concomitant STP) | 10, 20 | <i>'</i> (0') | taking concomitant |
| | V), XO | 25, | STP) |
| Placebo | Placebo | Placebo | Placebo |

After completion of the Titration Period, subjects enter the Maintenance Period and continue to receive the randomized dose of ZX008 or placebo and be treated for an additional 12 weeks.

Subjects who complete the Maintenance Period and do not be continue into Part 2, the open-label extension, and subjects who discontinue from Part 1 early, will be tapered off of study medication as outlined in Table 2.

Table 2: Taper Algorithm for Part 1

| Randomized Group | Taper Step 1 Day 1-4 after study completion or early termination | Taper Step 2 Days 5-8 after study completion or early termination |
|---|---|---|
| ZX008 0.2 mg/kg/day | Placebo | Placebo |
| ZX008 0.8 mg/kg/day (0.5 mg/kg/day for subjects taking concomitant STP) | ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day |

Sponsor: Zogenix International Limited; Protocol No.: ZX008-1601

| Randomized Group | Taper Step 1 Day 1-4 after study completion or early termination | Taper Step 2 Days 5-8 after study completion or early termination |
|---|---|---|
| Placebo | Placebo | Placebo |

Subjects who complete the Maintenance Period and will be continuing into the openlabel extension (Part 2) will be transitioned from double-blind study medication to open-label ZX008. All subjects entering the open-label extension (Part 2) will be transitioned from their blinded daily dose to the ZX008 0.2 mg/kg/day dose during the 2-week interval between Visits 12 and 15, without breaking the blind. The IWR system will assign two bottles of Investigational Medicinal Product (IMP) to the subject, one for each step in the transition. A new bottle of IMP will be started by the subject at each

| transitioned from their blinde<br>2-week interval between Visit<br>will assign two bottles of Inve | s entering the open-label extended daily dose to the ZX008 0.2 m<br>cs 12 and 15, without breaking the stigational Medicinal Product (Innew bottle of IMP will be started | ng/kg/day dose during the<br>the blind. The IWR system<br>MP) to the subject, one for |
|---|---|---|
| Table 3: Transition Algorithm | n for Part 1 | Marions |
| Dose Group in Double-<br>Blind Study<br>ZX008 0.2 mg/kg/day | Transition Step 1 Day 1-4 after Visit 12 ZX008 0.2 mg/kg/day | Transition Step 2 Day 5-14 after Visit 12 ZX008 0.2 mg/kg/day |
| ZX008 0.8 mg/kg/day (0.5 mg/kg/day for subjects taking concomitant STP) | ZX008 0.4 mg/kg/day | ZX008 0.2 mg/kg/day |
| Placebo | ZX008 0.2 mg/kg/day | ZX008 0.2 mg/kg/day |
| Placebo The full list and timing of study SAP Text Version 3 0 04-Feb-2022 | dany exter | |
| | This document is confidential. | |
| SAP Text Version 3.0 04-Feb-2022<br>Controlled Document ID: <b>3903A.02</b> , Effec<br>Filing requirements: TMF | | Page <b>20</b> of <b>160</b> |

Statistical Analysis Plan for Interventional Studies
Sponsor: Zogenix International Limited; Protocol No.: ZX008-1601

| | | | | able 4 | - Schedu | Table 4 – Schedule of Assessments | ssments | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | • | | rart I As | rart i Assessments | | | | | • | • | • | |
| Study Assessments - PART 1 | Baselin | e Perioda | a Ta | | | Titra | Titration + Maintenance Period | ntenance | Period | | | FO6/ | Doct | Cardiac |
| Visit Number | Screening | | Random-<br>ization | Ţ | Titration Period | riod | | Main | Maintenance Period | eriod | | EUS/ | rost-<br>Dosing <sup>1</sup> | rollow-<br>up <sup>c</sup> |
| | | 2<br>Phone) | 8 | | 4, 5 (Phone) | 9 | 7<br>(Phone) | ∞ | 9<br>(Phone) | 10 | 11<br>(Phone) | 12 | 13 | 14 |
| Study Day | -28 | 45 | -1 | 1 | 4,8 | 15 | 29 | 43 | 57 | 71 | 85 | 66 | 113 | 197 |
| Informed Consent (subject and parent/caregiver) | × | 7 | | 0 | | | | | | | | X<br>(Part 2) | | |
| Inclusion/Exclusion Criteria | × | Ó | X | , | 8 | | | | | | | | | |
| Demographics | × | | 7 | 6 | | . ( | | | | | | | | |
| Medical/Neurological History | × | | 0 | | | - ( | | | | | | | | |
| Epilepsy history | × | | | . 0 | 5 | 5 | | | | | | | | |
| Review retrospective seizure diary data | × | | | ,,,, | ),<br>}, | | 78 | | | | | | | |
| Prior Medication, including<br>AEDs | × | | × | | 2100 | 2/2 | | | | | | | | |
| Physical Examination, complete | × | | × | | | ď | | | | | | X | | Optional |
| Physical Examination, abbreviated | | | | | | Xm | 3 | Xm | | Xm | | | | × |
| Neurological Examination, complete | × | | | | | | S | 9 | \( \) | | | × | | |
| Neurological Examination,<br>abbreviated | | | × | | | Xm | | mX S | Tijs | Xm | | | | |
| Vital signs | X | | X | | | X | | X | ×, | × | | X | | |
| SAP Text Version 3.0 04-Feb-2022<br>Controlled Document ID: <b>3903A.02</b> , Effective Date 31-Aug-2020<br>Filing requirements: TMF | ctive Date 31. | Aug-202 | 0 | This d | ocument is | This document is confidential. | ifal. | Pag | Page 21 of 160 | of 160 | .HOİİL | Moil Lation | ~ | |

This document is confidential.

Statistical Analysis Plan for Interventional Studies Sponsor: Zogenix International Limited; Protocol No.: ZX008-1601

| CUIT | | | | Fable 4 | Table 4 – Schedule of Assessments Part 1 Assessments | le of Asse<br>sessment | ssments | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Assessments - PART 1 | Baseli | Baseline Period <sup>a</sup> | $\mathbf{d}^{\mathrm{a}}$ | | | Titra | Titration + Maintenance Period | intenance | Period | | | /504 | Dest | Cardiac |
| Visit Number | Screening | | Random-<br>ization | Ti | Titration Period | riod | | Main | Maintenance Period | eriod | | ET <sup>b</sup> | Fost-<br>Dosing <sup>1</sup> | rollow-<br>up <sup>c</sup> |
| COL | ari | 2<br>(Phone) | e | | 4, 5<br>(Phone) | 9 | 7<br>(Phone) | ∞ | 9<br>(Phone) | 10 | 11<br>(Phone) | 12 | 13 | 14 |
| Study Day | -28 | Q<br>S | -1 | 1 | 4,8 | 15 | 29 | 43 | 57 | 71 | 85 | 66 | 113 | 197 |
| Weight | X | Ó, | × | < | | × | | X | | × | | × | | |
| Height | × | 6 | | 5, | | | | | | | | × | | |
| Chest x-ray (France, Netherlands only) | | 0 | × ^ | 3 | 8) | | | | | | | × | | × |
| 12-lead ECG | × | • | ×G | > | | _ | | X | | | | × | | × |
| Doppler ECHO | × | | ** | × | 9 | | | $X^{\mathrm{d}}$ | | | | $X^{q}$ | | X |
| Urine or Serum Pregnancy Test | Xe | | Xe | e S | | | <b>(</b> | Xe | | | | Xe | | |
| Clinical laboratory evaluation (hematology/ chemistry/urinalysis°, etc) | × | | × | 6 | , (C | oc | 27 | X | | | | × | | |
| Plasma sample for ZX008 PK | | | | | 0. | | | $X^{\mathrm{f}}$ | | | | | | |
| Plasma sample for background<br>AEDs PK | | | Xg | | | 8 | dilly | X | | Xg | | Xg | | |
| Whole blood CBD/ THC Panel | × | | X | | | 70 | .0 | 2x | | | | × | | |
| Tanner Staging (for subjects >7 to 18 years old) | | | × | | | | | Oil | NL. | | | × | | |
| Subject Diary | D | R | C/R/D | | R | C/R/D | R | C/R/D | Š | C/R/D | N | C/R/Dh | C/R | |
| Epilepsy genotype panel (optional) | | | | | | | | S | | Ò | | | | |
| Study Medication | | | D | | $\mathbb{R}^{\mathrm{i}}$ | C/R/D | R | C/R/D | R | C/R/D | R | C/R/Dh | C/R | |
| SAP Text Version 3.0 04-Feb-2022<br>Controlled Document ID: <b>3903A.02</b> , Effective Date 31-Aug-2020<br>Filing requirements: TMF | ctive Date 3' | -Aug-203 | 50 | This do | This document is confidential | confiden | ial. | Pag | Page <b>22</b> of <b>160</b> | 0 | HOHIL | riValion | | |

This document is confidential.

Statistical Analysis Plan for Interventional Studies Sponsor: Zogenix International Limited; Protocol No.: ZX008-1601

| CUI | | | | rable 4 | – Schedu<br>Part 1 As | Table 4 – Schedule of Assessments<br>Part 1 Assessments | ssments | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Assessments - PART 1 | Baseli | Baseline Perioda | ďa | | | Titrat | Titration + Maintenance Period | ntenance | Period | | | 7201 | 4 | Cardiac |
| Visit Number | Screening | _ | Random-<br>ization | Tit | Titration Period | riod | | Main | Maintenance Period | eriod | | ET <sup>b</sup> | Fost-<br>Dosing <sup>1</sup> | rollow-<br>up <sup>c</sup> |
| Cor | di. | 2<br>(Phone) | 8 | | 4, 5<br>(Phone) | 9 | 7<br>(Phone) | ∞ | 9<br>(Phone) | 10 | 11<br>(Phone) | 12 | 13 | 14 |
| Study Day | -28 | 015 | -1 | - | 4,8 | 15 | 29 | 43 | 57 | 71 | 85 | 66 | 113 | 197 |
| C-SSRS | X | O, | × | < | | X | | X | | × | | X | | |
| Clinical Global Impression -<br>Improvement (assessed by<br>parent/caregiver) | | 90 | USE | 50 | (8) | × | | × | | × | | × | | |
| Clinical Global Impression -<br>Improvement (assessed by<br>Principal Investigator) | | | Jet | 9,0 | | × | | × | | × | | X | | |
| HADS (Effect of parent/caregiver) | | | × | ein' | | | R | | | | | × | | |
| BRIEF | | | × | 5, | C | CO | 7 | | | | | × | | |
| VABS | | | X | | 0 | | | × | | | | X | | |
| богсе | | | × | | ) | O. | S. | | | | | × | | |
| Zarit Burden | | | X | | | 1 | 7 | X | | | | X | | |
| Randomize subject | | | Xu | | | 70 | S | | | | | | | |
| First Day of Study Drug<br>Administration <sup>j</sup> | | | | × | | | Sil | dir | _16 | | | | | |
| Daily Diary Completion | | | | | | | × | 5 | | | | | | |
| Concomitant Medication | | | | | | | | S | ×× | | | | | |
| Adverse events | | | | | | | X | <b>.</b> | 2 | 0 | | | | |
| SAP Text Version 3.0 04-Feb-2022<br>Controlled Document ID: <b>3903A.02</b> , Effective Date 31-Aug-2020<br>Filing requirements: TMF | ective Date 31 | I-Aug-202 | 00 | This do | ocument is | This document is confidential | ial. | Pag | Page <b>23</b> of <b>160</b> | of 160 | *KOİİL | orilation | | |

This document is confidential.

# Statistical Analysis Plan for Interventional Studies

Sponsor: Zogenix International Limited; Protocol No.: ZX008-1601

| | | | | Fable 4 | Table 4 – Schedule of Assessments<br>Part 1 Assessments | le of Asse | ssments | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Assessments - PART 1 | Baseli | Baseline Period <sup>a</sup> | $\mathbf{d}^{\mathrm{a}}$ | | | Titrat | Titration + Maintenance Period | ntenance | Period | | | FOS/ | Post | Cardiac<br>Follow |
| Visit Number | Screening | | Random-<br>ization | Ti | Titration Period | riod | | Main | Maintenance Period | eriod | | ET <sup>b</sup> | ET <sup>b</sup> Dosing <sup>1</sup> up <sup>c</sup> | up <sup>c</sup> |
| Co | | 2<br>(Phone) | 8 | | 4, 5 (Phone) | 9 | 7<br>(Phone) | ∞ | 9<br>(Phone) | 10 | 11<br>(Phone) | 12 | 13 | 14 |
| Study Day | 82- | Ols | -1 | 1 | 4,8 | 15 | 29 | 43 | 57 | 71 | 82 | 66 | 113 | 197 |
| Adverse events of special interest | Ò | Q | | • | | | X | | | | | | | $\chi_{\mathrm{k}}$ |

Abbreviations: AED=antiepileptic drug; BMI=body mass index; C=Collect; CBD=cannabidiol; D=Dispense; ECG=electrocardiogram; EQ-5D-5L=standardized measure of health status; EOS=end of study; ET=early termination; HADS=Hospital Anxiety and Depression Scale; BRIEF=Behavior Rating Inventory of Executive Function; QoL=quality of life; R=Review; VABS=Vineland Adaptive Behavior Scale

- The Baseline Period is comprised of the initial screening for the study and the assessment of baseline seizure activity recorded daily in the diary. The procedures to be completed at the Screening visit may be completed in a single day or split so that they are completed over the 2-day period.
- Subjects who are discontinued early and those who complete the study and choose not to enroll in the separate open-label extension will be tapered off study medication over an up to 2-week þ:
- The safety follow-up visit will be conducted for subjects who either terminate early from Part 1, or who complete Part 1 but do not enter Part 2. Standard follow-up visits should occur 3 and 6 months after the last dose. For subjects enrolled in Germany, France and Netherlands, follow-ups will also occur 24 months after the last dose. If there are any findings at the last post-dose follow-up, a follow-up visit will be repeated every 3 months until resolved or stabilized.
  - The Visit 8 ECHO must be performed any time between Study Day 40 and Study Day 54. The Visit 12 ECHO must be performed any time between Study Day 90 and Study Day 113; if a subject discontinues early from the study, the ECHO should be scheduled as soon as practical. If the Study Day 43 ECHO was completed < 30 days prior to early termination, the Visit 12 ECHO will not be performed provided the parent/guardian agrees to bring the subject to the cardiac follow-up visit. <del>...</del>
    - Females of child-bearing potential
- Plasma sample for pharmacokinetic assessment will be conducted prior to the dose at Visit 8 and 1, 2, and 4.6 hours after dose administration.
- Plasma sample for assessment of background AED(s) will be conducted prior to the dose of AED(s) at Visits 3. 8 and 12 (Visits 6 and 10 only if clinically indicated). AED plasma sample may be collected after the morning dose of AEDs are taken, if preferable, as long as the time of last dose is accurately recorded. ä
  - þ:
- Study drug administration begins in the morning of Study Day 1. Study Day 1 is considered the first day of dosing, even though subjects may receive an in-clinic dose on Study Day -1. If the drug/diary unspecified to unspecified to unspecified the subject diary; the unspecified administration begins in the morning of Study Day 1. Study Lay 1... at dose is taken in the clinic, it will be recorded in the eCRF, but not the subject diary; the unspecified staken in the clinic, it will be collected at this visit.

  Visit 13 may be conducted as a phone call, provided diaries and study medication are returned by this time.

  An abbreviated physical and/or neurological examination to be conducted as appropriate based on last exam and reported AEs.

  This document is confidential.

Controlled Document ID: 3903A.02, Effective Date 31-Aug-2020 SAP Text Version 3.0 04-Feb-2022 Filing requirements: TMF

Statistical Analysis Plan for Interventional Studies

Sponsor: Zogenix International Limited; Protocol No.: ZX008-1601

| ocument | SAP Text Version 3.0 04-Feb-2022 Controlled Document ID: <b>3903A.02</b> , Effective Date 31-Aug-2020 Filing requirements: TMF |
|---|---|

The targeted study day and allowable windows for visits in Part 1 are reproduced from the protocol below. Early termination visits will be mapped to a visit based on these windows.

Table 5: Visit windows for Part 1 Visits

| Table 5. Visit Willdows for Part 1 Visits | |
|---|---|
| | Time window (relative to |
| | scheduled visit / |
| Visit / Procedure | procedure) |
| Visit 1 (Clinic; Study Day -29 to -28 or -28 to -27): | Not Applicable |
| Visit 2 (Phone; Study -15) | ± 3 days |
| Visit 3 (Clinic; Study Day -1; Randomization | ± 4 days <sup>a</sup> |
| Visits 4, 5 (Phone: Study Days 4, 8) | ± 3 days |
| Visit 6 (Clinic; Study Day 15) | ± 4 days |
| Visit 7 (Phone; Study Day 29) | ± 4 days |
| Visit 8 (Clinic; Study Day 43) | ± 4 days |
| Visit 9 (Phone: Study Day 57) | ± 4 days |
| Visit 10 (Clinic; Study Day 71) | ± 4 days |
| Visit 11 (Phone: Study Day 85) | ± 4 days |
| Visit 12 (Clinic: Study Day 99) | ± 4 days |
| Visit 13 (Clinic; Study Day 113; post dosing) | ± 4 days |
| Visit 14 (ECHO clinic; 3-24 months after last dose) <sup>b</sup> | + 30 days |

AED=antiepileptic drug (s); ECHO=echocardiogram

## 5. ENDPOINTS

### 5.1. PRIMARY EFFICACY ENDPOINT

Percent change from baseline in DSF in T+M in the ZX008 0.8 mg/kg/day group compared to the placebo group. Seizures that result in drops are GTC, SGTC, TS, AS, and TA confirmed for each subject as a drop seizure by the ESC.

### 5.2. KEY SECONDARY EFFICACY ENDPOINTS

The key secondary endpoints are:

<sup>&</sup>lt;sup>a</sup> In cases where the screening period is extended beyond 28 days, the immediate 28 days before the Randomization visit will be used to calculate the baseline seizure frequency

<sup>&</sup>lt;sup>b</sup> All subjects are required to have follow-ups at 3 and 6 months post-treatment. Subjects enrolled in Germany, France and Netherlands will have an additional 24-month follow-up.

- Change from baseline in DSF in T+M in the ZX008 0.2 mg/kg/day group compared to the placebo group.
- Proportion of subjects who achieve a ≥50% reduction from baseline in DSF
- rioportion of subjects who achieve improvement (minimally, much, or very much improved) in the Clinical Global Impression Improvement as assessed by the Principal Investigator, comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo.

  ADDITIONAL SECONDATE:

### 5.3.

The additional secondary endpoints are:

ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups compared independently versu placebo on the

- Change from baseline during T+M in frequency of all seizures that (typically) result in drops (i.e., GTC, SGTC, TS, AS, TA) whether ESC confirmed as drop or not.
- Change from baseline during T+M in frequency of all countable motor seizures (GTC, SGTC, TS, AS, TA, CS, FS, and HS).
- Change from baseline during T+M in frequency of all countable non-motor seizures (absence, myoclonic, focal without clear observable motor signs, infantile spasms, and epileptic spasms).
- Change from baseline during T+M in the frequency of all countable seizures (i.e., motor and non-motor).
- Change from baseline during W in DSF
- Change from baseline during M in the frequency of seizures that typically result
- Change from baseline during M in the frequency of all countable motor seizures.
- Change from baseline during M in the frequency of all countable non-motor
- Change from baseline during M in the frequency of all countable seizures (i.e., motor and non-motor).
- Proportion of subjects who achieve a worsening from baseline (ie,  $\leq 0$ % reduction), or > 0%,  $\ge 25\%$ ,  $\ge 50\%$ ,  $\ge 75\%$ , or 100% reduction between baseline and T+M, and baseline and M, in seizures that result in drops (ESC confirmed), seizures that typically result in drops, all countable motor seizures, all countable non-motor seizures, and all countable seizures.
- Number of seizure-free days in the baseline, M, and T+M periods, defined as 1) days with no seizures that results in drops (ESC confirmed), and 2) days with no countable motor seizures

- The longest interval (days) between seizures that result in drops (ESC Laboratory safety (hematology, chemistry, urinalysis)
  Vital signs (blood pressure, heart rate, temperature, and respiratory (ate)
  Body weight and BMI
  Physical examination
  Neurological examination
  BRIEF to measure changes in cognition of the subject
  Columbia Suicidality Severity Rating Scale (C-SSRS)
  12-lead ECGs
  )oppler ECHOs
  Thest x-ray (for subjects enrolled in France and EG (for subjects enrolled in Italy confirmed) comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups

### 5.4.

The safety endpoints for Part 1 of the study are:

### **EXPLORATORY ENDPOINTS** 5.5.

The exploratory endpoints for Part 1 of the study are

- The change from baseline in behavior using the VABS
- The change from baseline in QoL using the QOLCE
- The change from baseline in caregiver burden using the Zarit Caregiver Burden Inventory
- The change from baseline in affective symptoms of parent/caregiver using the HADS scale
- Incidence of SE in the M and T+M period.
- Incidence of rescue medication usage in the T+M and M periods
- Number of days rescue medication used in the T+M and M periods
- Incidence in use of medical services to treat seizures in the M and T+M periods

### 6. ANALYSIS SETS

Separate analysis datasets will be produced for Cohort A and Cohort B. Cohort A will include subjects from North America, Europe, and Australia; Cohort B will include subjects from Japan.

### 6.1. ENROLLED POPULATION

The Enrolled Population is defined as all subjects who signed the informed consent form.

### 6.2. SAFETY (SAF) POPULATION

All Part 1 safety analyses will be performed on the SAF Population, defined as all randomized subjects who receive at least one dose of ZX008 or placebo.

### 6.3. MODIFIED INTENT-TO-TREAT (MITT) POPULATION

The mITT Population is defined as all randomized subjects who receive at least one dose of ZX008 or placebo and for whom at least one week of diary data are available. Subjects will be analyzed according to the treatment group to which they were randomized. The primary comparison of ZX008 0.8 mg/kg/day to placebo, as well as key secondary analyses, will be performed on the mITT Population.

### 6.4. PER PROTOCOL (PP) POPULATION

The PP Population is defined as all randomized subjects who receive at least one dose of ZX008 or placebo, who complete at least 4 weeks of diary data in the maintenance period, and who have no major protocol deviations that would have a significant impact on clinical outcome of Part 1 data, and who have met the inclusion criteria for baseline drop seizure count. Protocol deviations that occurred during Part 1 will be reviewed and the list of deviations warranting exclusion from the PP Population will be finalized prior to study unblinding.

# 6.5. PROTOCOL DEVIATIONS

Major protocol deviations will be summarized overall and by treatment group based on the SAF Population. Major protocol deviations are those that have the potential to impact subject safety and/or affect data integrity and/or the efficacy conclusions. Major protocol deviations will be grouped into categories and may include categories such as:

- Violation of inclusion/exclusion criteria
- Violation of randomization inclusion criteria
- Non-compliance regarding intake of IMP
- Inappropriate intake of concomitant medication
- Subject not discontinued as per protocol
- Other non-compliance

Multiple deviations can occur in the same subject and thus a subject can be counted in more than 1 deviation category.

For each study part and cohort, major protocol deviations will be presented in a subject data listing for the Enrolled Population, sorted by treatment, site, subject, and type.

Deviations will be reviewed prior to the database lock of Part 1 data for each cohort to determine which deviations will be classified as leading to exclusion from the PP Population.

During the determination of the PP Population for Part 1 Cohort A, the decision was made to exclude from the PP Population those subjects who had a baseline ESC-confirmed drop seizure count value of < 6 per 28 days as well as subjects who had less than 4 weeks (28 days) of DSD data collected during the Maintenance Period.

### 6.6. GENERAL ASPECTS FOR STATISTICAL ANALYSIS

### 6.6.1. General Methods

All statistical analyses will be performed using SAS statistical software (Version 9.4 or later).

Part 1 summaries will be presented by treatment group (Placebo, 2X008 0.2 mg/kg/day, ZX008 0.8 mg/kg/day).

Continuous data will be summarized using descriptive statistics including means, standard deviations, medians, lower and upper quartiles, minimum and maximum values. Categorical variables will be summarized with frequencies and percentages. Confidence intervals will be calculated for key parameters or estimates as warranted.

Two-sided statistical significance testing ( $\alpha$ = 0.05) comparing each active treatment to placebo will be performed for the primary and secondary endpoints as described below, unless otherwise noted.

All relevant collected subject data will be included in listings. All subjects entered into the database will be included in data listings.

Unless otherwise specified in the subsequent sections, in the event of multiple assessments at a given planned time point, the latest collected value will be used for the summarization.

### 6.6.2. Definitions

<u>First Dose Date</u>: First Dose Date of Investigational Drug: If the first diary date on the day after randomization indicates that investigational drug was taken on this day, then the first dose date (Study Day 1) will be the date after randomization. In all other situations where it is known that the subject took at least one dose of medication, the first dose date will be assumed to be 1 day after the date of randomization.

<u>Study Day:</u> Study day will be calculated relative to the First Dose Date in the Titration Period. For any date on or after the date of first dose, study day will be calculated as

assessment date - first dose date + 1. For any date prior to the date of first dose, study day will be calculated as assessment date - first dose date. There will be no Study Day 0.

<u>Baseline Value:</u> For non-seizure frequency assessments, the Part 1 baseline value will be the last non-missing assessment collected on or prior to the first date of dosing in Part 1. Unscheduled assessments prior to First Dose Date will be considered for selection of the baseline value. Baseline values for seizure frequency endpoints will be determined from the immediate 28 days prior to study day 1 (ie, the First Dose Date) using methods described below.

### 6.6.3. Missing Data

The term missing date refers to a completely missing date or to an incomplete date/partial date where parts are not available, eg, missing month/day/year.

### Missing Adverse Event Start and End Dates

Missing start and end date will be imputed conservatively, ie, missing values will be imputed in such a way that the duration of the AE is considered with the longest possible duration and such that, whenever the AE may potentially start after first date of study medication, the AE will be handled as a treatment-emergent adverse event (TEAE).

The missing Start date and End date of an AE will be imputed for the purpose of calculating treatment emergent status and assigning events to treatment periods using definitions given in the following table.

| | Adverse event |
|---|---|
| Partial<br>/Missing<br>Start date | Missing day - If adverse event day is missing but month and year is present then impute the 1st of the month unless month is same as month of first dose of study drug in Part 1 then impute first dose date in Part 1. |
| c 3 | Missing day and month - If adverse event day and month are both missing but year is present then impute 1st January unless year is the same as first dose date in Part 1 then impute first dose date in Part 1. |
| inglic | Completely missing - impute first dose date in Part 1 unless the end date suggests it could have started prior to this in which case impute the 1st January of the same year as the end date. |
| 271, 3166, | When imputing a start date, ensure that the new imputed date is sensible ie, is prior to the end date of the AE. |
| Partial<br>/Missing End<br>date | Missing day - If AE end day is missing but month and year are present then impute the last day of the month unless month is same as month of last dose of study drug then impute last dose date. |

Missing day and month - If AE has missing day and month but year is present then impute 31st December unless year is the same as first dose date then impute last dose date.

Completely Missing - need to look at whether the AE is still ongoing before imputing a date and also when it started in relation to study drug. If the ongoing flag is missing then assume that AE is still present (ie, do not impute a date). If the AE has stopped and start date is prior to first dose date then impute the 1st dose date. If the AE started on or after the first dose date then impute the last dose date.

### **Data Handling for Seizure Diaries**

Seizures are recorded in the Daily Seizure Diary (DSD). On each day, subjects are asked a question of whether there is a seizure to report that day. Subjects may either answer "Yes" and continue to complete more details about the seizure, or answer "No, this day has been seizure free". There will be no explicit imputation of intermittent missing data for seizure diaries. Missing DSD data will be handled as follows:

- If no seizures are entered in the DSD and the response to the question, is there a seizure to report that day, is "No, this day has been seizure free" then that day will have the seizure count set to 0.
- If seizures are entered in the DSD and the response to the question, is there a seizure to report that day, is "No this day has been seizure free" the seizures entered in the DSD will supersede the seizure freedom affirmation.
- If no seizures are entered in the DSD and there is no response to the question, is there a seizure to report that day, that day will be considered to have missing diary data.
- If no seizures are entered in the DSD and it is indicated that there were seizures that day, that day will be considered to have missing diary data.

### 6.7. VISIT WINDOWS

The following rules will be used to window data into treatment periods for by-treatment period tabulations. For all by-visit tabulations, the nominal visit as recorded on the electronic Case Report Form (eCRF) will be used.

The following are the definitions for associating dates with the treatment periods of Part 1.

| Baseline Period | The Baseline Period will be the 28 days immediately prior to the date of the Study Day 1. |
|---|---|
| | The Double-Blind Treatment Period start date is the date of first full daily dose (ie, Study Day 1). The Double-Blind |

| Titration Period | Treatment Period end date is the last date the subject was on study treatment in Part 1. The Double-Blind Treatment Period consists of 16 weeks from first treatment start date, which includes 2 weeks of Titration Period, 12 weeks of Maintenance Period and 2 weeks of Taper/Transition Period. The end date for efficacy analyses is the last day of Maintenance treatment or Visit 12; the end date for safety analyses is the last day of Taper/Transition, which would be considered the date at Visit 15. For subjects who discontinue early from the study, the Double-Blind Treatment Period end date for efficacy analyses will be the date at the Early Termination Visit (Visit 12); the end date for safety analyses would be the date of Visit 13. If a taper is not conducted, the end date for both analyses would be Visit 12. The Titration Period begins on the first full day of treatment (Study Day 1) and extends through Visit 6 (when the subject has reached their randomization dose). The Titration Period applies to all subjects including placebo recipients. If a subject withdraws from the study prior to treatment in the | Ori Zation |
|---|---|---|
| Maintenance<br>Period | Maintenance Period, all safety assessments and events up to and including the date of study withdrawal will be tabulated in the Titration Period. The Maintenance Period covers the 12 weeks following the end of the Titration Period. It begins on the date of Visit 6 + 1 day and extends through the End of Study/Early Termination Visit (Visit 12). | |
| Titration + Maintenance Period (T+M) | The T+M Period combines the Titration and Maintenance periods, beginning on the date of first treatment (Study Day 1) and extending through the End of Study/End of Treatment Visit (Visit 12). | |
| Taper/Transition<br>Period | The Taper/Transition Period consists of 2 weeks starting from End of Study/Early Termination Visit (Visit 12) + 1 day through Visit 13 (Taper) or Visit 15 (Transition to Part 2). For subjects who are not entering into the Part 2 of the study, subjects will gradually be tapered off of study medication. For subjects who are entering Part 2, subjects will enter the Transition Period where all subjects will be on a dose of ZX008 0.2 mg/kg/day at the end of this period. | |

### 6.8. POOLING OF CENTERS

Analysis will be pooled by cohort (A vs. B).

### 6.9. SUBGROUPS

The following subgroups may be utilized for some efficacy analyses and/or AE summarizations:

Age: 2- < 6 years, 6-< 12 years, 12 - < 18, 2-<18 years,  $\geq$  18 - 35 years

Sex: Male, Female

Baseline Weight: < 37.5 kg vs. ≥ 37.5 kg

Number of Concomitant Antiepileptic Medications Used:  $\leq 2$ , 3,  $\geq 4$  medications

Number of Prior Antiepileptic Medications Used: 0-3, 4-6, 7-9, ≥ 10 medications

Baseline Frequency of Seizures that Result in Drops (events/28 days): based on observed tertiles

Usage of a specific concomitant medication(s) (top 3 concomitant AEDs to be determined by data review) (Yes / No)

# 7. DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION

### 7.1. SUBJECT DISPOSITION AND WITHDRAWALS

The Part 1 subject disposition will be presented per treatment group and overall for Cohort A and B independently.

For describing the Part 1 subject disposition, the following will be summarized by number and percentage:

- Subjects enrolled (only overall)
- Subjects enrolled but not randomized (ie, screen failures) and reason for notrandomized (only overall)
- Subjects randomized
- Number of randomized subjects discontinued the trial per trial period (overall Double-Blind Treatment Period, Titration Period, Maintenance Period, Taper/Transition Period).
- Reasons for discontinuation
- Part 1 completers
  - Completers continuing into Part 2
  - Completers who discontinued prior to Visit 12

Part 1 trial completers include: 1.) subjects who did not discontinue prior to the Visit 12, and 2.) subjects who completed at least through Visit 8 and enrolled into the Part 2 open label extension.

For subjects enrolled but not randomized to treatment in Part 1, and for the tallies listed under each reason for not being randomized, the denominator used to calculate the percentage will be the number of enrolled subjects. For all other calculations in the Part 1 disposition table, the denominator will be the number of subjects randomized.

All subject disposition data will be listed using the Enrolled Population and sorted by randomized treatment and site.

The number and percentage of subjects in the following populations will be summarized by treatment group and overall for Cohort A and B independently:

- Enrolled Population
- Randomized (Intent-to-Treat) Population
- mITT Population
- PP Population
- SAF Population

Allocation to each analysis population will be presented by subject in a listing, by Cohort A and B.

### 7.2. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Part 1 subject demographics and baseline characteristics will be summarized descriptively per treatment group and overall, for the SAF and mITT Populations for Cohort A and B.

The following demographic characteristics will be summarized:

- Age [Years]
- Categorized age as: 2 < 6 years, ≥ 6 < 12 years; ≥ 12 < 18 years, 2 < 18 years, ≥ 18 35 years</li>
- Sex
- Race
- Ethnicity
- Height [m]
- Weight [kg]
- BMI [kg/m²]

• Geography: (Cohort A) North America, Europe, Australia; (Cohort B) Japan only All subject demographics data will be listed for the Enrolled Population, by Cohort A and B.

For Cohort B, a summary table will be added for the mITT Population that will summarize the number and percentage of subjects who experienced at least one seizure event of each type during the baseline period. For the seizure types that are typical drop seizures, the number and percentage of subjects where that seizure type was or was not classified as ESC confirmed drop seizures will be summarized.

# 7.3. MEDICAL HISTORY, NEUROLOGIC HISTORY, AND CONCOMITANT DISEASES

Medical history and neurologic history will be summarized and sorted alphabetically, by primary System Organ Class (SOC) and Preferred Term (PT) coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 or later. The number and percentage of subjects will be displayed for each SOC and PT within treatment group.

Medical history will be presented for the SAF population, separated by Cohort A and B.

All medical history data of subjects will be listed for the Enrolled Population, by Cohort A and B.

### 7.4. MEDICATION

Medication (collected on the prior antiepileptic medications, prior medications, and concomitant medications eCRF page) will be coded using the World Health Organization Drug Dictionary (WHO-DD) Format B3 Version Sep 2017 or later.

The following algorithm will be used to define prior and concomitant in Part 1.

Prior medications will be those with a stop date prior to first dose of study drug administration in Part 1. Summaries of prior medications only include medications that stopped during the period from 30 days prior to the screening date to the day before first date of study treatment.

Concomitant medications in Part 1 will be defined as those medications that were initiated after first study drug administration in Part 1 (but excluding medications that started on or after the first dose of study medication in Part 2) or those medications that were ongoing at the date of first study drug administration in Part 1.

The medication will be assumed to be prior medication if it cannot be definitively shown that the medication did not start or continue during the Part 1 treatment period.

If the start date or stop date of a medication is partially missing, the date will be compared as far as possible with the date of the start of administration of study drug. The following approach will be taken:

• If the start date of medication is complete and occurs on or after the day of the first full dose, the medication will be assumed concomitant. If the start date
occurs prior to the first full dose date but the end date is on or after the first dose date or the medication is recorded as ongoing, the medication will be considered concomitant.

- If the start day is missing but the start month and year are complete, a medication will only be excluded as being concomitant if the start month/year is before the month/year of study drug administration and if the stop date (either full date, month and year if missing day, or year if missing month and day) is before study drug administration.
- If the start day and month are missing but the start year is complete, a
  medication will only be excluded as concomitant if the start year is before the
  year of study drug administration and if the stop date (either full date, month
  and year if missing day, or year if missing month and day) is before study drug
  administration.
- If the start date is completely missing and the stop date is prior to first dose or completely missing, the medication will be assumed to be a prior medication.

A medication may be counted as concomitant in Part 1 and in Part 2. By definition, a prior medication cannot be counted as concomitant in Part 1. Medication will be summarized and sorted alphabetically separately for prior and concomitant medication by Anatomical Therapeutic Chemical (ATC) categories (Level 2: pharmacological or therapeutic subgroup and Level 3: chemical or therapeutic or pharmacological subgroup) and WHO-DD drug code. For each medication, the number and percentage of subjects will be displayed by treatment group and overall.

Part 1 medication summary tables will be presented for the SAF Population.

Prior and concomitant medications/treatments will be listed for the Enrolled Population.

### 7.4.1. Prior and Concomitant Antiepileptic Treatments

Medication (collected on the prior antiepileptic medications, prior medications, and concomitant medications eCRF page) will be coded using the World Health Organization Drug Dictionary (WHO-DD) Format B3 Version Sep 2017 or later. Antiepileptic medications will be identified using any drug entered on the prior-antiepileptic medication page and anti-seizure concomitant medications with indication of "Lennox-Gastaut Syndrome," that have an ATC2 level of 'Antiepileptics'. Medications with a frequency of use specified as "as needed" (PRN) are excluded from the prior and concomitant antiepileptic treatments. Usages of Valproate (all forms) will be summarized on the prior and concomitant antiepileptic medications tables. Subjects may have used multiple forms of the medication. The following preferred names will be summarized into a combined term called "Valproate (all forms)"

- Valproate Magnesium
- Valproate Semisodium

- Valproate Sodium
- Valproate Sodium; Valproic Acid
- Valproic Acid

Prior and concomitant antiepileptic medications will be defined and analyzed for the SAF Population similar to concomitant medications as described in Section 7.4. In addition, the number of prior antiepileptic medications and the number of concomitant antiepileptic medications will be summarized using descriptive statistics and presented by treatment group and overall. Only prior medications that stopped during the period from 30 days prior to the screening date to the day before first date of study treatment will be summarized.

Prior and concomitant antiepileptic treatments will be listed for the Enrolled Population.

Note that further summaries of rescue medications recorded on the daily medication diary are described in the efficacy section.

#### 8. EFFICACY

The analysis of the Part 1 primary and secondary efficacy parameters will be performed on the mITT Population for Cohort A and B independently.

The Part 1 primary efficacy endpoint and key secondary efficacy endpoint analyses will be repeated on the PP Population for Cohort A and B independently, in order to assess the impact of major protocol deviations on the key inference.

All primary and key secondary variables will be analyzed for data obtained for the T+M Period and will be repeated for data obtained during the M Period only.

### 8.1. MULTIPLICITY STRATEGY AND TESTING HIERARCHY

The Part 1, Cohort A efficacy analyses will employ a serial gatekeeper strategy to maintain the Type 1 error rate at a=0.05 across the family of analyses that support the primary and key secondary objectives. The strategy specifies a hierarchy of significance tests where each test acts as a gatekeeper to the tests below it.

Note that the serial gatekeeper strategy does not apply to Part 1 Cohort B since, as noted in the protocol, the relatively small sample size of Cohort B is expected to afford only a descriptive assessment of study endpoints in Cohort B.

The hierarchy starts with the primary analysis comparing ZX008 0.8 mg/kg/day to placebo on the change in number of seizures that results in drops from baseline. The next steps in the hierarchy entail the comparisons for the key secondary endpoints.

• Change from baseline in frequency of seizures that result in drops in T+M in the ZX008 0.2 mg/kg/day group compared to placebo.

- Proportion of subjects who achieve a ≥50% reduction from baseline in the frequency of seizures that result in drops in the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo.
- Proportion of subjects who achieve improvement (minimally, much, or very much improved) in the CGI-I as assessed by the Principal Investigator comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo.

Below is a complete list of steps in the testing hierarchy in order:

- 1. Compare ZX008 0.8 mg/kg/day to placebo on the change in frequency in seizures that result in drops per 28 days between the Baseline and T+M periods.
- 2. Compare ZX008 0.8 mg/kg/day to placebo on the proportion of subjects who achieve a  $\geq$  50% reduction from baseline in the number of seizures that result in drops.
- 3. Compare ZX008 0.8 mg/kg/day to placebo on the CGI-I at Visit 12.
- 4. Compare ZX008 0.2 mg/kg/day to placebo on the change in frequency in seizures that result in drops per 28 days between the Baseline and T+M periods.
- 5. Compare ZX008 0.2 mg/kg/day to placebo on the proportion of subjects who achieve a  $\geq$  50% reduction from baseline in the number of seizures that result in drops.
- 6. Compare ZX008 0.2 mg/kg/day to placebo on the CGI-I at Visit 12

### 8.2. PRIMARY EFFICACY ENDPOINT AND ANALYSIS

### 8.2.1. Primary Efficacy Endpoint Definition

The Part 1 primary efficacy endpoint is the percentage change from Baseline in the frequency in seizures that result in drops per 28 days in the T+M Period. The following seizure types from the DSD will be included in the frequency count of seizures resulting in drops, if for an individual subject, the seizure as listed in the eCRF has been confirmed and approved by the ESC as a 'drop seizure':

- AS
- TS
- TA
- GTO
- SGTC

For each subject, the frequency of drop seizures will be calculated from all available data collected during the Baseline and T+M Periods. Subjects in the ZX008 0.8 mg/kg/day treatment group will be compared to those in the placebo group on the DSF) during T+M adjusted for the frequency during Baseline using a non-parametric ANCOVA model.

The Baseline Period is the 28 days immediately preceding the date of Study Day 1. The T+M Period is planned for 14 weeks. However, actual durations will be computed for each subject based on the individual subject's start and stop dates for each period, except that if the Baseline Period is longer than 28 days, the frequency for the Baseline Period will be calculated with data from the 28 days immediately preceding the Study Day 1.

The frequency of drop seizures will be counted from the DSD records provided by the subject or parent/caregiver.

Responses to the DSD question about the frequency of seizure episodes will be handled differently according to the following response options.

| Response | Number of seizures |
|---|---|
| No seizures | 0 |
| A single seizure | 1 |
| An episode of many discrete seizures | Based on the response to the Question 12 for frequency of episodes |
| A cluster of seizures back-to-back | This will be determined empirically dependent on the duration of the cluster event and the number of events reported in a discrete seizure event for subjects in the study. |

#### **Seizure Clusters**

Seizure clusters are entered in the DSD by estimating the duration of the cluster in hours: minutes; seconds. For seizure clusters the number of discrete seizures that occurred during a cluster is not entered in the DSD. In order to estimate the number of seizures during a cluster, the number of seizures will be imputed using the seizure count and duration of seizures recorded for "an episode of many discrete seizures".

Specifically, episodes of discrete seizures include both an estimate of the number of seizures, and an estimate of the duration, categorized into 1 of 3 buckets: < 2 minutes; 2-10 minutes.

Study-level summary statistics using seizure events reported in the T+M Period will be calculated for each bucket to determine the median number of seizures occurring in each bucket.

The median number of seizures will then be used to impute counts for seizure clusters:

• 'short' clusters (ie, ≤ 59 minutes) will be the median number of seizures reported in discrete seizure events < 2 minutes

- 'medium' clusters (ie, 1-5 hours) will be the median number of seizures reported in discrete seizure events 2-10 minutes
- 'long' clusters (ie, > 5 hours) will be the median number of seizures reported in discrete seizure events > 10 minutes.

#### **Sensitivity Analysis of Cluster Imputation**

A sensitivity analysis using an alternative method for imputing the count associated with cluster events was described in the Part 1 SAP Note to File (NTF) document dated 31Jun2021. This analysis will be completed for Cohort A and Cohort B.

This analysis is an alternative method for imputation of the number of seizure events associated with episodes that were described in the diary as "A cluster of seizures backto-back." The "A cluster of seizure back-to-back" episodes did not have a number of seizure events associated with it. In order to associate a number of seizure events with it, the following alternative method for imputation was defined.

- 1.) Cluster episodes described in the diary as "A cluster of seizures back-to-back" were classified according to duration, as in the primary analysis.
  - Short: < 1 hour duration</li>
  - Medium: 1 5 hours, inclusive
  - Long: > 5 hours
- 2.) Seizure cluster episodes described as "An episode of many discrete seizures" that occurred during the Titration or Maintenance Period of Part 1 were identified, as in the primary analysis. These episodes were reported in the diary with information about the number of discrete seizures in the cluster episode and the duration of a single discrete seizure within the cluster episode.
- 3.) The duration of a single seizure within the discrete seizure cluster episode was defined as:
  - 2 minutes, if the duration of the discrete seizure was answered as "Less than 2 minutes"
  - 10 minutes, if the duration of the discrete seizure was answered as "2 10 minutes"
  - 15 minutes, if the duration of the discrete seizure was answered as "More than 10 minutes"
- 4.) The total duration of the overall discrete seizure cluster episode was calculated as the duration from step 3 multiplied by the number of seizures reported in the discrete seizure cluster episode.
- 5.) The total duration from step 4 was categorized into categories as:

• Short: ≤ 59 minutes

Medium: 60 minutes - 300 minutes (ie, 1 - 5 hours, inclusive)

• Long: > 300 minutes

6.) The median number of seizures reported within a discrete seizure cluster episode was determined for all discrete cluster episodes in the Short, Medium, and Long discrete cluster duration categories in the population. The median value was then imputed into the Short, Medium, and Long duration back-to-back cluster categories.

The frequency of drop seizures was then determined using the alternative cluster event imputation. The same summary statistics, nonparametric model, and parametric models as used for the primary endpoint were used for the cluster event sensitivity analysis.

#### Calculation of seizure frequency / 28 days

For any individual subject, the frequency of drop seizures per 28 days during the baseline period (DSF $_B$ ) will be derived as follows:

 $DSF_B = \frac{28 \times Total \ number \ of \ drop \ seizures \ during \ the \ Baseline \ Period}{Total \ number \ of \ days \ in \ the \ Baseline \ Period \ with \ nonmissing \ diary \ data}$ 

For each treatment group, the median and mean DSF will be calculated.

Similarly, for each subject, the frequency of DSF per 28 days for the T+M period (DSF<sub>T+M</sub>) is derived as below:

$$DSF_{T+M} = \frac{28 \times Total \ number \ of \ drop \ seizures \ during \ the \ T+M \ Period}{Total \ number \ of \ days \ in \ the \ T+M \ Period \ with \ nonmissing \ diary \ data}$$

The percentage change from baseline for any individual subject will be estimated by  $PCDSF_{T+M} = (DSF_{T+M} - DSF_B)*100/DSF_B$ 

The difference from baseline (CDSF<sub>T+M</sub>) will be estimated by CDSF<sub>T+M</sub> = DSF<sub>T+M</sub> – DSF<sub>B</sub>.

For each treatment group, descriptive statistics for DSF during baseline, T+M and M only, as well as the differences and % changes from baseline, will include the number of observations, mean, standard deviation, median, minimum and maximum, overall.

#### 8.2.2. Part 1 Primary Efficacy Endpoint Analyses

#### T+M Period:

The primary analysis will compare the ZX008 0.8 mg/kg/day group to the placebo group for Cohort A using a two-sided test at the  $\alpha$ =0.05 level of significance. The same comparison will be done for Cohort B but will be considered descriptive.

The primary endpoint will be analyzed using a non-parametric analysis of covariance (ANCOVA) model with treatment group (three levels; Placebo, ZX008 0.2 mg/kg/day, ZX008 0.8 mg/kg/day) and weight strata group (< 37.5 kg,  $\geq$  37.5 kg) as factors, rank of baseline DSF<sub>B</sub> as a covariate and rank of percentage CDSF<sub>T+M</sub> as response. Treatment group mean differences from placebo will be estimated via least squares means from the analysis model along with 95% confidence intervals (CIs). Note that the treatment difference estimated from the model is based on rank-transformed data; thus, it cannot be interpreted as an estimate of the size of the difference between groups in percentage CDSF. Instead, the size of the difference between groups in percentage CDSF will be estimated using the Hodges-Lehmann method, described in Section 8.2.3.

The null hypothesis

```
H_0: \mu_{Z_{0.8}} - \mu_P = 0,
```

will be tested against the alternative

$$H_A$$
:  $\mu_{Z0.8} - \mu_P \neq 0$ ,

where  $\mu_{Z0.8}$  and  $\mu_P$  represent the ZX008 0.8 mg/kg and Placebo group location parameter, respectively.

Rejection of the null hypothesis in favor of the alternative, in the presence of a statistically significantly smaller seizure frequency for the treatment group compared to the placebo group, (two-sided p-value <.05) will be regarded as evidence of a treatment benefit in favor of the ZX008 0.8 mg/kg group. A similar comparison of the location parameter for ZX008 0.2 mg/kg/day vs. placebo will be regarded as evidence of a treatment benefit of the ZX008 0.2 mg/kg group. This is the 3rd key secondary endpoint.

Sample SAS code for the non-parametric ANCOVA described above is as follows:

```
Proc rank data=temp ties=mean out=ranktemp;
Var bsrd csrd;
Rank r_bsrd r_csrd;
Run;
proc glm data=ranktemp;
class wtgrp trtp;
model r_csrd = r_bsrd wtgrp trtp / SS3;
lsmeans trtp / pdiff stderr;
```

where trtp = randomized treatment group (with codes 1, 2, 3 indicating placebo, ZX008 0.2 mg/kg, and ZX008 0.8 mg/kg groups).

```
r_bsrd = rank of baseline DSF_B,
r_csrd = rank of percentage CDSF_{T+M}
wtgrp = weight group.
```

Additional statements may be used to obtain estimates and associated 95% Cls.

This document is confidential.

SAP Text Version 3.0 04-Feb-2022 Controlled Document ID: **3903A.02**, Effective Date 31-Aug-2020 Filing requirements: TMF A second analysis of the primary endpoint will be completed using a parametric analysis of covariance (ANCOVA) model with treatment group (three levels; Placebo, ZX008 0.2 mg/kg/day, ZX008 0.8 mg/kg/day) and weight group (<37.5 kg,  $\geq$ 37.5 kg) as factors, log baseline DSF<sub>B</sub> as a covariate and log (CDSF<sub>T+M</sub> +1) as response. Treatment group mean differences from placebo will be estimated via least squares means from the analysis model along with 95% CIs. Since the least square means and confidence intervals will be on the log scale, these least square means and CIs will be exponentiated back to the original scale.

The null hypothesis

$$H_0$$
:  $m_{Z_{0.8}} - m_P = 0$ ,

will be tested against the alternative

$$H_A: m_{Z_{0.8}} - m_P \neq 0$$
,

where  $m_{Z0.8}$  and  $m_P$  represent the ZX008 0.8 mg/kg and Placebo group means (on the log scale), respectively.

Sample SAS code for the parametric ANCOVA described above is as follows:

```
proc glm data=temp;
    class wtgrp trtp;
    model cdsf = bdsf wtgrp trtp / SS3;
    lsmeans trtp / pdiff stderr;
```

where trtp = randomized treatment group (with codes 1, 2, 3 indicating placebo, ZX008 0.2 mg/kg, and ZX008 0.8 mg/kg groups).

```
bdsf = log(DSF_B +1),
cdsf = log(DSF_{T+M} +1)
wtgrp = weight group.
```

Additional statements may be used to obtain estimates and associated 95% confidence intervals. Endpoints of the CIs will be translated to the original scale using the ranks.

#### M Period only:

The primary endpoint analysis described above will be repeated using data from the Maintenance period only as response. For subjects who did not reach the Maintenance period, their Transition period data will be used to represent their M period data.

Similar non-parametric and parametric ANCOVA models will be used.

#### Treatment by baseline seizure category interaction:

Treatment by baseline seizure category interaction: The non-parametric and parametric analysis for the T+M and M period described above will be repeated with baseline seizure frequency as a categorical variable, rather than a covariate, and will include

baseline seizure frequency by treatment interaction. Baseline seizure frequency per 28 days will be categorized using tertiles.

#### 8.2.3. Sensitivity Analyses of Part 1 Primary Efficacy Endpoint

#### Wilcoxon Rank-sum Test

The ZX008 0.8 mg/kg/day group will be compared to the placebo group on the percentage change from baseline in seizures resulting in drops using a Wilcoxon rank sum test. The median difference between the groups, and its 95% CI, will be estimated using the Hodges-Lehmann estimator.

#### Impact of Antiepileptic Drugs (AED)

Subjects in the study are required to be on stable background therapy. Using the mITT population, an additional nonparametric ANCOVA analysis will be performed to assess the impact on the primary analysis of changes in dose or type of concomitant AED, which are protocol violations that may occur during the course of the study.

For this analysis, each subject will be classified according to the number of concomitant AEDs used during the T+M period. Fisher's exact tests will be used to compare the ZX008 dose groups with the placebo group on the percentage of subjects within each group who have a change in concomitant AEDs.

#### Per Protocol Analysis

The primary efficacy ANCOVA will be repeated on the PP Population (which excludes subjects with important protocol deviations that may affect the inference on efficacy such as a change in dose or type of concomitant AED).

### No Imputation for Seizure Clusters

The primary efficacy ANCOVA will be repeated on the mITT Population with no imputation for seizure clusters; ie, seizure clusters will not be calculated in the frequency of seizures that result in drops.

### **Exclusion of Outliers**

The distribution of the primary endpoint is inherently asymmetric since no subject can have more than a 100% decrease in seizures, but there is no reason a subject couldn't have a 200% or even 1000% increase. In fact, there is no theoretical upper bound to the possible magnitude of an increase in a percentage change statistic. To assess the sensitivity of the primary analysis to extreme outliers in percentage change in drop seizure frequency, the primary analysis will be repeated excluding any PCDSF value that satisfies Tukey's criterion for a "far out" outlier (Tukey 1977). Specifically, any PCDSF value that satisfies

$$[\hat{q}_{.25} - 3(\hat{q}_{.75} - \hat{q}_{.25}), \qquad \hat{q}_{.75} + 3(\hat{q}_{.75} - \hat{q}_{.25})]$$

will be excluded where  $\hat{q}_{.25}$  and  $\hat{q}_{.75}$  are the sample lower and upper quartiles of all PCDSF data combined.

#### Imputation for Dropouts

Two different methods for imputation of missing values due to subject drop out will be incorporated into the analysis of the primary efficacy endpoint. When referring to frequency in the paragraphs below, it refers to the number of seizure events per 28 days. The imputation for dropouts may be omitted if fewer than 5% of subjects drop out prior to Visit 12.

S1: Worst value substituted: In this analysis, for a subject who drops out of treatment, if the DSF during T+M is lower than the baseline value, the baseline value will be substituted for the subject from the point of withdrawal to the end of the planned duration of T+M. However, if the seizure frequency during T+M is higher than the baseline value, there will be no substitution. The DSF for the planned duration of T+M will then be computed as a weighted mean of the value before dropout, and the imputed value after dropout. The weights will be the proportion of planned duration of T+M before and after dropout. The statistical analysis (nonparametric ANCOVA) described at the start of Section 8.2.2will then be performed on the resulting dataset. Treatment comparisons will be based on the least squares means and standard errors obtained from the ANCOVA.

S2: Differential imputation method: In this analysis, subjects who drop out due to an AE, lack of compliance, loss to follow-up or subject choice will have their DSF for the remainder of the time during the planned T+M period replaced with the worse of the observed value or the baseline value as described for S1. However, for other withdrawal reasons (e.g., "lack of efficacy") their observed DSF during T+M will be imputed for the remainder of the time between dropout and end of planned T+M. The DSF for the planned duration of T+M will then be computed as a weighted mean of the value before dropout and the imputed value after dropout. The weights will be the proportion of time before and after dropout. The statistical analysis (nonparametric ANCOVA) described at the start of Section 8.2.2will then be performed on the resulting dataset. Treatment comparisons will be based on the least squares means and standard errors obtained from the ANCOVA.

#### Pre-Data Change Request (DCR) Analyses

The following posthoc analyses of the DSF for Cohort A were described in the Part 1 SAP NTF dated 31Jun2021.

A pre-edited version of the seizure datasets for Cohort A was requested for regulatory submissions, intended to represent the original instance of data prior to modifications made as a result of cleaning for Part 1 Cohort A database lock. Upon sponsor request, Syneos Health created 2 versions of pre-edited ("pre-DCR") datasets that were used as sensitivity analyses. The changes made in the DSD data are described below:

 Pre-DCR 2) any edits made through the Trial Manager portal or directly on the device itself were removed

 Pre-DCR 3) any edits made through the Trial Manager portal or directly on the device itself were removed, with the exception of the seizure classification field (this field is not subject-reported and is subject to review/query/approval by the ESC)

Using the different versions of the pre-DCR seizure dataset, the seizure frequency rates were reproduced with each set. The following sensitivity analyses of seizures that result in drops were completed using these sets.

- Summary statistics for observed rate, change from baseline, and percentage change from baseline in rate for the T+M period, M period, up to 2 weeks, up to 6 weeks, up to 10 weeks, and up to 14 weeks. This analysis was completed for the mITT Population
- Summary statistics for observed rate, change from baseline, and percentage change from baseline in rate for the T+M period, M period, up to 2 weeks, up to 6 weeks, up to 10 weeks, and up to 14 weeks using the cluster sensitivity values. This analysis was completed for the mITT Population.
- Nonparametric analysis for the T+M period and M period using the original values and alternative cluster imputation method. This analysis was completed for the mITT Population.
- Imputation methods for dropouts described in Section 8.2.3of the Part 1 SAP
- Wilcoxon rank-sum test, including Hodges-Lehmann confidence interval for differences from placebo, described in Section 8.2.3
- The number and percentage of subjects who had a worsening or no change, 0% reduction, ≥25% reduction, ≥50% reduction, ≥75% reduction, 100% reduction in seizure frequency, and near seizure freedom (ie, 0 or 1 seizures) between Baseline and T+M and between Baseline and M.
- Cumulative response curve for percentage of subjects experiencing various % reductions in seizures (mITT Population)
- Summary statistics for observed rate, change from baseline, and percentage change from baseline in rate for the T+M and M period by individual seizure type. This analysis was completed for the mITT Population
- The number and percentage of subjects who had a worsening or no change, > 0% reduction, ≥ 25% reduction, ≥ 50% reduction, ≥ 75% reduction, 100% reduction in seizure frequency, and near seizure freedom by individual seizure type between Baseline and T+M and between Baseline and M

For Cohort B, the need for pre-DCR analyses will be determined based on regulatory interactions, and any analyses to be performed will be detailed separately.

#### ESC Confirmed Drop Seizures - Sensitivity to the Supplementary Drop Seizure File

This document is confidential.

SAP Text Version 3.0 04-Feb-2022 Controlled Document ID: **3903A.02**, Effective Date 31-Aug-2020 Filing requirements: TMF After the Part 1 Cohort A database lock occurred, an updated version of the supplementary drop seizure file for Cohort A, which lists each seizure type per subject that was reconciled to be an ESC-confirmed drop seizure, was provided that contained corrections to the reconciliation based on findings discovered after database lock. The updated file was used to create a new version of the frequencies of ESC-confirmed drop seizures, and the same analyses used for the primary analyses of ESC-confirmed drop seizures were applied to this data.

#### Criteria for Establishing Efficacy

While several supportive and/or supplementary analyses are specified above, the main criterion for demonstrating efficacy will be the primary non-parametric analysis for the mITT population from Cohort A.

#### KEY SECONDARY EFFICACY ENDPOINTS AND ANALYSES 8.3.

#### 50% Reduction in Seizures Resulting in Drops 8.3.1.

The first key secondary endpoint compares treatment groups on the percentage of subjects with at least a 50% reduction from baseline in seizures resulting in drops. That is, the percentage of subjects in the ZX008 0.8 mg/kg/day group who have a decrease in frequency of seizures resulting in drops of at least 50 percentage points will be compared to the analogous percentage in the placebo group. This the 1st key secondary efficacy endpoint.

The comparison of the percentage of subjects with at least a 50% decrease in DSF from baseline between treatment groups will be made using a logistic regression model that incorporates the factors treatment and weight strata and the baseline seizure frequency. Separate models will be fit for ZX008 0.2 mg/kg/day vs. placebo and ZX008 0.8 mg/kg/day vs. placebo. Achievement of the 50 percentage point reduction or greater (yes or no) will be modeled as a function of treatment group (2 levels; ZX008 0.8 mg/kg/day (or ZX008 0.2 mg/kg/day) and placebo) and baseline weight strata group (< 37.5 kg, ≥ 37.5 kg). If the model with treatment and weight strata is not convergent (eg, due to a 0 count in a treatment by weight strata combination, the model will be refit using treatment only and the baseline seizure frequency. If the model still does not converge, no odds ratio and p-value from the logistic regression will be reported.

The model estimated odds ratio (including a 95% CI) and p-value for comparison of ZX008 0.8 mg/kg/day to placebo and ZX008 0.2 mg/kg/day to placebo will be provided. A supplementary Fisher's exact test comparing treatment groups will be provided.

Similarly, the number and percentage of subjects who have a worsening or no change, ≥ 0% reduction, ≥ 25% reduction, ≥ 50% reduction, ≥ 75% reduction, 100% reduction in seizure frequency and near seizure-freedom will be tabulated for each treatment. Near seizure-freedom will be defined as having 0 or 1 seizures leading to a drop in the T+M

period. These are additional secondary endpoints. For Cohort B, an additional exploratory analysis of the number and percentage of subjects who have a > 25% worsening from baseline will be included. This had been added by Zogenix as a posthoc analysis in the report of Cohort A results.

For the Pre-DCR datasets for Cohort A, the following sensitivity analyses of the change in seizures that result in drops were added.

The number and percentage of subjects who had a worsening or no change, 0% reduction, ≥ 25% reduction, ≥ 50% reduction, ≥ 75% reduction, 100% reduction, and near seizure freedom in the frequency of each individual seizure type between Baseline and T+M and between Baseline and M will be summarized by treatment group. This analysis was completed for the mITT Population.

# 8.3.2. Clinical Global Impression - Improvement (CGI-I) Rating, as assessed by the Principal Investigator

The Principal Investigator will rate their global impression of the subject's condition at each clinic visit after randomization: at the end of the Titration period Visit 6 (Day 15), during the Maintenance period at Visit 8 (Day 43) and Visit 10 (Day 71), and at Visit 12 (End of Study / Early Termination).

The CGI-I scale measures the change in the subject's clinical status from a specific point in time, i.e., the Baseline Period. The CGI-I rating scale permits a global evaluation of the subject's improvement over time. The severity of a subject's condition is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows:

1=very much improved
2=much improved
3=minimally improved
4= no change
5=minimally worse
6=much worse
7=very much worse

Descriptive statistics for the CGI-I score, and the number and percentage of subjects who showed improvement (i.e., had a score of 3 or lower) will be presented for each for each treatment group at each assessment time point. Each assessment time point will include a comparison of the percentage of subjects with improvement between each ZX008 group and the placebo group using the Cochran-Mantel-Haenszel test (CMH) stratified by weight strata, and also a frequency distribution of the number and percentage of subjects rated in each category in the scale. A graphic showing the percentage of subjects rated in each category will be presented.

The number and percentage of subjects who showed clinically meaningful improvement (ie, had a score of 2 or lower) and a comparison of the percentage of subjects with clinically meaningful improvement between each ZX008 group and the placebo group

will be presented for each treatment group at each assessment time point as an exploratory analysis.

Individual subject CGI-I data will be listed.

#### 8.4. ADDITIONAL EFFICACY ENDPOINTS AND ANALYSES

#### 8.4.1. Countable Motor Seizures Definition and Analysis

The change in the frequency of countable motor seizures per 28 days between the Baseline and T+M periods will be calculated using the same methodology described for the primary endpoint. Countable motor seizures include:

- GTC
- SGTC
- TS
- AS
- TA
- clonic seizures [CS]
- hemiclonic seizures [HS]
- focal seizures [FS] with clear observable motor signs

The change in the frequency of countable motor seizures per 28 days between the Baseline and M period will also be calculated.

The same non-parametric and parametric ANCOVA models described for the primary endpoint will be used for the analyses of countable motor seizures (change in the frequency between Baseline and T+M periods). The mITT Population will be used for this analysis. The difference between ZX008 0.8 mg/kg/day and placebo in the change between Baseline and T+M is a secondary endpoint. The analyses will be repeated for the change in frequency between the Baseline and M periods. The analysis of the change between Baseline and the M period is one of the additional secondary endpoints.

The number and percentage of subjects who had a worsening or no change, 0% reduction,  $\ge 25\%$  reduction,  $\ge 50\%$  reduction,  $\ge 75\%$  reduction, and 100% reduction in the frequency of countable motor seizures between Baseline and T+M and between Baseline and M will be summarized by treatment group and overall. For Cohort B, the number and percentage of subjects who had a > 25% worsening will be determined. Except for the latter, which is exploratory, these analyses are part of the additional secondary endpoints.

#### 8.4.2. Additional Seizure Counts

The other efficacy endpoints of change in the frequency per 28 days between Baseline and T+M Period and between Baseline and M Period of:

- Seizures that Typically Result in Drops (i.e., GTC, SGTC, TS, AS, TA regardless of whether ESC confirmed as drop or not)
- All Countable Non-Motor Seizures
- All Countable Seizures
- All Countable Seizures That Did Not Result in Drops (ESC Confirmed) Added as
  posthoc analysis for Cohort A. It will also be included in the analysis of Cohort B.

Each of these endpoints will be calculated using the same method as the primary endpoint. The same non-parametric ANCOVA, parametric ANCOVA, and logistic regressions used for the primary efficacy endpoint will be used. The mITT Population and PP Populations will be used for these analyses.

Refer to Appendix 1 for the seizure types that are included in each of these endpoints.

#### Pre-DCR Sensitivity Analyses of Seizures that Typically Result in Drops

Analyses of Typical Drop Seizure endpoints for Cohort A, Part 1 using the Pre-DCR versions of the dataset were added and described in the Part 1 SAP NTF dated 31Jun2021. The following summaries were included. For Cohort B, the need for pre-DCR analyses will be determined based on regulatory interactions, and any analyses to be performed will be detailed separately.

- Summary statistics for observed rate, change from baseline, and percentage change from baseline in rate for the T+M period, M period, up to 2 weeks, up to 6 weeks, up to 10 weeks, and up to 14 weeks. This analysis was completed for the mITT Population.
- Summary statistics for observed rate, change from baseline, and percentage change from baseline in rate for the T+M period, M period, up to 2 weeks, up to 6 weeks, up to 10 weeks, and up to 14 weeks using the cluster sensitivity values. This analysis was completed for the mITT Population.
- Nonparametric analysis for the T+M period and M period using the original values and alternative cluster imputation method. This analysis was completed for the mITT Population
- Wilcoxon rank-sum test, including Hodges-Lehmann confidence interval for differences from Placebo, described in section 8.2.3 of the Part 1 SAP
- The number and percentage of subjects who had a worsening or no change, 0% reduction, ≥ 25% reduction, ≥ 50% reduction, ≥ 75% reduction, 100% reduction in seizure frequency, and near seizure freedom (ie, 0 or 1 seizures) between Baseline and T+M and between Baseline and M. This analysis is completed for the mITT Population.

- Cumulative response curve for percentage of subjects experiencing various % reductions in seizures (mITT Population)
- Summary statistics for observed rate, change from baseline, and percentage change from baseline in rate for the T+M and M period by individual seizure type. This analysis was completed for the mITT Population
- The number and percentage of subjects who had a worsening or no change, 0% reduction,  $\geq 25\%$  reduction,  $\geq 50\%$  reduction,  $\geq 75\%$  reduction, 100% reduction, and near seizure freedom in the frequency of each individual seizure type between Baseline and T+M and between Baseline and M will be summarized by treatment group. This analysis is completed for the mITT Population.

#### All Countable Seizures That Did Not Result in Drops (ESC Confirmed)

The SAP v2.0 08Jan2020 described increasingly broad groupings of seizure types for efficacy analyses, from the primary endpoint (drop seizures only) to all countable (motor + non-motor) seizures; however, it did not describe a seizure grouping that does not include drop seizures as defined for the primary endpoint. The calculation of the change in the frequency of all countable seizures that did not result in drops (ESC confirmed; ie, non-drop seizures) between Baseline and the T+M Period and M Period will be completed similarly to the method described for the primary endpoint. All countable seizures recorded from the diary that did not meet the criteria of drop seizures as defined in the primary endpoint analysis, ie, are CS, HS, FS with or without observable signs, myoclonic, absence/atypical absence, infantile spasms, epileptic spasms, other, or are seizures of the following classifications that were approved for each subject as non-drop seizure types by the ESC: GTC, SGTC, TS, AS, or TA seizures, will be included. The analysis of this parameter will also be included in the analysis of Part 1, Cohort B. In addition, the number and percentage of subjects who had a worsening or no change, 0% reduction,  $\geq$  25% reduction,  $\geq$  50% reduction,  $\geq$  75% reduction, 100% reduction in frequency and near seizure freedom for non-drop seizures between Baseline and T+M and between Baseline and M will be summarized. For Cohort B, the number and percentage of subjects who had a > 25% worsening will also be determined.

#### 8.4.3. Seizure-Free Days

Seizure-free days will be taken from the DSD data.

A seizure-free day with no seizures leading to drops will be defined as a day for which diary data are available and with no ESC-confirmed drop seizures. A day without countable motor seizures will be defined as a day for which diary data are available and with no countable motor seizures. The total number of drop seizure-free days and countable motor seizure-free days will be summarized for the entire T+M period and similarly for the Baseline Period.

Seizure-free days per 28 days at baseline = (number of seizure free days during baseline)\*28/ (number of days during baseline with non-missing diary data)

Seizure-free days per 28 days during T+M Period = (number of seizure free days during T+M Period)\*28/ (number of days during T+M Period with non-missing diary data)

Statistical comparison of the ZX008 groups and placebo group on the number of drop seizure-free days per 28 days and countable motor seizure-free days per 28 days during T+M using the baseline as covariate will be done with a similar non-parametric ANCOVA model as described for the primary analysis.

### 8.4.4. Duration of the Longest Interval Between Seizures Resulting in Drops

The duration of the longest interval between seizures resulting in drops (in days) will be analyzed using nonparametric methods.

For each subject, the duration of the longest interval between seizures resulting in drops (ie, ESC confirmed) will be calculated over the entire T+M period. This will be derived as the maximum of the number of consecutive days between seizures resulting in drops. The length of the intervals between seizures resulting in drops will be calculated as below, after which the duration of the longest interval between convulsive seizures will be derived.

If a subject has a missing diary day within an otherwise seizure-free interval, that day is counted towards the duration of the seizure free interval. However, if a subject has two consecutive days of missing diary data, the current seizure-free interval will end on the first date of missing diary data, and a new one begun on the next date that diary data are available, and no seizure occurs. [In that case, for purpose of calculation of this variable, all intervening days, after the 2nd day, with missing diary data, will be assumed to have a seizure with drops occurrence, until the first available date with non-missing diary data.]

Let Date0 (=Day1) be the first day of treatment. If a seizure resulting in a drop occurs on five days having dates as Date1, Date2, Date3, Date4, and Date5, where Date5>Date4>Date3>Date2>Date1≥Date0, and let LDT = Last date of treatment in the maintenance period, where LDT ≥ Date5, then the time interval between convulsive seizures will be calculated as follows:

11=Date2 - Date1

12=Date3 - Date2

l3=Date4 - Date3,

14=Date5 - Date4.

For completeness, we calculate the time to the first seizure as

10=Date1 - Date0,

and the time from the last seizure to end of treatment as

15 = LDT - Date5.

Here the duration of the longest interval =Maximum (10, 11, 12, 13, 14, 15).

If the subject does not experience a seizure during treatment, then the last available diary date will be used to compute the duration of the longest interval as follows:

The longest interval=last available diary date - Date0

The median time of the longest interval between seizures resulting in drops (in days) will be presented. Additional summary statistics will be presented, including mean, minimum, maximum, and the 25th and 75th percentiles, 95% CIs on the difference in medians between groups (Hodges-Lehman estimator).

The Wilcoxon rank sum test will be used to test for differences between each ZX008 group and the placebo group, and the p-value from this test will be presented. A boxplot summarizing the duration of the longest interval between seizures will be provided.

# 8.4.5. Clinical Global Impression - Improvement Rating, as assessed by the Parent/Caregiver

CGI-I ratings assessed by the parent/caregiver will be summarized and analyzed using the same methods used for CGI-I ratings recorded by the Principal Investigator as above.

#### 8.4.6. Incidence of Status Epilepticus

The incidence of SE will be evaluated based on: 1.) seizures entered as serious adverse events (SAEs), and 2.) seizures lasting longer than 10 minutes from the DSD. A single seizure meeting more than one of these criteria will be counted once.

The number and percentage of subjects with SE during the Baseline and T+M Periods recorded as an AE will be presented by treatment group. Statistical comparisons of the difference in incidence will be tested using a Fisher's Exact Test.

From the diary data, change from Baseline in the number of seizures with duration > 10 minutes per 28 days for the T+M Period will be reported. A nonparametric ANCOVA will be completed to compare ZX008 groups vs. placebo. As well, the number of unique days where SE was reported (normalized per 28 days) will be summarized and analyzed using the nonparametric ANCOVA.

All seizures recorded in the AE database as SE should also be included in the DSD. An edit check will be performed to identify the overlap between seizures identified as AE

of SE and seizures entered into the diary as seizures > 10 min. The "calculated" number and percentage of subjects experiencing SE will be presented by treatment group, defined as individuals who experience either an AE of SE, medical treatment for SE, or a seizure lasting longer than 10 minutes. Each subject will be represented once regardless of incidence. Statistical comparisons of the differences in incidence between treatment and placebo groups will be based on Fisher's exact test.

A second calculation will present the number of incidences of SE, according to the above definition, by treatment group normalized to per 28 days. In this analysis, a single subject may have more than one episode of SE, but an episode of SE recorded as both an AE and as a seizure longer than 10 minutes will be counted as a single episode. Statistical comparisons of the differences between treatment and placebo groups will be based on a Fisher's Exact Test. A difference in percentages between baseline and the T+M period will be calculated and summarized within each treatment group.

#### Sensitivity Analysis of Status Epilepticus

The following analysis was added as a posthoc analysis for Cohort A, Part 1. This was included in the Part 1 SAP NTF dated 31Jun2021. This analysis will be completed for Cohort B.

A sensitivity analysis of SE cases determined from the DSD was conducted, based on seizure types officially recognized as SE by the International League Against Epilepsy (ILAE). Seizure events with duration > 10 minutes that were of one of the following types were identified.

- Absence/atypical absence
- Focal with clear observable motor signs
- Focal without clear observable motor signs
- GTC
- SGTC

Such events were further divided in order of increasing risk/emergency, ie, into those events that required

- No Rescue Medications
- 1 Rescue Medications
- > 1 Rescue Medications

The number of events of each type was counted in the Baseline Period, T+M Period, and M Period as well as the rate (events/ 28 days) was determined. The number of subjects with at least one event was summarized and the incidence rate between the ZX008 groups and the placebo group was compared using a Fisher's Exact Test.

#### 8.4.7. Rescue Medication Usage

Use of rescue medication is recorded on the daily diary. In the event of prolonged seizures or SE, rescue medication is administered according to each subject's personalized regimen consisting of one or more medications. If the first rescue administration does not control the seizures, a second or even third round might be administered. The second and third round might use different medications or different doses than the first round of rescue medications.

Rescue medication will be summarized by treatment group and comparisons of ZX008 treatment vs. placebo performed for the following:

- The number of days rescue medication was taken (normalized to 28 days) will be summarized separately for the Baseline and T+M periods by the mean (SD) as well as the median, minimum and maximum values. Multiple medications taken on the same day will be counted once for that day. The ZX008 groups will be compared to the placebo group using a non-parametric ANCOVA analogous to that described in the primary efficacy endpoint section. Specifically, the rank ANCOVA will use the ranks of rescue medication frequency during T+M or M period as the response and will incorporate treatment group as a factor and the ranks of rescue medication frequency during Baseline as a covariate.
- The number of medications used per episode will be summarized using similar descriptive statistics as above. Rescue medications related to an episode of SE are considered to be all rescue administered on the day of the SE (or seizure lasting >10 min). If more than one episode of SE or a seizure lasting >10 min occurred in a single day, the rescue medication for that episode is all rescue administered after the seizure until the start time of the next prolonged seizure.

#### 8.4.8. Incidence of Medical Services to Treat Seizures

Data on hospitalization and healthcare resource use to treat seizures will be captured in the CRF and will be used to calculate incidence.

Details of the hospitalizations, including reasons for hospitalization and use of resources during the study will be summarized.

#### 8.4.9. Vineland Adaptive Behavior Scale (VABS)

The VABS is a parent/caregiver completed assessment that looks at the personal and social skills of individuals from birth through adulthood (Sparrow, S. S. & Cicchetti, D. V. (1989)). Because adaptive behavior refers to an individual's typical performance of the day-to-day activities required for personal and social sufficiency, these scales assess what a person actually does, rather than what he or she is able to do. The VABS assesses adaptive behavior in 4 domains:

- Communication
- Daily living skills
- Socialization

## Motor skills

In Part 1, the VABS is collected at Visit 3 (Randomization), Visit 8 (Day 43), and Visit 12 (End of Study/Early Termination).

As noted in the Part 1 SAP NTF dated 21Jun2021, the Vineland Adaptive Behavior Scale data was not analyzed due to issues with the collection on the eDiary device. The questionnaire was not administered in a way that allowed for determination of the domain scores.

### 8.4.10. Quality of Life in Childhood Epilepsy (QOLCE) Scale

The parent/caregiver will complete the QOLCE. This assessment looks at how epilepsy affects day-to-day functioning of their child in various life areas, including physical activities, well-being, cognition, social activities, behavior and general health (Sabaz et al., 2000; Talarska 2007). There is also one question on overall quality of life, administered as part of the QOLCE.

The QOLCE is collected at Visit 3 (Randomization) and at Visit 12 (End of Study/Early Termination).

The QOLCE scores items with a possible 5-point response. To calculate subscale scores, the 5-point item scores will first be reverse coded as necessary so that scores of 5 represent the best possible response and 1 represents the worst possible response. [Details of the reverse coding are provided in the shells for the TLFs]. Item scores will then be transformed to a 0-100 scale as follows: 1 -> 0, 2 -> 25, 3 -> 50, 4 -> 75, 5 -> 100. After transformation, a score for each subject for each subscale is calculated by averaging that subject's responses to each item in the subscale. A value of 0 represents the lowest or poorest score and 100 reflects the highest level of functioning. The 16 subscale scores per subject are then averaged to obtain an overall quality of life score for each subject.

Summary descriptive statistics including the n, mean, standard deviation, median, minimum, and maximum will be generated for the index score at each scheduled collection time point.

A higher subscale and overall quality of life score indicate a better response.

Table 6: Subscale of QOLCE:

| Domain | Subscale | Item |
|-----------------------|-------------------------|---------------------|
| Section 3: Physical | Physical Restrictions | 3.1 a-j |
| Section 3: Physical | Energy/Fatigue | 3.2 a,b |
| Section 4: Well-being | Depression | 4.1 a,d,e,l |
| Section 4: Well-being | Anxiety | 4.1 b,g,j,n,o,p |
| Section 4: Well-being | Control/helplessness | 4.1 c,f,h,i |
| Section 4: Well-being | Self-esteem | 4.1 k,m,q,r,s |
| Section 5: Cognition | Attention/Concentration | 5.1 a,d,e,f,g |
| Section 5: Cognition | Memory | 5.1 j,k,l,m,n,o |
| Section 5: Cognition | Language | 5.1 p,q,r,s,t,u,v,w |

| Section 5: Cognition | Other Cognitive | 5.1 b,c,h |
|---|---|---|
| Section 6: Social Activities | Social Interactions | 6.1 c,f,h |
| Section 6: Social Activities | Social Activities | 6.1 a, e, 6.2 |
| Section 6: Social Activities | Stigma Item | 6.1 i |
| Section 7: Behavior | Behavior | 7.1 a, |
| | | c,f,g,h,i,j,k,l,m,o,q,r,s,t |
| Section 8: General Health | General Health | 8.1 |
| Section 2 (USA Version) or | Quality of Life Item | 2.1 or 9.1 |
| Section 9 (Australia Version): | | , KI |
| Quality of Life | | |
| Overall Quality of Life * | | Average of 16 subscale scores* |

<sup>\*</sup>An Overall Quality of Life Score will be computed by adding each subscale score for each individual and then dividing by 16.

For each treatment group and at each schedule visit, the descriptive statistics will be presented for each QOLCE subscale and for the overall quality of life score.

In addition, the change from baseline in the overall QOLCE will be calculated for each subject by subtracting the Part 1 baseline score from the score measured at each scheduled postbaseline visit. The change from baseline for each treatment group will be summarized by summary statistics. Treatment groups will be compared using pairwise Wilcoxon Rank-sum tests.

Individual subject data for the domains will be listed.

## 8.4.11. Zarit Caregiver Burden Inventory





Patient/Caregiver Assessment using HADS Scale 8.4.12.





#### 8.4.13. **New Seizure Types**

The analysis of New Seizure Types was added in the Part 1 SAP NTF dated 31Jun2021.

In Cohort A, a posthoc analysis of the emergence of new seizure types was to be pase are types c of study transpect's unique sold from the following performed. The summary of this variable will be based on the Seizure History eCRF (a form that lists both previous and current seizure types experienced by each subject), seizures reported on the DSD prior the start of study treatment, and seizures reported during the T+M Period of Part 1. Each subject's unique seizure types experienced prior to study treatment will be determined from the following types:

#### **Seizure Types**

**GTC** 

**SGTC** 

TS

AS

TA

CS

**HS L Body** 

HS R Body

HS with Independent L and R

FS with clear observable signs

FS without clear observable signs

Myoclonic

Absence/atypical absence

Infantile Spasms

**Epileptic Spasms** 

Other

Subjects with emergence of at least one new seizure type during the T+M Period will be summarized by randomized treatment group. A new seizure type is defined as a seizure type recorded in the DSD that was not recorded in the Seizure History eCRF as occurring before the first study drug dose date and that also did not occur during the Baseline Period.

#### 9. SAFETY

All Part 1 safety analyses will be performed for the SAF Population, as defined in Section 6.2. Results will be reported by treatment group for the 16-week treatment period, unless noted otherwise.

#### 9.1. **EXTENT OF EXPOSURE**

Part 1 treatment exposure data will be summarized for the SAF Population.

Duration of total exposure during Part 1 (ie, time on treatment (in days)) will be calculated per subject as the number of days with IMP intake during the trial and will be summarized using n, mean, standard error, median, minimum,  $Q_1$ ,  $Q_3$  and maximum.

This will be calculated as:

Date of last IMP intake in Part 1 - Date of first full daily IMP intake in Part 1 + 1

Time on treatment will be summarized by the Part 1 treatment group.

#### TREATMENT COMPLIANCE (DIARY) 9.2.

Study medication is to be administered twice daily, and self-reported compliance is recorded in the daily diary as full (both doses), partial (less than full daily dose) or missed (both doses) each day. From this, compliance will be calculated by assuming that a missed dose = 0% of dose consumed, partial =50% of dose consumed, and full = 100% of dose consumed. For each subject, a daily diary compliance score will be thus obtained.

Compliance will also be determined based on the actual quantity taken, determined using the weight of the dispensed drug kit and weight of the returned drug kit. The expected quantity taken will be determined using the assigned dosage in mg/kg/day and the number of days they were assigned at that dosage. If a kit was not returned, the compliance for the period will be missing.

For Part 1, compliance will be summarized for the SAF and mITT Populations over the course of T+M period and M period only per recorded visit dates, reported by treatment group.

#### 9.3. ADVERSE EVENTS

An AE is defined as any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. For Part 1, the period of observation for AEs extends from the time the subject gives informed consent until the end of the Titration/Transition Period (Visit 13 or 15).

A TEAE in Part 1 is defined as any AE that based on start date information occurs after the first intake of study treatment in Part 1, but not on or after the first dose of study treatment in Part 2. For subjects who participate in Part 2, the Part 1 TEAE will include events with onset up to the day prior to the date of first dosing in Part 2. A Part 1 TEAE will be further classified into the Titration Period, Maintenance Period, and Transition/Taper Period. The Titration Period will include all events with onset from the date of the first dose in Part 1 to date of the Visit 6. The Maintenance Period will include all events with onset from the day after Visit 6 through the date of Visit 12. The Transition/Taper Period will include all events with onset starting with the day after Visit 12 through Visit 15.

For Part 1, tables will present TEAE data by assigned treatment group received in Part 1. AEs occurring after enrollment and prior to the first administration of study treatment in Part 1 are defined as non-treatment emergent AEs (non-TEAEs).

AEs are categorized by the Investigator as related or unrelated to study drug. If the AE is thought to be definitely, probably or possibly related to study drug then it is to be categorized as related. Possibly or definitely unrelated is categorized as unrelated. Any TEAE with missing relationship will be considered as "related."

The severity of AEs (for both non-serious and serious AEs) will be assessed by the Investigator as follows:

### Severity Definition of Adverse Events:

Mild - A type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living.

Moderate - A type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant.

Severe - A type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.

Any AE with missing severity will be imputed as "severe."

The original terms used by the investigators in the eCRFs to identify AEs will be coded using the MedDRA Version 20.1 or later.

#### 9.3.1. Overview of Adverse Events

ating authorization as the street of the str For Cohort A and B, separately, the number and percentage of subjects with at least one of the following events will be summarized in an overall summary table:

- **TEAE**
- Treatment-related TEAE
- Treatment-emergent SAE
- Treatment-related treatment-emergent SAE
- Severe TEAEs
- Severe treatment-related TEAE
- Adverse events of special interest
- TEAEs leading to premature discontinuation of study treatment
- TEAEs leading to premature discontinuation from the study
- Death

This overall summary table will be presented for the full Part 1 period, Titration Period, Maintenance Period, Titration + Maintenance Period, and Taper/Transition Period.

For the full Part 1 period, Titration Period, and Titration + Maintenance Period, the denominator for the calculation of percentage will be the number of subjects in the SAF Population for the treatment group. For the Maintenance Period, the denominator for the calculation of the percentage will be the number of subjects for the treatment group with Part 1 last dose strictly greater than the date of Visit 6. For the Taper/Transition Period, the denominator for the calculation of the percentage will be the number of subjects for the treatment group with last dose strictly greater than the date of Visit 12.

#### **Treatment-Emergent Adverse Events** 9.3.2.

For Cohort A and B, separately, the following summaries will display the number and percentage of subjects with an adverse event as well as the corresponding number of events by SOC and PT (sorted alphabetically):

- All TEAEs
- Treatment-emergent SAEs
- TEAEs by Maximum Severity
- Study Drug-Related TEAEs
- All TEAEs leading to premature discontinuation from the study

These summaries will present the TEAEs presented for the full Part 1 period, Titration Period, Maintenance Period, T+M Period, and Taper/Transition Period.

Summaries of TEAEs and study drug-related TEAEs will be summarized for the following subgroups:

- Age: 2- < 6 years (Cohort A only), 6-< 12 years (Cohort A only), 12 < 18 (Cohort A only), 2 < 18 years (Cohort B only) ≥ 18 35 years (Cohort A and B)</li>
- Sex (Cohort A only)
- Concomitant usage of most commonly used concomitant antiepileptic medications (eg, valproate or other medications of interest; to be determined)
- Number of concomitant AEDs (Cohort A only)

An additional summary table will summarize the number and percentage of subjects in each treatment group who experience an AE that occurs in at least 5% in Cohort A (at least 10% of subjects for Cohort B) of subjects in any treatment group. For AEs occurring in at least 5% of subjects in Cohort A (at least 10% of subjects for Cohort B), another table will present the mean and median time to onset and the median duration of the onset. The summaries will be presented by preferred term in decreasing order of incidence. For subjects who have multiple occurrences of the same event during the study, the first event will be used in the summary. For unresolved events, the duration will be calculated using the last date of follow-up in Part 1.

Another summary of the most commonly occurring adverse events ( $\geq$  10% incidence overall or in any treatment group) in Part 1 will be provided by treatment group, first showing the number of subjects, number of events (noting that a subject may have multiple occurrences of the same event), and the number of resolved events.

No inferential statistical methods (ie, methods that yield p-values) will be used to compare treatment groups on the frequency or severity of AEs.

The following listings will be produced for all enrolled subjects:

- All AEs; events considered to be TEAEs will be identified in the listing
- SAEs
- AEs that lead to premature discontinuation from the study
- Deaths

### 9.3.3. Adverse Events of Special Interest (AESI)

As per International Conference on Harmonisation (ICH) guidance (E2F Development Safety Update Report [2011]), the sponsor has identified the following AESIs for the study:

Table 7 - Adverse Events of Special Interest:

#### Metabolic/Endocrine

- 1. Elevated prolactin level  $\ge 2x$  above the upper limit of normal (ULN)

ror Part 1 AEs, the AESIs will be identified on the eCRF.
For Part 1, AESIs will be summarized by treatment group and by SOC and PT.
All AESIs will be listed separately.

9.4. PHYSICAL EXAMINATION

A complete physical examination will be performed at Visit 1 (Screen Randomization) prior to first dose of study medication study/Early Termination). An abbreviated 5), Visit 8 (Day 43), and Vicin 1 and be performed at Visit 8 (Day 43), and Vicin 1 and be performed at Visit 8 (Day 43), and Vicin 1 and be performed at Visit 9 (Day 43). may be performed at the Cardiac follow-up visit for subjects who do not enter the open-label extension study if clinically warranted. Clinically significant findings at screening will be reported on the medical history page. New clinically significant findings starting with after the first dose in Part 1 will be reported as AEs.

A summary of subjects with clinically significant physical examination findings at each visit will be provided for the T+M Period.

All physical examination results will be presented in a subject data listing.

#### 9.5. **NEUROLOGIC EXAMINATION**

In Part 1, a complete neurological examination will be performed at Visit 1 (Screening) and Visit 12 (End of Study/Early Termination). An abbreviated neurological examination will be performed at Visit 3 (Randomization) and at Visit 6 (Day 15), Visit 8 (Day 43), and Visit 10 (Day 71). Clinically significant findings at screening will be reported on the medical history page. New clinically significant findings starting with after the first dose in Part 1 will be reported as adverse events.

A summary of subjects with clinically significant neurologic examination findings at each visit will be provided for the T+M Period.

All neurological examination results will be presented in a subject data listing.

#### VITAL SIGNS, WEIGHT, AND BMI

Vital signs and weight and BMI data will be documented for subjects at Visit 1 (Screening), Visit 3 (Randomization) prior to first dose of study medication, at the end of the Titration Period at Visit 6 (Day 15), during the Maintenance Period at Visit 8 (Day 43) and Visit 10 (Day 71), and at Visit 12 (End of Study/Early Termination). The

measurements will include blood pressure, heart rate, temperature, respiratory rate, weight, and BMI.

For each vital sign and weight and BMI, observed values and change from baseline to each on-study evaluation will be summarized.

For weight, the occurrence of at least a  $\geq 7\%$  gain/reduction or  $\geq 10\%$  gain/reduction from baseline will be summarized by visit and at any time during the T+M Period. For subjects with an occurrence of a  $\geq 7\%$  reduction in weight, the number who achieved a recovery to their baseline weight, the duration of time to recovery, and whether that recovery was achieved as a result of a reduction or withdrawal of the subject's study medication, will be summarized. Recovery will be defined as achieving a weight after the  $\geq 7\%$  reduction, that is at least 99% of the baseline weight and having a weight at Visit 12 that is at least 99% of the baseline weight. The number of days until weight recovery will be determined using the date of the first date when the weight loss was observed and the first date when the subject's weight had recovered to, and maintained for the duration of the study period, at least 99% of the baseline weight. For Cohort B, the summary will also be presented by subgroups of subjects 2 to < 18 and  $\geq$  18 years of age.

For subjects with at least a 7% reduction in body weight, a spaghetti plot showing the subject's weight values by study day will be presented by actual treatment group. For Cohort B, the plot will also be presented by subgroups of subjects 2 to < 18 and  $\geq$  18 years of age.

Vital signs, weight, height, and BMI data will be presented in a data listing. In addition, change and percentage change from baseline in weight and BMI will be presented in a data listing.

For each subject with a clinically meaningful abnormality in vital signs (to be supplied by Zogenix International), a listing will be produced organized by parameter that lists each subject, age, sex, day of most abnormal value, and the most abnormal value. The listing will also include subjects with at least a 7% reduction in weight or clinically meaningful abnormality in BMI.

#### 9.7. ELECTROCARDIOGRAM

Analysis of ECGs will be included in a separate report from ERT (formerly Biomedical Systems).

#### 9.8. DOPPLER ECHOCARDIOGRAPHY

Results of ECHOs will be presented in a separate report from ERT (formerly Biomedical Systems).

### 9.9. TANNER STAGING

In Part 1, Tanner Staging will be assessed for subjects > 7 to 18 years old during the study at Visit 3 (Randomization) and Visit 12 (End of Study/Early Termination).

Conceptually, pubertal maturation can be described in terms of sequence, timing, and tempo. Puberty consists of a series of predictable events, and the sequence of changes in secondary sexual characteristics has been categorized by several groups. The onset and progress of pubertal changes will be recorded on a 5-point scale for boys and girls separately. Boys are rated for genital development and pubic hair growth through stage I to stage V. Girls are rated for breast development and pubic hair growth through stage I to stage V.

The number and percentage of subjects in each Tanner Stage will be presented for all visits by treatment group separately for boys and girls overall and broken out for the following age groups:

- > 7 years to ≤11 years
- > 11 years to  $\leq$  15 years
- > 15 years to ≤ 18 years

All Tanner staging data will be presented in the subject data listing

#### 9.10. LABORATORY PARAMETERS

Laboratory safety parameters will be analyzed by a central laboratory using standard validated methods.

All laboratory safety data will be collected as per the schedule of assessments given in Table 4

The following continuous laboratory parameters will be analyzed:

- Hematology: hemoglobin, hematocrit, erythrocytes, erythrocyte mean corpuscular volume, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets
- Blood Biochemistry: albumin (ALB), alkaline phosphatase (AP), alanine aminotransferase (ALT; SGPT), aspartate aminotransferase (AST; SGOT), blood urea nitrogen (BUN), calcium (Ca), carbon dioxide (CO2), chloride (Cl), creatinine, creatine kinase, gamma-glutamyl transferase (GGT), globulin, glucose, lactate dehydrogenase (LDH), phosphorus, potassium (K), sodium (Na), thyroid function, thyroid stimulating hormone (TSH), total bilirubin, direct bilirubin, total cholesterol, total protein, triglycerides, uric acid.
- Tests of growth and precocious puberty: Growth hormone (GH), insulin-like growth factor-1 (IGF-1, low sensitivity), prolactin, Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH), testosterone, estradiol
- Coagulation: Prothrombin time, International normalized ratio (INR), activated partial thromboplastin time (PTT)
- Whole blood cannabidiol
- Urinalysis: analysis for pH, glucose, ketones, nitrite, protein, bilirubin, urobilinogen, leukocyte esterase, and occult blood. Microscopic analysis will be performed for blood, all cell types, and casts.

- Pregnancy test: Urine or serum pregnancy testing will be performed in female subjects of childbearing potential.
- Urine or serum THC panel

Observed continuous laboratory data will be descriptively summarized by type of laboratory test/parameter change from baseline. For Cohort B, tests of growth and precocious puberty will be summarized by age groups and/or sex groups.

Categorical laboratory parameters will be summarized by presenting the number and % of subjects by visit and by treatment arm.

For each laboratory parameter for which upper or low limits of normal are defined, shift tables will be created comparing the baseline status with the status at each postbaseline visit. Status will be classified as:

- below lower limit of normal and clinically significant
- below lower limit of normal,
- within normal limits,
- above upper limit of normal,
- above upper limit of normal and clinically significant.

Listings of the most extreme values for a subject recorded during Part 1 will be created for each parameter for which normal limits are defined. These will show the lowest recorded value and the highest recorded value noted for the subject. A listing of subjects with markedly abnormal laboratory results will be provided, and additional explorations of the data may be conducted as warranted.

Additionally, summaries of abnormal lab results by parameter will be provided to investigate changes in platelet count and prolactin in detail. The summaries include:

- Subjects with decrease (≥ 25% from baseline) in platelets count with normal platelet count at baseline
- Subjects with decrease (≥ 25% from baseline) in platelets count relative to baseline (whether normal or abnormal) platelet count
- Subjects with decrease (≥ 25% from baseline) in platelets count with normal platelet count at baseline, by valproate use
- Subjects with decrease (≥ 25% from baseline) in platelets count with normal platelet count at baseline, by presence/absence of infection event prior to 7 days of the lab assessment
- Subjects with increase (≥ 25% from baseline) in prolactin with normal baseline

• Subjects with increase (≥ 25% from baseline) in prolactin with normal baseline, and had seizure event within 48 hours prior to prolactin

#### 9.11. COLUMBIA-SUICIDE SEVERITY RATING SCALE

During Part 1, the Columbia-Suicide Severity Rating Scale (C-SSRS) data will be collected at Visit 1 (Screening), at Visit 3 (Randomization), at the end of the Titration Period at Visit 6 (Day 15), during the Maintenance Period at Visit 8 (Day 43) and Visit 10 (Day 71), and at Visit 12 (End of Study/Early Termination).

Subjects who are younger than 7 years of age, or who are judged by the investigator not to have the mental capacity to understand the questions as specified on the C-SSRS, will not complete the rating. The investigator should use his/her judgment to substitute intellectually appropriate questions to probe the tendency for self-harm.

An electronic tablet will be used to collect C-SSRS data and will only ask about a subject's capability to complete C-SSRS during the Baseline visit. If the site records that the subject is incapable of answering the questions, the C-SSRS will be removed from their list of required questionnaires for the remainder of the study.

The following outcomes are C-SSRS categories for and have binary responses (yes/no):



is assessed as a "yes" answer at any time during the T+M Period to any one of the five questions (1-5) above. In Part 1, the number and percentage of subjects with at baseline and the number and the number and percentage of subjects with at least once during the T+M Period will be presented. The denominator will be the number of subjects completing the C-SSRS at least once during the period.

The following outcomes are C-SSRS categories for and have binary responses (yes/no):





# 10. INTERIM ANALYSES

No formal interim analysis is planned for this study. However, the analysis of the Part 1 Cohort A will occur prior to the completion of Part 1 Cohort B. The unblinding of Part 1 Cohort A will not occur until data cleaning is completed and all decisions regarding protocol deviations warranting exclusion from the PP Population have been made for the Cohort A subjects. The review of deviations and exclusion from the PP Population for Cohort B subjects will occur independently. An unblinded team from Zogenix International and Syneos Health will be assigned to complete the unblinding of Part 1 Cohort A. The unblinded team will not participate in any decision-making regarding the Cohort B subjects' Part 1 data. Access to aggregated data (ie, group-level tables or figures) does not constitute unblinding and for the purpose of data cleaning these

subjects will be considered blinded. A separate unblinding plan will be developed to further define this process.

There have been several changes to the Additional Secondary Objectives specified for Part 1 in the protocol, and consequently to the associated Additional Secondary Efficacy Endpoints. These mainly fell into the following categories:

• Addition of new objectives
• Clarification of seizure types involved
• Specification of when seizure types needed ESC confirmation
• Clarification of the treatment period involved.

The following is a list of the Additional Secondary Objectives as specified in the SAP to support the support of the support of the SAP to support the support of the SAP to support the support of the SAP to support the SAP to support the support of the SAP to support the same of the same of the

| Protocol Versions 2.1 and later | Statistical Analysis Plan Version 2.0 | |
|---|---|--|
| To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints: | To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the following endpoints: | |
| PUBLIO | Added: Change in frequency of all seizures that (typically) result in drops (i.e., GTC, SGTC, TS, AS, TA) between baseline and the combined T+M whether ESC confirmed as drop or not. | |
| <ul> <li>Change in the frequency of all countable motor seizures between baseline and T+M (countable seizures include: generalized tonic-clonic seizures [GTC], tonic seizures [TS], clonic seizures [CS], atonic seizures [AS], tonic/atonic seizures [TA], clearly recognizable focal seizures [FS], and myoclonic seizures [MS] that result in a drop)</li> </ul> | <ul> <li>Modified to:</li> <li>Change in the frequency of all countable motor seizures between baseline and T+M (countable seizures include: GTC, SGTC, TS, AS, TA, clonic seizures [CS], focal seizures with clear observable motor signs [FS], and hemiclonic seizures [HS]).</li> </ul> | |
| Change in the frequency of all countable seizures (ie, motor and nonmotor) between baseline and T+M | Change in the frequency of all countable seizures (i.e., motor and non-motor) between baseline and T+M | |
| Change in frequency of seizures that<br>result in drops between baseline and<br>the Maintenance Period (M) | <ul> <li>Modified to:</li> <li>Change in frequency of seizures that result in drops (ESC confirmed) between</li> </ul> | |
| | baseline and the Maintenance Period (M) |
|---|---|
| | Added: |
| | <ul> <li>Change in frequency of seizures that<br/>(typically) result in drops between<br/>baseline and the Maintenance Period<br/>(M)</li> </ul> |
| Change in the frequency of countable | Deleted and replaced with: |
| motor seizures that do not result in drops between baseline and M | Change in the frequency of all countable motor seizures between baseline and M |
| | <ul> <li>Change in the frequency of all<br/>countable non-motor seizures between<br/>baseline and M</li> </ul> |
| | <ul> <li>Change in the frequency of all<br/>countable seizures (i.e., motor and non-<br/>motor) between baseline and M</li> </ul> |
| <ul> <li>The proportion of subjects who have a worsening or no change (ie, ≤ 0% reduction), &gt; 0%, ≥ 25%, ≥ 50%, ≥ 75%, 100% reduction, and "near seizure freedom" (ie, 0 or 1 seizures) between baseline and T+M, and baseline and M, in all countable motor seizures (GTC, TS, AS, TA, FS, MS with a drop); in countable motor seizures that do not result in drops; in all countable seizures; in all countable seizures that do not result in drops; and in all seizures that result in drops</li> </ul> | Modified to: The proportion of subjects who achieve a worsening, > 0 - < 25%, ≥ 25%, ≥ 50%, ≥ 75%, 100% reduction, and "near seizure freedom" (ie, 0 or 1 seizures) between baseline and T+M, and baseline and M, in seizures that result in drops (ESC confirmed), seizures that typically result in drops, all countable motor seizures, all countable non-motor seizures, and all countable seizures |
| Number of seizure-free days, defined as 1) days with no countable seizures and 2) days with no seizures that result in drops | <ul> <li>Modified to:</li> <li>Number of seizure-free days, defined as <ol> <li>no seizures that result in drops (ESC confirmed), and 2) days with no countable motor seizures</li> </ol> </li> </ul> |
| Longest interval between seizures that | Modified to: |
| result in drops | Longest interval between seizures that result in drops (ESC confirmed) |
| To evaluate the effect of ZX008 0.2 and 0.8 mg/kg/day (independently) versus placebo on the Clinical Global | <ul> <li>To evaluate the effect of ZX008 0.2 and<br/>0.8 mg/kg/day (independently) versus<br/>placebo on the Clinical Global</li> </ul> |

| Impression - Improvement rating, as | Impression - Improvement (CGI-I) rating, |
|---|---|
| assessed by the parent/caregiver | as assessed by the parent/caregiver. |

Below is a list of the Additional Secondary Efficacy Endpoints as specified in the protocol:

| Protocol Version 2.1 | Statistical Analysis Plan Version 2.0 |
|---|---|
| <ul> <li>Change from baseline in the frequency of all countable motor seizures in T+M</li></ul> | Added: Change from baseline during T+M in frequency of all seizures that (typically) result in drops (i.e., GTC, SGTC, TS, AS, TA) whether ESC confirmed as drop or not. Modified to: Change from baseline during T+M in frequency of all countable motor seizures (GTC, SGTC, TS, AS, TA, CS, FS, and HS). Modified to: Change from baseline during T+M in the frequency of all countable seizures (i.e., motor and non-motor). Change from baseline during M in the frequency of seizures that result in drops. |
| Change from baseline in the frequency of countable seizures that do not result in drops | Deleted; This was added as a post-hoc analysis for the Part 1 analysis of Cohort A, and will be included in the Part 1 analysis of Cohort B as noted in the SAP version 3.0. Added: Change from baseline during T+M in frequency of all countable non-motor seizures (absence, myoclonic, focal |

| | <ul> <li>without clear observable motor signs, infantile spasms, and epileptic spasms).</li> <li>Change from baseline during M in the frequency of seizures that typically result in drops.</li> </ul> |
|---|---|
| | Change from baseline during M in the frequency of all countable motor seizures. |
| | <ul> <li>Change from baseline during M in the<br/>frequency of all countable non-motor<br/>seizures.</li> </ul> |
| | <ul> <li>Change from baseline during M in the<br/>frequency of all countable seizures<br/>(i.e., motor and non-motor).</li> </ul> |
| Proportion of subjects who achieve a | Modified to: |
| worsening from baseline (ie, ≤ 0% reduction), or >0%, ≥ 25%, ≥ 50%, ≥ 75%, 100% reduction, and "near seizure freedom" (ie, 0 or 1 seizures) between baseline and T+M, and baseline and M, in all countable motor seizures; in countable motor seizures that do not result in drops; in all countable seizures; in all countable seizures that do not result in drops; and in all seizures that result in drops | <ul> <li>Proportion of subjects who achieve a worsening from baseline (ie, ≤ 0% reduction), or &gt; 0%, ≥ 25%, ≥ 50%, ≥ 75%, or 100% reduction between baseline and T+M, and baseline and M, in seizures that result in drops (ESC confirmed), seizures that typically result in drops, all countable motor seizures, all countable non-motor seizures, and all countable seizures.</li> </ul> |
| <ul> <li>Number of seizure-free days in the baseline, M, and T+M period, defined as</li> <li>1) days with no countable seizures and</li> <li>2) days with no seizures that result in drops</li> </ul> | <ul> <li>Modified to:</li> <li>Number of seizure-free days in the baseline, M and T+M period, defined as 1) days with no seizures that results in drops (ESC confirmed), and 2) days with no countable motor seizures</li> </ul> |
| The longest interval (days) between<br>seizures that result in drops comparing<br>the ZX008 0.8 mg/kg/day and 0.2<br>mg/kg/day groups independently versus<br>placebo | <ul> <li>Modified to:</li> <li>The longest interval (days) between seizures that result in drops (ESC confirmed) comparing the ZX008 0.8 mg/kg/day and 0.2 mg/kg/day groups independently versus placebo</li> </ul> |
| <ul> <li>Clinical Global Impression -<br/>Improvement as assessed by the<br/>parent/caregiver</li> </ul> | Clinical Global Impression - Improvement as assessed by the parent/caregiver |

Changes and additions to the analyses described in the Part 1 SAP version 2.0 were described in the Part 1 SAP NTF dated 31Jun2021. They have been added to the Version 3.0 Part 1 SAP.

### 12. PROGRAMMING CONSIDERATIONS

All tables, data listings, figures (TLFs), and statistical analyses will be generated using SAS® for Windows, Release 9.4 (SAS® Institute Inc., Cary, NC, USA). Computergenerated table, listing and figure output will adhere to the following specifications.

#### 12.1. GENERAL CONSIDERATIONS

- One SAS program can create several outputs. / A separate SAS program will be created for each output.
- One output file can contain several outputs. / Each output will be stored in a separate file.
- Output files will be delivered in Word format / pdf format.
- Numbering of TLFs will follow ICH E3 guidance.

# 12.2. TABLE, LISTING, AND FIGURE FORMAT

#### 12.2.1. General

- All TLFs will be produced in landscape format, unless otherwise specified.
- All TLFs will be produced using the Courier New font, size 8
- The data displays for all TLFs will have a minimum 1-inch margin on all 4 sides.
- Headers and footers for figures will be in Courier New font, size 8.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TLFs will be in black and white (no color), unless otherwise specified
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TLFs, unless otherwise specified. On some occasions, superscripts 1, 2, or 3 may be used (see below).
- Only standard keyboard characters will be used in the TLFs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used. Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g., μ). Certain subscripts and superscripts (e.g., cm2, Cmax) will be employed on a case-by-case basis.
- Mixed case will be used for all titles, footnotes, column headers, and programmersupplied formats, as appropriate.

#### 12.2.2. Headers

- All output should have the following header at the top left of each page:
   <Sponsor Name> Protocol XXX (Syneos Health study number xxx)
   Draft/Final Run <date>
- All output should have Page n of N at the top or bottom right corner of each page.
   TLFs should be internally paginated in relation to the total length (i.e., the page
   number should appear sequentially as page n of N, where N is the total number of
   pages in the table).
- The date output was generated should appear along with the program name as a footer on each page.

# 12.2.3. Display Titles

- Each TLF should be identified by the designation and a numeral. (i.e., Table 14.1.1). ICH E3 numbering is strongly recommended but sponsor preferences should be obtained prior to final determination (see also template 03.007C "Table of Contents for Tables Listings and Figures in Statistical Analysis Plan"). A decimal system (x.y and x.y.z) should be used to identify TLFs with related contents. The title is centered. The analysis set should be identified on the line immediately following the title. The title and table designation are single spaced. A solid line spanning the margins will separate the display titles from the
- Column headers. There will be 1 blank tine between the last title and the solid line.

Table x,y,z
First Line of Title
Second Line of Title if Needed
ITT Analysis Set

## 12.2.4. Column Headers

- Column headings should be displayed immediately below the solid line described above in initial upper-case characters.
- In the case of efficacy tables, the variable (or characteristic) column will be on the
  far left-followed by the treatment group columns and total column (if applicable).
   P-values may be presented under the total column or in separate p-value column (if
  applicable). Within-treatment comparisons may have p-values presented in a row
  beneath the summary statistics for that treatment.
- For numeric variables, include "unit" in column or row heading when appropriate.
- Analysis set sizes will be presented for each treatment group in the column heading as (N=xx) (or in the row headings if applicable). This is distinct from the 'n' used for the descriptive statistics representing the number of subjects in the analysis set.

The order of treatments in the tables and listings will be Placebo first in the case of placebo controlled studies and Active comparators first in the case of active comparator trials, followed by a total column (if applicable).

#### Body of the Data Display 12.2.5.

### 12.2.5.1. General Conventions

Data in columns of a table or listing should be formatted as follows:

- alphanumeric values are left-justified;
- numbers in table cells are center aligned.

### 12.2.5.2. Table Conventions

- Units will be included where available
- between t'
  e, even
  num If the categories of a parameter are ordered, then all categories between the maximum and minimum category should be presented in the table, even if n=0 for all treatment groups in a given category that is between the minimum and maximum level for that parameter. For example, the frequency distribution for symptom severity would appear as:

| Severity<br>Rating | N |
|--------------------|---|
| severe C | 0 |
| moderate | 8 |
| mild | 3 |

Where percentages are presented in these tables, zero percentages will not be presented and so any counts of 0 will be presented as 0 and not as 0 (0%).

- If the categories are not ordered (e.g., Medical History, Reasons for Discontinuation from the Study, etc.), then only those categories for which there is at least 1 subject represented in 1 or more groups should be included.
- An Unknown or Missing category should be added to any parameter for which information is not available for 1 or more subjects.
- Unless otherwise specified, the estimated mean and median for a set of values should be printed out to 1 more significant digit than the original values, and standard deviations should be printed out to 2 more significant digits than the original values. The minimum and maximum should report the same significant digits as the original values. For example, for systolic blood pressure:

| N | XX |
|---------|-------|
| Mean | XXX.X |
| Std Dev | X.XX |
| Median | XXX.X |
| Minimum | XXX |

#### Maximum

#### XXX

- P-values should be output in the format: "0.xxxx", where xxxx is the value rounded to 4 decimal places. Any p-value less than 0.0001 will be presented as <0.0001. If the p-value is returned as >0.9999 then present as >0.9999
- Percentage values should be printed to one decimal place, in parentheses with no spaces, one space after the count (e.g., 7 (12.8%), 13 (5.4%)). Unless otherwise noted, for all percentages, the number of subjects in the analysis set for the treatment group who have an observation will be the denominator. Percentages after zero counts should not be displayed and percentages equating to 100% should be presented as 100%, without any decimal places.
- Tabular display of data for medical history, prior / concomitant medications, and all tabular displays of adverse event data should be presented by the body system, treatment class, or SOC, assuming all terms are coded. Within the body system, drug class and SOC, medical history (by preferred term), medications (by preferred name), and adverse events (by preferred term) should be displayed. SOC terms are sorted alphabetically. Preferred tems are sorted in order of incidence within SOC terms.
- The percentage of subjects is normally calculated as a proportion of the number of subjects assessed in the relevant treatment group (or overall) for the analysis set presented. However, careful consideration is required in many instances due to the complicated nature of selecting the denominator, usually the appropriate number of subjects exposed. Describe details of this in footnotes or programming notes.
- For categorical summaries (number and percentage of subjects) where a subject can be included in more than one category, describe in a footnote or programming note if the subject should be included in the summary statistics for all relevant categories or just 1 category and the criteria for selecting the criteria.
  - Where a category with a subheading (such as system organ class) has to be split over more than one page, output the subheading followed by "(cont)" at the top of each subsequent page. The overall summary statistics for the subheading should only be output on the first relevant page.
- For each table, a reference to the source listing(s) will be provided in the footer.

# **Listing Conventions**

- Listings will be sorted for presentation in order of subject num, visit/collection day, and visit/collection time.
- Missing data should be represented on subject listings as either a hyphen ("-") with a corresponding footnote ("- = unknown or not evaluated"), or as "N/A", with the footnote "N/A = not applicable", whichever is appropriate.

- Dates should be printed in SAS® DATE9.format ("ddMMMyyyy": 01JUL2000). Missing portions of dates should be represented on subject listings as dashes (--JUL2000). Dates that are missing because they are not applicable for the subject are output as "N/A", unless otherwise specified.
- All observed time values must be presented using a 24-hour clock HH:MM or HH:MM:SS format (e.g., 11:26:45, or 11:26). Time will only be reported if it was measured as part of the study.
- Units will be included where available

#### 12.2.5.3. Figure Conventions

 Unless otherwise specified, for all figures, study visits will be displayed on the X-axis and endpoint (e.g., treatment mean change from Baseline) values will be displayed on the Y-axis.

#### 12.2.6. Footnotes

- A solid line spanning the margins will separate the body of the data display from the footnotes.
- All footnotes will be left justified with single-line spacing immediately below the solid line underneath the data display.
- Footnotes should always begin with "Note:" if an informational footnote, or 1, 2, 3, etc. if a reference footnote. Each new footnote should start on a new line where possible.
- Subject specific footnotes should be avoided, where possible.
- Footnotes will be used sparingly and must add value to the table, figure, or data listing. If more than six lines of footnotes are planned, then a cover page may be used to display footnotes, and only those essential to comprehension of the data will be repeated on each page.
- The last line of the footnote section will be a standard source line that indicates the name of the program used to produce the data display, date the program was run, and the listing source (i.e., 'Program: myprogram.sas Listing source: 16.x.y.z').

# 13. QUALITY CONTROL

SAS programs are developed to produce output such as analysis data sets, summary tables, data listings, figures or statistical analyses. Syneos Health SOP 03.010 and 03.013 provide an overview of the development of such SAS programs.

Syneos Health SOP 03.009 describes the quality control procedures that are performed for all SAS programs and output. Quality control is defined here as the operational techniques and activities undertaken to verify that the SAS programs produce the output by checking for their logic, efficiency and commenting and by review of the produced output.

This document cannot be used any extensions or validations the real to support any national declination and any extensions or validations to the superior of t

# 14. INDEX OF TABLES, FIGURES, AND LISTINGS

The data analyses from Cohort B subjects in Japan will not be performed during the initial, principal analysis of the trial but will be conducted later. In general, the same analyses that apply to Cohort A subjects in North America, Europe and Australia will be applied to Cohort B subjects in Japan except for those where the smaller sample size in Cohort B makes the analysis untenable. In particular, subset analyses will generally not be applied to Cohort B data.

| Table/<br>Figure/<br>Listing | Number | Description of Modification from Version 2.0 SAP |
|---|---|---|
| | 14.1 | Demographic data and other baseline characteristics |
| | 14.1.1 | Subject disposition |
| Table | 14.1.1.1.1 | Overall Subject Disposition in Part 1 (Cohort A – North America, Europe, Australia) – All Enrolled Subjects |
| Table | 14.1.1.1.2 | Overall Subject Disposition in Part 1 (Cohort B - Japan) – All Enrolled Subjects |
| Table | 14.1.1.2.1 | Major Protocol Deviations in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population |
| Table | 14.1.1.2.2 | Major Protocol Deviations in Part 1 (Cohort B - Japan) – Safety Population |
| Table | 14.1.1.3.1 | Study Populations in Part 1 (Cohort A – North America,<br>Europe, Australia) |
| Table | 14.1.1.3.2 | Study Populations in Part 1 (Cohort B - Japan) |
| | 14.1.2 | Demographic and other baseline characteristics |

| Table/<br>Figure/<br>Listing | Number | Table Header | Description of Modification from Version 2.0 SAP |
|---|---|---|---|
| Table | 14.1.2.1.1 | Demographic and Baseline Characteristics (Cohort A – North America, Europe, Australia) – Safety Population | illos |
| Table | 14.1.2.1.2 | Demographic and Baseline Characteristics (Cohort B - Japan) – Safety Population | |
| Table | 14.1.2.2.1 | Demographic and Baseline Characteristics (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.1.2.2.2 | Demographic and Baseline Characteristics (Cohort B-Japan) – mITT Population | |
| Table | 14.1.2.3.1 | Demographic and Baseline Characteristics by Baseline Weight Stratum (Cohort A – North America, Europe, Australia) – Safety Population | Adhoc Table request |
| Table | 14.1.2.4.1 | Seizure Types Reported on the Seizure Diary During the Baseline Period (Cohort B – Japan) – Safety Population | New Table |
| | 14.1.3 | Medical history | |
| Table | 14.1.3.1.1 | Medical and Neurologic History (Cohort A – North America, Europe, Australia) – Safety Population | Title Change; Neurologic History included in this table. |
| Table | 14.1.3.1.2 | Medical and Neurologic History (Cohort B – Japan) – Safety Population | Title Change; Neurologic History included in this table. |
| | 14.1.4 | Prior and concomitant medication/treatment | |
| Table | 14.1.4.1.1 | Medications and Therapies/Treatments Stopped during or up to 30 Days prior to Screening (Cohort A – North America, Europe, Australia) – Safety Population | Title Changed. Only medications that had stopped during screening or up to and |

|---|---|---|---|
| | | | including 30 days prior to the screening were included. |
| Table | 14.1.4.1.2 | Medications and Therapies/Treatments Stopped during or up to 30 Days prior to Screening (Cohort B – Japan) Safety Population | Title Changed. Only medications that had stopped during screening or up to and including 30 days prior to the screening were included. |
| Table | 14.1.4.2.1 | Concomitant Medications and Therapies/Treatments in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.1.4.2.2 | Concomitant Medications and Therapies/Treatments in Part 1 (Cohort B – Japan) – Safety Population | |
| Table | 14.1.4.3.1 | Prior Antiepileptic Treatment (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.1.4.3.2 | Prior Antiepileptic Treatment (Cohort B – Japan) – Safety<br>Population | |
| Table | 14.1.4.4.1.1 | Concomitant Antiepileptic Treatment in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.1.4.4.1.2 | Concomitant Antiepileptic Treatment in Part 1 (Cohort B – Japan) - Safety Population | |
| Table | 14.1.4.4.2.1 | Rescue Medications in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | Title Change from Concomitant Rescue<br>Medications |

|---|---|---|---|
| Table | 14.1.4.4.2.2 | Rescue Medications in Part 1 (Cohort B – Japan) - Safety Population | Title Change from Concomitant Rescue<br>Medications |
| | 14.1.5 | Treatment Exposure and compliance | 6 |
| Table | 14.1.5.1.1 | Duration of IMP Treatment Exposure in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.1.5.1.2 | Duration of Study Drug Treatment Exposure in Part 1<br>(Cohort B – Japan) – Safety Population | Title Adjustment |
| Table | 14.1.5.2.1.1 | Compliance to IMP intake in Part 1 (Cohort A – North America, Europe, Australia) - mITT Population | |
| Table | 14.1.5.2.1.2 | Compliance to Study Drug Intake in Part 1 (Cohort B – Japan) - mITT Population | Title Adjustment |
| Table | 14.1.5.2.2.1 | Compliance to IMP intake in Part 1 (Cohort A – North America, Europe, Australia) - Safety Population | This table was described in the shells but was not included in the table of contents. |
| Table | 14.1.5.2.2.2 | Compliance to Study Drug Intake in Part 1 (Cohort B – Japan) - Safety Population | This table was described in the shells but was not included in the table of contents. |
| | | | Title Adjustment |
| Table | 14.1.5.2.3.1 | Compliance to IMP Intake in Part 1 based on Bottle Weight (Cohort A – North America, Europe, Australia) - mITT Population | |
| Table | 14.1.5.2.3.2 | Compliance to Study Drug Intake in Part 1 Based on Bottle Weight (Cohort B – Japan) - mITT Population | Title Adjustment |

|---|---|---|---|
| Table | 14.1.5.2.4.1 | Compliance to IMP Intake in Part 1 based on Bottle Weight (Cohort A – North America, Europe, Australia) - Safety Population | This table was described in the shells but was not included in the table of contents. |
| Table | 14.1.5.2.4.2 | Compliance to Study Drug Intake in Part 1 Based on Bottle Weight (Cohort B – Japan) - Safety Population | This table was described in the shells but was not included in the table of contents. Title Adjustment |
| | 14.2 | Efficacy, pharmacokinetics, and pharmacodynamics | |
| | 14.2.1 | Efficacy – ZX008 0.8 and 0.2 mg/kg/day vs Placebo<br>Seizures resulting in drops | |
| Table | 14.2.1.1.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort A. North America, Europe, Australia) – mITT Population | |
| Table | 14.2.1.1.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplementary Seizure File updated post-Part 1 Database Lock. |
| Table | 14.2.1.1.1b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |

|---|---|---|---|
| Table | 14.2.1.1.1.1c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version |
| Table | 14.2.1.1.1.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort B – Japan) – mITT Population | Table number clarified in shells. |
| Table | 14.2.1.1.1.3 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cluster Event Sensitivity Analysis) (Cohort A – North America, Europe, Australia) – mITT Population | Post-hoc table addition. The shell used is the same as 14.2.1.1.1.1. The different methodology of imputing the number of seizure events associated with Cluster events was added. |
| Table | 14.2.1.1.1.3s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cluster Event Sensitivity Analysis) (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplementary Seizure<br>File updated post-Part 1 Database Lock |
| Table | 14.2.1.1.1.4 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cluster Event Sensitivity Analysis) (Cohort B – Japan) – mITT Population | Post-hoc table addition. The shell used is the same as 14.2.1.1.1. The different methodology of imputing the number of seizure events associated with Cluster events was added. |
| Table | 14.2.1.1.2.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics | |

|---|---|---|---|
| | | (Cohort A – North America, Europe, Australia) – PP<br>Population | insere |
| Table | 14.2.1.1.2.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – PP Population | New Table using Supplementary Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.1.2.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort B – Japan) – PP Population | |
| Table | 14.2.1.2.1.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | Table Number Update |
| Table | 14.2.1.2.1.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplementary Seizure<br>File updated post-Part 1 Database Lock |
| Table | 14.2.1.2.1.1b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.2.1.1c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric | New Table using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | | Analysis (Cohort A – North America, Europe, Australia)<br>(Pre-DCR Seizure Event Dataset Version 3) – mITT<br>Population | in the le |
| Table | 14.2.1.2.1.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort B – Japan) – mITT Population | Planned table per SAP. This Table number was added to the Table of Contents. |
| Table | 14.2.1.2.1.3 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis with Categorized Baseline Seizure Frequency and Baseline Seizure Frequency by Treatment Interaction (Cohort A – North America, Europe, Australia)- MITT Population | Table was described in the SAP, but shell had not been produced. This was added to the shells. |
| Table | 14.2.1.2.1.3s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis with Categorized Baseline Seizure Frequency and Baseline Seizure Frequency by Treatment Interaction (Cohort A – North America, Europe, Australia)-MITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.2.1.4 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis with Categorized Baseline Seizure Frequency and Baseline Seizure Frequency by Treatment Interaction (Cohort B – Japan)- MITT Population | Table was described in the SAP, but shell had not been produced. This was added to the shells. |
| Table | 14.2.1.2.2.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric | Table Number Update |

|---|---|---|---|
| | | Analysis (Cohort A – North America, Europe, Australia) – PP Population | insele |
| Table | 14.2.1.2.2.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.2.2.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort B – Japan) – PP Population | Planned table per SAP. This Table number was added to the Table of Contents. |
| Table | 14.2.1.3.1.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | Table Number Update |
| Table | 14.2.1.3.1.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.3.1.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort B—Japan) — mITT Population | Planned table per SAP. This Table number was added to the Table of Contents. |
| Table | 14.2.1.3.1.3 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis with Categorized Baseline Seizure Frequency and Baseline | Table was described in the SAP, but shell had not been produced. This was added to the shells. |

|---|---|---|---|
| | | Seizure Frequency by Treatment Interaction (Cohort A – North America, Europe, Australia) – mITT Population | illogic |
| Table | 14.2.1.3.1.3s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis with Categorized Baseline Seizure Frequency and Baseline Seizure Frequency by Treatment Interaction (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.3.1.4 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis with Categorized Baseline Seizure Frequency and Baseline Seizure Frequency by Treatment Interaction (Cohort B – Japan) – mITT Population | Table was described in the SAP, but shell had not been produced. This was added to the shells. |
| Table | 14.2.1.3.2.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | Table Number Update |
| Table | 14.2.1.3.2.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.4.1.1 | Percent Improvement in Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic | |

|---|---|---|---|
| | | Regression (Cohort A – North America, Europe, Australia) – mITT Population | insele |
| Table | 14.2.1.4.1.1s | Sensitivity Analysis of Percent Improvement in Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.4.1.1b | Percent Improvement in Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.4.1.1c | Percent Improvement in Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version 3 |
| Table | 14.2.1.4.1.2 | Percent Improvement in Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic Regression (Cohort B – Japan) – mITT Population | |
| Table | 14.2.1.4.2.1 | Percent Improvement in Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – PP Population | |

|---|---|---|---|
| Table | 14.2.1.4.2.1s | Sensitivity Analysis of Percent Improvement in Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – PP Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.4.2.2 | Percent Improvement in Frequency of Seizures resulting in Drops (ESC Confirmed) per 28 days during Part 1: Logistic Regression (Cohort B – Japan) – PP Population | |
| Figure | 14.2.1.5.1.1 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures Resulting in Drops (ESC Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | |
| Figure | 14.2.1.5.1.1s | Sensitivity Analysis of Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures Resulting in Drops (ESC Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | New Figure using Supplemental Seizure<br>File updated post-Part 1 Database Lock |
| Figure | 14.2.1.5.1.1b | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures Resulting in Drops (ESC Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Figure using Pre-DCR dataset Version 2 |
| Figure | 14.2.1.5.1.1c | Cumulative Response Curve for Percent of Subjects<br>Experiencing Various % Reductions in Seizures Resulting<br>in Drops (ESC Confirmed) during Part 1 (Cohort A – North | New Figure using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | | America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | |
| Figure | 14.2.1.5.1.2 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures Resulting in Drops (ESC Confirmed) during Part 1 (Cohort B - Japan) – mITT Population | S |
| Table | 14.2.1.6.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Age Subgroup: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | |
| Table | 14.2.1.6.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Age Subgroup: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.6.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Sex: Nonparametric Analysis – (Cohort A – North America, Europe, Australia) - mITT Population | |
| Table | 14.2.1.6.2s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Sex: Nonparametric Analysis – (Cohort A – North America, Europe, Australia) - mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.6.3 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Weight Subgroup: | |

|---|---|---|---|
| | | Nonparametric Analysis – (Cohort A – North America, Europe, Australia) - mITT Population | illogie |
| Table | 14.2.1.6.3s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Weight Subgroup: Nonparametric Analysis – (Cohort A – North America, Europe, Australia) - mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.6.4 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Number of Concomitant Antiepileptic Medications Used: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | |
| Table | 14.2.1.6.4s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Number of Concomitant Antiepileptic Medications Used: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.6.5 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Number of Prior Antiepileptic Medications Used: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | |
| Table | 14.2.1.6.5s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Number of Prior Antiepileptic Medications Used: | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |

|---|---|---|---|
| | | Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | insere |
| Table | 14.2.1.6.6 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Baseline Frequency of Seizures that Result in Drops: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | ns in |
| Table | 14.2.1.6.6s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Baseline Frequency of Seizures that Result in Drops: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.6.7 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Race Group: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | New Table requested. |
| Table | 14.2.1.6.8 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1 by Geographic Region: Nonparametric Analysis (Cohort A – North America, Europe, Australia) mITT Population | New Table requested. |
| Table | 14.2.1.6.9 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 Days During Part 1 by Age Group: Nonparametric Analysis (Cohort B – Japan) - mITT Population | New Table requested. |

|---|---|---|---|
| Table | 14.2.1.6.10 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 Days During Part 1 by Sex: Nonparametric Analysis (Cohort B – Japan) - mITT Population | New Table requested. |
| Table | 14.2.1.7.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 1 (Worst Value Substituted for Dropouts) (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.1.7.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 1 (Worst Value Substituted for Dropouts) (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.7.1b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 1 (Worst Value Substituted for Dropouts) (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.7.1c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 1 (Worst Value Substituted for Dropouts) (Cohort A – North America, Europe, | New Table using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | | Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | insele |
| Table | 14.2.1.7.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 1 (Worst Value Substituted for Dropouts) (Cohort B – Japan) – mITT Population | ns in |
| Table | 14.2.1.7.3 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 2 (Differential Imputation Method for Dropouts) (Cohort A – North America, Europe, Australia) – mITT Population | Correction of Table Title for Cohort A |
| Table | 14.2.1.7.3s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 2 (Differential Imputation Method for Dropouts) (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.7.3b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 2 (Differential Imputation Method for Dropouts) (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.7.3c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 2 (Differential Imputation | New Table using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | | Method for Dropouts) (Cohort A – North America,<br>Europe, Australia) (Pre-DCR Seizure Event Dataset<br>Version 3) – mITT Population | instelle |
| Table | 14.2.1.7.4 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity Analysis 2 (Differential Imputation Method for Dropouts) (Cohort B – Japan) – mITT Population | Correction of Table Title for Cohort B |
| Table | 14.2.1.8.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Wilcoxon Analysis – Sensitivity to Analysis Method (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.1.8.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Wilcoxon Analysis – Sensitivity to Analysis Method (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.8.1b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Wilcoxon Analysis – Sensitivity to Analysis Method (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.8.1c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Wilcoxon Analysis – Sensitivity to Analysis Method (Cohort A – North | New Table using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | | America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | insele |
| Table | 14.2.1.8.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Wilcoxon Analysis – Sensitivity to Analysis Method (Cohort B – Japan) – mITT Population | ns in |
| Table | 14.2.1.9.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Outliers (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.1.9.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Outliers (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.9.1b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Outliers (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.9.1c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Outliers (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version 3 |

|---|---|---|---|
| Table | 14.2.1.9.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Outliers (Cohort B – Japan) – mITT Population | ing inerec |
| Table | 14.2.1.10.1 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Seizure Clusters (Cohort A North America, Europe, Australia) – mITT Population | |
| Table | 14.2.1.10.1s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Seizure Clusters (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.10.1b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Seizure Clusters (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.10.1c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis – Sensitivity to Seizure Clusters (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version 3 |
| Table | 14.2.1.10.2 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric | |

|---|---|---|---|
| | | Analysis – Sensitivity to Seizure Clusters (Cohort B – Japan) – mITT Population | ins le |
| Table | 14.2.1.10.3 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cluster Event Sensitivity Analysis) (Cohort A – North America, Europe, Australia) – mITT Population | Sensitivity Analysis to assess the impact of imputation of number of events associated with cluster events. |
| Table | 14.2.1.10.3s | Sensitivity Analysis of Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cluster Event Sensitivity Analysis) (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.1.10.3b | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cluster Event Sensitivity Analysis) (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.1.10.3c | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cluster Event Sensitivity Analysis) (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version 3 |
| Table | 14.2.1.10.4 | Frequency of Seizures Resulting in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric | Sensitivity Analysis to assess the impact of imputation of number of events associated with cluster events. |

|---|---|---|---|
| | | Analysis (Cluster Event Sensitivity Analysis) (Cohort B – Japan) – mITT Population | ins ele |
| | 14.2.2 | Efficacy – Clinical Global Impression – Improvement rating by Investigator | S |
| Table | 14.2.2.1.1.1 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.1.2 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 (Cohort B – Japan) – mITT Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.2.1 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 (Cohort A – North America, Europe, Australia) – PP Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.3.1 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Age Subgroup (Cohort A – North America, Europe, Australia) – mITT Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.3.2 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Sex (Cohort A – North America, Europe, Australia) – mITT Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.3.3 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Weight Subgroup (Cohort A – North America, Europe, Australia) – mITT Population | Table Title adjustment to align with shell. |

|---|---|---|---|
| Table | 14.2.2.1.3.4 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Number of Concomitant Antiepileptic Medications Used (Cohort A – North America, Europe, Australia) – mITT Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.3.5 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Number of Prior Antiepileptic Medications Used (Cohort A – North America, Europe, Australia) – mITT Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.3.6 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Baseline Frequency of Seizures that Result in Drops (Cohort A – North America, Europe, Australia) – mITT Population | Table Title adjustment to align with shell. |
| Table | 14.2.2.1.3.6s | Sensitivity Analysis of Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Baseline Frequency of Seizures that Result in Drops (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.2.1.3.7 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Age Group (Cohort B – Japan) - mITT Population | New Table |
| Table | 14.2.2.1.3.8 | Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 by Sex (Cohort B – Japan) - mITT Population | New Table |

|---|---|---|---|
| Figure | 14.2.2.2.1 | Distribution of Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | Figure Title adjustment to align with shell. |
| Figure | 14.2.2.2.2 | Distribution of Clinical Global Impression – Improvement (CGI-I) Rating by Investigator in Part 1 (Cohort B – Japan) – mITT Population | Figure Title adjustment to align with shell. |
| | 14.2.3 | Countable Motor Seizures | |
| Table | 14.2.3.1.1.1 | Frequency of Countable Motor Seizures per 28 days during Part 1: Summary Statistics (Cohort A - North America, Europe, Australia) – mITT Population | |
| Table | 14.2.3.1.1.2 | Frequency of Countable Motor Seizures per 28 days during Part 1: Summary Statistics (Cohort B – Japan) – mITT Population | |
| Table | 14.2.3.1.2.1 | Frequency of Countable Motor Seizures per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – PP Population | |
| Table | 14.2.3.2.1.1 | Frequency of Countable Motor Seizures per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.3.2.1.2 | Frequency of Countable Motor Seizures per 28 days during Part 1: Nonparametric Analysis (Cohort B – Japan) – mITT Population | |

|---|---|---|---|
| Table | 14.2.3.2.2.1 | Frequency of Countable Motor Seizures per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | ing ite |
| | | | S |
| Table | 14.2.3.3.1.1 | Frequency of Countable Motor Seizures per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.3.3.1.2 | Frequency of Countable Motor Seizures per 28 days during Part 1: Parametric Analysis (Cohort B – Japan) – mITT Population | |
| Table | 14.2.3.3.2.1 | Frequency of Countable Motor Seizures per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | |
| | | 60. 70. | |
| Table | 14.2.3.4.1.1 | Percent Improvement in Frequency of Countable Motor<br>Seizures per 28 days during Part 1: Logistic Regression<br>(Cohort A – North America, Europe, Australia) – mITT<br>Population | |
| Table | 14.2.3.4.1.2 | Percent Improvement in Frequency of Countable Motor<br>Seizures per 28 days during Part 1: Logistic Regression<br>(Cohort B – Japan) – mITT Population | |
| Table | 14.2.3.4.2.1 | Percent Improvement in Frequency of Countable Motor<br>Seizures per 28 days during Part 1: Logistic Regression | |

|---|---|---|---|
| | | (Cohort A – North America, Europe, Australia) – PP<br>Population | ins is |
| Figure | 14.2.3.5.1.1 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Countable Motor Seizures during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | |
| Figure | 14.2.3.5.1.2 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Countable Motor Seizures during Part 1 (Cohort B – Japan)– mITT Population | |
| | 14.2.4.1 | Efficacy – Typical Drop Seizures | |
| Table | 14.2.4.1.1.1.1 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.1.1s | Sensitivity Analysis of Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.4.1.1.1.1b | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.4.1.1.1.1c | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort A – | New Table using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | | North America, Europe, Australia) (Pre-DCR Seizure<br>Event Dataset Version 3) – mITT Population | insere |
| Table | 14.2.4.1.1.1.2 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort B – Japan) – mITT Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.1.2.1 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – PP Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.1.2.1b | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – PP Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.4.1.1.2.1c | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – PP Population | New Table using Pre-DCR dataset Version 3 |
| Table | 14.2.4.1.2.1.1 | Frequency of Seizures that Typically Result in Drops per | Title update made at the request of Zogenix |
| 1 aute | 14.2.4.1.2.1.1 | 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | The update made at the request of Zogemx |
| Table | 14.2.4.1.2.1.1b | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Nonparametric Analysis (Cohort A – | New Table using Pre-DCR dataset Version 2 |
|---|---|---|---|
| | | North America, Europe, Australia) (Pre-DCR Seizure<br>Event Dataset Version 2) – mITT Population | inspire |
| Table | 14.2.4.1.2.1.1c | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version |
| Table | 14.2.4.1.2.1.2 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Nonparametric Analysis (Cohort B – Japan) – mITT Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.2.2.1 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.2.2.1b | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2)– PP Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.4.1.2.2.1c | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – PP Population | New Table using Pre-DCR dataset Version 3 |
| | | 63, 70 | |

|---|---|---|---|
| Table | 14.2.4.1.3.1.1 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.3.1.1b | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.4.1.3.1.1c | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version 3 |
| Table | 14.2.4.1.3.1.2 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Parametric Analysis (Cohort B – Japan) – mITT Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.3.2.1 | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.3.2.1b | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2)– PP Population | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.4.1.3.2.1c | Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Parametric Analysis (Cohort A – | New Table using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | | North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3)– PP Population | insere |
| Table | 14.2.4.1.4.1.1 | Percent Improvement in Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – mITT Population | Title update made at the request of Zogenix |
| Table | 14.2.4.1.4.1.1b | Percent Improvement in Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – mITT Population (Pre-DCR Seizure Event Dataset Version 2) | New Table using Pre-DCR dataset Version 2 |
| Table | 14.2.4.1.4.1.1c | Percent Improvement in Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – mITT Population (Pre-DCR Seizure Event Dataset Version 3) | New Table using Pre-DCR dataset Version 3 |
| Table | 14.2.4.1.4.1.2 | Percent Improvement in Frequency of Seizures that Typically Result in Drops per 28 days during Part 1: Logistic Regression (Cohort B – Japan)– mITT Population | Title update made at the request of Zogenix |
| Figure | 14.2.4.1.5.1.1 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures that Typically Result in Drops during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | Title update made at the request of Zogenix |

|---|---|---|---|
| Figure | 14.2.4.1.5.1.1b | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures that Typically Result in Drops during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population (Pre-DCR Seizure Event Dataset Version 2) | New Figure using Pre-DCR dataset Version 2 |
| Figure | 14.2.4.1.5.1.1c | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures that Typically Result in Drops during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population (Pre-DCR Seizure Event Dataset Version 3) | New Figure using Pre-DCR dataset Version 3 |
| Figure | 14.2.4.1.5.1.2 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures that Typically Result in Drops during Part 1 (Cohort B – Japan)– mITT Population | |
| Table | 14.2.4.1.6.1.1b | Change in Seizures that Typically Result per 28 days in Drops from Baseline during Part 1: Wilcoxon Analysis - Sensitivity to Analysis Method) (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) - mITT Population | New Figure using Pre-DCR dataset Version 2 |
| Table | 14.2.4.1.6.1.1c | Change in Seizures that Typically Result per 28 days in Drops from Baseline during Part 1: Wilcoxon Analysis - Sensitivity to Analysis Method) (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) - mITT Population | New Figure using Pre-DCR dataset Version 3 |

|---|---|---|---|
| | 14.2.4.2 | Efficacy – Countable Non-Motor Seizures | 100 100 |
| Table | 14.2.4.2.1.1.1 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | Sille |
| Table | 14.2.4.2.1.1.2 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Summary Statistics (Cohort B – Japan) + mITT Population | |
| Table | 14.2.4.2.1.2.1 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – PP Population | |
| Table | 14.2.4.2.2.1.1 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.4.2.2.1.2 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Nonparametric Analysis (Cohort B – Japan) – mITT Population | |
| Table | 14.2.4.2.2.1 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | |
| Table | 14.2.4.2.3.1.1 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | |

|---|---|---|---|
| Table | 14.2.4.2.3.1.2 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Parametric Analysis (Cohort B – Japan) – mITT Population | ingelen |
| Table | 14.2.4.2.3.2.1 | Frequency of Countable Non-Motor Seizures per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | 100 |
| Table | 14.2.4.2.4.1.1 | Percent Improvement in Frequency of Countable Non-<br>Motor Seizures per 28 days during Part 1: Logistic<br>Regression (Cohort A – North America, Europe,<br>Australia)– mITT Population | |
| Table | 14.2.4.2.4.1.2 | Percent Improvement in Frequency of Countable Non-<br>Motor Seizures per 28 days during Part 1: Logistic<br>Regression (Cohort B – Japan)– mITT Population | |
| Figure | 14.2.4.2.5.1.1 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Countable Non- Motor Seizures during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | |
| Figure | 14.2.4.2.5.1.2 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Countable Non- Motor Seizures during Part 1 (Cohort B – Japan)– mITT Population | |
| | 14.2.4.3 | Efficacy – All Countable Seizures (Motor + Non-Motor) | |

|---|---|---|---|
| Table | 14.2.4.3.1.1.1 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | ingie |
| Table | 14.2.4.3.1.1.2 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Summary Statistics (Cohort B – Japan) – mITT Population | |
| Table | 14.2.4.3.1.2.1 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – PP Population | |
| Table | 14.2.4.3.1.2.2 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Summary Statistics (Cohort B – Japan) – PP Population | |
| Table | 14.2.4.3.2.1.1 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.4.3.2.1.2 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Nonparametric Analysis (Cohort B – Japan) – mITT Population | |
| Table | 14.2.4.3.2.2.1 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) – PP Population | |

|---|---|---|---|
| Table | 14.2.4.3.3.1.1 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) – mITT Population | ing elec |
| Table | 14.2.4.3.3.1.2 | Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Parametric Analysis (Cohort B – Japan) – mITT Population | <b>1</b> |
| Table | 14.2.4.3.3.2.1 | Frequency of All Countable Seizures (Motor + Non-Motor)<br>per 28 days during Part 1: Parametric Analysis (Cohort A –<br>North America, Europe, Australia) – PP Population | |
| Table | 14.2.4.3.4.1.1 | Percent Improvement in Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.4.3.4.1.2 | Percent Improvement in Frequency of All Countable Seizures (Motor + Non-Motor) per 28 days during Part 1: Logistic Regression (Cohort B – Japan) | Title correction |
| Figure | 14.2.4.3.5.1.1 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in All Countable Seizures (Motor + Non-Motor) during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | Title correction |
| Figure | 14.2.4.3.5.1.2 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in All Countable Seizures (Motor + Non-Motor) during Part 1 (Cohort B – Japan)– mITT Population | Title correction |

| Table/<br>Figure/ | | | Description of Modification from Version |
|---|---|---|---|
| Listing | Number | Table Header | 2.0 SAP |
| Table | 14.2.4.4.1.1 | Change from Baseline in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) - mITT Population | Table Number Correction; This table was also updated to summarize the seizure types that were typically associated with drop seizures that were classified as ESC Confirmed Drop Seizures. |
| Table | 14.2.4.4.1.1s | Sensitivity Analysis of Change from Baseline in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) - mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock; The only sections affected by the update are the summary of seizure types that were typically associated with drop seizures that were classified as ESC Confirmed Drop Seizures. |
| Table | 14.2.4.4.1.1b | Change from Baseline in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) - mITT Population | New Table using Pre-DCR dataset Version 2. The only sections affected by the DCR update are the summary of seizure types that were typically associated with drop seizures that were classified as ESC Confirmed Drop Seizures. |
| Table | 14.2.4.4.1.1c | Change from Baseline in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) - mITT Population | New Table using Pre-DCR dataset Version 3. The only sections affected by the DCR update are the summary of seizure types that were typically associated with drop seizures that were classified as ESC Confirmed Drop Seizures. |

|---|---|---|---|
| Table | 14.2.4.4.1.2 | Change from Baseline in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort B – Japan) - mITT Population | Table Number Correction |
| Table | 14.2.4.4.2.1 | Percent Improvement in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | Table Number Correction |
| Table | 14.2.4.4.2.1s | Sensitivity Analysis of Percent Improvement in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock; The only sections affected by the update are the summary of seizure types that were typically associated with drop seizures that were classified as ESC Confirmed Drop Seizures. |
| Table | 14.2.4.4.2.1b | Percent Improvement in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) – mITT Population | New Table using Pre-DCR dataset Version 2. The only sections affected by the DCR update are the summary of seizure types that were typically associated with drop seizures that were classified as ESC Confirmed Drop Seizures. |
| Table | 14.2.4.4.2.1c | Percent Improvement in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) – mITT Population | New Table using Pre-DCR dataset Version 3. The only sections affected by the DCR update are the summary of seizure types that were typically associated with drop seizures that were classified as ESC Confirmed Drop Seizures. |

|---|---|---|---|
| Table | 14.2.4.4.2.2 | Percent Improvement in Seizure Frequency by Types during Part 1: Summary Statistics (Cohort B – Japan) – mITT Population | Table Number Correction |
| | 14.2.4.5 | All Countable Seizures that Did Not Result in Drops<br>(ESC Confirmed) | C <sup>o</sup> |
| Table | 14.2.4.5.1.1.1 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) - mITT Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.1.1.2 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort B – Japan) - mITT Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.1.2.1 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) - PP Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.2.1.1 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.2.1.2 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort B – Japan) - mITT Population | New defined analysis after initial Cohort A analysis |

|---|---|---|---|
| Table | 14.2.4.5.2.2.1 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Nonparametric Analysis (Cohort A – North America, Europe, Australia) - PP Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.3.1.1 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.3.1.2 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort B – Japan) - mITT Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.3.2.1 | Frequency of All Countable Seizures that did not Result in Drops (ESC Confirmed) per 28 days during Part 1: Parametric Analysis (Cohort A – North America, Europe, Australia) - PP Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.4.1.1 | Percent Improvement in Frequency of All Countable<br>Seizures that did not Result in Drops (ESC Confirmed) per<br>28 days during Part 1: Logistic Regression (Cohort A –<br>North America, Europe, Australia) - mITT Population | New defined analysis after initial Cohort A analysis |
| Table | 14.2.4.5.4.1.2 | Percent Improvement in Frequency of All Countable<br>Seizures that did not Result in Drops (ESC Confirmed) per<br>28 days during Part 1: Logistic Regression (Cohort B –<br>Japan) - mITT Population | New defined analysis after initial Cohort A analysis |

|---|---|---|---|
| Figure | 14.2.4.5.5.1.1 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in All Countable Seizures that did not Result in Drops (ESC Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) - mITT Population | New defined analysis after initial Cohort A analysis |
| Figure | 14.2.4.5.5.1.2 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in All Countable Seizures that did not Result in Drops (ESC Confirmed) during Part 1 (Cohort B – Japan) - mITT Population | New defined analysis after initial Cohort A analysis |
| | 14.2.4.6 | New Seizure Types | |
| Table | 14.2.4.6.1.1 | New Seizure Types During Part 1 (Cohort A – North America, Europe, Australia) - mITT Population | New Post-hoc defined analysis |
| Table | 14.2.4.6.1.2 | New Seizure Types During Part 1 (Cohort B – Japan) - mITT Population | New defined analysis |
| | 14.2.4.7 | Seizures Resulting in Drops (Caregiver Determination) | |
| Table | 14.2.4.7.1.1.1 | Frequency of Seizures Resulting in Drops (Caregiver Determination) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) – mITT Population | New Post-hoc defined endpoint |
| Table | 14.2.4.7.2.1.1 | Frequency of Seizures Resulting in Drops (Caregiver Determination) per 28 days during Part 1: Nonparametric | New Post-hoc defined endpoint |

|---|---|---|---|
| | | Analysis (Cohort A – North America, Europe, Australia) – mITT Population | insere |
| Table | 14.2.4.7.4.1.1 | Percent Improvement in Frequency of Seizures Resulting in Drops (Caregiver Determination) per 28 days during Part 1: Logistic Regression (Cohort A – North America, Europe, Australia) – mITT Population | New Post-hoc defined endpoint |
| Figure | 14.2.4.7.5.1.1 | Cumulative Response Curve for Percent of Subjects Experiencing Various % Reductions in Seizures Resulting in Drops (Caregiver Determination) during Part 1 (Cohort A – North America, Europe, Australia)– mITT Population | New Post-hoc defined endpoint |
| | 14.2.5 | Efficacy – Seizure-free Days | |
| Table | 14.2.5.1.1 | Number of Seizure Free Days per 28 Days during Part 1:<br>Nonparametric Analysis: (Cohort A – North America,<br>Europe, Australia) - mITT Population | |
| Table | 14.2.5.1.2 | Number of Countable Motor Seizure-Free Days per 28 Days during Part 1: Nonparametric Analysis (Cohort B – Japan) - mITT Population | New Table title for Cohort B |
| Table | 14.2.5.2.1 | Number of Drop Seizure Free Days per 28 Days (ESC Confirmed) during Part 1: Nonparametric Analysis: (Cohort A – North America, Europe, Australia) - mITT Population | |
| Table | 14.2.5.2.1s | Sensitivity Analysis of Number of Drop Seizure Free Days per 28 Days (ESC Confirmed) during Part 1: | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |

|---|---|---|---|
| | | Nonparametric Analysis: (Cohort A – North America, Europe, Australia) - mITT Population | The start of the s |
| Table | 14.2.5.2.2 | Number of Drop Seizure Free Days per 28 Days (ESC Confirmed) during Part 1: Nonparametric Analysis (Cohort B – Japan) - mITT Population | NS III |
| | 14.2.6 | Efficacy – Duration of the Longest Interval between Seizures Resulting in Drops | |
| Table | 14.2.6.1 | Duration of Longest Interval between Seizures Resulting in Drops (ESC Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.6.1s | Sensitivity Analysis of Duration of Longest Interval between Seizures Resulting in Drops (ESC Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |
| Table | 14.2.6.2 | Duration of Longest Interval between Seizures during<br>Titration and Maintenance Resulting in Drops (ESC<br>Confirmed) in Part 1 (Cohort B – Japan)– mITT Population | Adjusted title |
| Figure | 14.2.6.3 | Boxplot of the Duration of Longest Interval between Seizures Resulting in Drops (ESC Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | |
| Figure | 14.2.6.3s | Sensitivity Analysis of Boxplot of the Duration of Longest<br>Interval between Seizures Resulting in Drops (ESC | New Table using Supplemental Seizure File updated post-Part 1 Database Lock |

|---|---|---|---|
| | 1,444 | Confirmed) during Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | ingeled |
| Figure | 14.2.6.4 | Boxplot of the Duration of Longest Interval between Seizures during Titration and Maintenance Resulting in Drops (ESC Confirmed) during Part 1 (Cohort B – Japan) mITT Population | Adjusted title |
| | 14.2.7 | Efficacy – Clinical Global Impression – Improvement rating by Parent/Caregiver | |
| Table | 14.2.7.1.1 | Clinical Global Impression – Improvement Rating by Parent/Caregiver in Part 1 (Cohort A – North America, Europe, Australia) – mITT Population | |
| Table | 14.2.7.1.2 | Clinical Global Impression – Improvement Rating by Parent/Caregiver in Part 1 (Cohort B – Japan) – mITT Population | |
| Figure | 14.2.7.2.1 | Distribution of Clinical Global Impression – Improvement<br>Rating by Parent/Caregiver in Part 1 (Cohort A – North<br>America, Europe, Australia)– mITT Population | |
| Figure | 14.2.7.2.2 | Distribution of Clinical Global Impression – Improvement Rating by Parent/Caregiver in Part 1 (Cohort B – Japan) – mITT Population | |
| | 14.2.8 | Efficacy – Incidence of Status Epilepticus | |

|---|---|---|---|
| Table | 14.2.8.1.1 | Number of Episodes of Status Epilepticus (SE) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) - mITT Population | The le |
| Table | 14.2.8.1.2 | Number of Episodes of Status Epilepticus (SE) per 28 days during Part 1: Summary Statistics (Cohort B – Japan) - mITT Population | |
| Table | 14.2.8.1.3 | Sensitivity Analysis of Number of Episodes of Status Epilepticus (SE) per 28 days during Part 1: Summary Statistics (Cohort A – North America, Europe, Australia) - mITT Population Sensitivity Analysis of Number of Episodes of Status | New Analysis of Status Epilepticus using the diary events that were generalized tonic/clonic, secondarily generalized tonic/clonic, focal with clear observable signs, focal without clear observable signs, or absence/atypical absence. These events were further separated into those events that required 0 rescue medications, 1 rescue medication, or > 1 rescue medications associated with the seizure event. |
| Table | 14.2.8.1.4 | Sensitivity Analysis of Number of Episodes of Status<br>Epilepticus (SE) per 28 days during Part 1: Summary<br>Statistics (Cohort B – Japan) - mITT Population | New Analysis of Status Epilepticus using the diary events that were generalized tonic/clonic, secondarily generalized tonic/clonic, focal with clear observable signs, focal without clear observable signs, or absence/atypical absence. These events were further separated into those events that required 0 rescue medications, 1 rescue |

|---|---|---|---|
| | | | medication, or > 1 rescue medications associated with the seizure event. |
| Table | 14.2.8.2.1 | Number of Days where Episodes of Status Epilepticus (SE) Occurred per 28 Days during Part 1: Summary Statistics and Nonparametric Analysis (Cohort A – North America, Europe, Australia) - mITT Population | S |
| Table | 14.2.8.2.2 | Number of Days When Episodes of Status Epilepticus (SE)<br>Occurred per 28 Days during Part 1: Summary Statistics<br>and Nonparametric Analysis (Cohort B – Japan) - mITT<br>Population | Minor Table Title Update. |
| | 14.2.9 | Efficacy – Rescue Medication | |
| Table | 14.2.9.1.1 | Days with Rescue Medication Usage in Part 1:<br>Nonparametric Analysis (Cohort A – North America,<br>Europe, Australia) – mITT Population | |
| Table | 14.2.9.1.2 | Days with Rescue Medication Usage in Part 1:<br>Nonparametric Analysis (Cohort B – Japan) – mITT<br>Population | |
| Table | 14.2.9.2.1 | Number of Rescue Medications Used per Status Epilepticus<br>Episode in Part 1: Nonparametric Analysis (Cohort A –<br>North America, Europe, Australia) – mITT Population | |
| Table | 14.2.9.2.2 | Number of Rescue Medications Used per Status Epilepticus<br>Episode in Part 1: Nonparametric Analysis (Cohort B –<br>Japan) - mITT Population | |

|---|---|---|---|
| Table | 14.2.9.3.1 | Categorical Analysis of Change from Baseline in the<br>Number of Days with Rescue Medication Usage in Part 1<br>(Cohort A – North America, Europe, Australia) – mITT<br>Population | sihere |
| Table | 14.2.9.3.2 | Categorical Analysis of Change from Baseline in the Number of Days with Rescue Medication Usage in Part 1 (Cohort B – Japan) – mITT Population | |
| | 14.2.10 | Efficacy – Hospitalization and Resource Utilization for Treatment of Seizures | |
| Table | 14.2.10.1.1 | Hospitalization and Other Healthcare Resource Utilization during the Study: Summary statistics (Cohort A – North America, Europe, Australia) – mITT Population | Table Title updated. |
| Table | 14.2.10.1.2 | Hospitalization and Other Healthcare Resource Utilization during the Study: Summary Statistics (Cohort B – Japan) – mITT Population | Table Title updated. |
| | 14.2.12 | Exploratory Efficacy — Quality of Life in Childhood<br>Epilepsy Scale | |
| Table | 14.2.12.1.1 | Quality of Life in Childhood Epilepsy (QOLCE) in Part 1:<br>Summary Statistics and Nonparametric Analysis (Cohort A<br>North America, Europe, Australia) – mITT population | |
| Table | 14.2.12.1.2 | Quality of Life in Childhood Epilepsy (QOLCE) in Part 1:<br>Summary Statistics and Nonparametric Analysis (Cohort B<br>Japan) – mITT population | |

| Table/<br>Figure/ | | | Description of Modification from Version |
|---|---|---|---|
| Listing | Number | Table Header | 2.0 SAP |
| | 14.2.13 | Exploratory Efficacy – Zarit Caregiver Burden Inventory | illo de la companya della companya d |
| Table | 14.2.13.1.1 | Zarit Caregiver Burden Inventory during Part 1: Normal;<br>Borderline Abnormal; and Abnormal Categories (Cohort A – North America, Europe, Australia) – mITT population | |
| Table | 14.2.13.1.2 | Zarit Caregiver Burden Inventory during Part 1: Normal,<br>Borderline Abnormal; and Abnormal Categories (Cohort B<br>– Japan) – mITT population | |
| Table | 14.2.13.2.1 | Zarit Caregiver Burden Inventory Index Score during Part 1: Summary Descriptive Statistics (Cohort A – North America, Europe, Australia) – mITT population | Title updated; Added Burden. |
| Table | 14.2.13.2.2 | Zarit Caregiver Burden Inventory Index Score during Part 1: Summary Descriptive Statistics (Cohort B – Japan) – mITT population | Title updated; Added Burden. |
| | 14.2.14 | Exploratory Efficacy – Parent / Caregiver Ratings using HADS Scale | |
| Table | 14.2.14.1.1 | Parent/Caregiver Ratings Based on Hospital Anxiety and Depression Scale (HADS) during Part 1: Normal; Borderline Abnormal, and Abnormal Categories (Cohort A North America, Europe, Australia) – mITT population | |
| Table | 14.2.14.1.2 | Parent/Caregiver Ratings Based on Hospital Anxiety and Depression Scale (HADS) during Part 1: Normal; | |

|---|---|---|---|
| | | Borderline Abnormal, and Abnormal Categories (Cohort B – Japan)– mITT population | insele |
| Table | 14.2.14.2.1 | Parent/Caregiver Ratings Based on Hospital Anxiety and Depression Scale (HADS) during Part 1: Summary Descriptive Statistics (Cohort A – North America, Europe, Australia) -mITT population | S |
| Table | 14.2.14.2.2 | Parent/Caregiver Ratings Based on Hospital Anxiety and Depression Scale (HADS) during Part 1: Summary Descriptive Statistics (Cohort B – Japan) – mITT population | |
| | 14.3 | Safety | |
| | 14.3.1 | Summary of adverse events | |
| Table | 14.3.1.1.1 | Overview of Number of Subjects with TEAE during Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.1.2 | Overview of Number of Subjects with TEAE during Part 1 (Cohort B – Japan) – Safety Population | |
| Table | 14.3.1.2.1.1 | Treatment-Emergent Adverse Events in Part 1 by MedDRA<br>System Organ Class and Preferred Term (Cohort A – North<br>America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.2.1.2 | Treatment-Emergent Adverse Events in Part 1 by MedDRA<br>System Organ Class and Preferred Term (Cohort B –<br>Japan) – Safety Population | |

|---|---|---|---|
| Table | 14.3.1.2.2.1 | Treatment-Emergent Adverse Events in Part 1 by MedDRA System Organ Class and Preferred Term by Age Group (Cohort A – North America, Europe, Australia) – Safety Population | ille le |
| Table | 14.3.1.2.2.2 | Treatment-Emergent Adverse Events in Part 1 by MedDRA<br>System Organ Class and Preferred Term by Age Group<br>(Cohort B – Japan) – Safety Population | |
| Table | 14.3.1.2.3.1 | Treatment-Emergent Adverse Events in Part 1 by MedDRA<br>System Organ Class and Preferred Term by Sex (Cohort A<br>– North America, Europe, Australia)– Safety Population | |
| Table | 14.3.1.2.4.1 | Treatment-Emergent Adverse Events in Part 1 by MedDRA System Organ Class and Preferred Term by Usage of Most Commonly Used Anti-Epileptic Medications (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.2.4.2 | Treatment-Emergent Adverse Events in Part 1 by MedDRA<br>System Organ Class and Preferred Term by Usage of Most<br>Commonly Used Anti-Epileptic Medications (Cohort B –<br>Japan) Safety Population | |
| Table | 14.3.1.3.1.1 | TEAEs Leading to Study Discontinuation in Part 1 by MedDRA System Organ Class and Preferred Term (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.3.1.2 | Treatment-Emergent Adverse Events Leading to Study Discontinuation in Part 1 by MedDRA System Organ Class and Preferred Term (Cohort B – Japan) – Safety Population | |

|---|---|---|---|
| Table | 14.3.1.4.1.1 | Serious TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term (Cohort A – North America, Europe, Australia) – Safety Population | ingile |
| Table | 14.3.1.4.1.2 | Treatment-Emergent Serious Adverse Events in Part 1 by MedDRA System Organ Class and Preferred Term (Cohort B – Japan) – Safety Population | |
| Table | 14.3.1.5.1.1 | Treatment Related TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.5.1.2 | Treatment-Related TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term (Cohort B – Japan) Safety Population | |
| Table | 14.3.1.5.2.1 | Treatment Related TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term by Age Group (Cohort A – North America, Europe, Australia)— Safety Population | |
| Table | 14.3.1.5.2.2 | Treatment-Related TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term by Age Group (Cohort B – Japan)– Safety Population | |
| Table | 14.3.1.5.3.1 | Treatment Related TEAEs in Part 1 by MedDRA System<br>Organ Class and Preferred Term by Sex (Cohort A – North<br>America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.5.4.1 | Treatment Related TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term by Usage of Most | |

|---|---|---|---|
| | | Common Concomitant Antiepileptic Medications (Cohort A – North America, Europe, Australia) – Safety Population | illo ile |
| Table | 14.3.1.6.1.1 | TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term, and Maximum Severity (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.6.1.2 | TEAEs in Part 1 by MedDRA System Organ Class and Preferred Term, and Maximum Severity (Cohort B – Japan)– Safety Population | |
| Table | 14.3.1.7.1.1 | Treatment-Emergent Adverse Events in Part 1 occurring in ≥ 5% of Subjects by MedDRA System Organ Class and Preferred Term (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.7.1.2 | Treatment-Emergent Adverse Events in Part 1 Occurring in ≥ 10% of Subjects in Any Treatment Group by MedDRA Preferred Term (Cohort B – Japan) – Safety Population | Use 10% as the cutoff for Cohort B because the total sample size for Cohort B is smaller than Cohort A, leading the 5% cut to show almost all events. |
| Table | 14.3.1.8.1.1 | Overview of Treatment-Emergent Adverse Events of Special Interest during Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.1.8.1.2 | Overview of Treatment-Emergent Adverse Events of Special Interest during Part 1 (Cohort B – Japan) – Safety Population | |

|---|---|---|---|
| Table | 14.3.1.9.1.1 | Treatment-Emergent Adverse Events of Special Interest (AESI) by SOC and PT (Cohort A – North America, Europe, Australia) – Safety Population | in the le |
| Table | 14.3.1.9.1.2 | Treatment-Emergent Adverse Events of Special Interest (AESI) by SOC and PT (Cohort B – Japan) – Safety Population | No. |
| Table | 14.3.1.10.1.1.9 | Treatment-Emergent Adverse Events that Occurred in at Least 5% of Subjects During the Part 1 Titration + Maintenance Period by System Organ Class and Preferred Term with Number of Events and Number of Resolved Events (Cohort A – North America, Europe, Australia) - Safety Population | New Post-hoc AE Table request. Table number adjusted to align with Part 2 SAP. |
| Table | 14.3.1.10.1.1.10 | Treatment-Emergent Adverse Events that Occurred in at Least 5% of Subjects During the Part 1 Titration + Maintenance Period by System Organ Class and Preferred Term with Mean Onset and Mean Duration (Cohort A – North America, Europe, Australia) - Safety Population | New Post-hoc AE Table request. Table number adjusted to align with Part 2 SAP. |
| Table | 14.3.1.10.1.1.11 | Treatment-Emergent Adverse Events During the Part 1 Titration + Maintenance Period that Occurred in at Least 2% of Subjects in Either ZX008 Treatment Group and With Higher Percentage Than the Placebo Group by System Organ Class and Preferred Term (Cohort A – North America, Europe, Australia) - Safety Population | New Post-hoc AE Table request. Table number adjusted to align with Part 2 SAP. |

|---|---|---|---|
| Table | 14.3.1.10.1.2.9 | Treatment-Emergent Adverse Events that Occurred in at Least 10% of Subjects in Any Treatment Group During the Part 1 Titration + Maintenance Period by Preferred Term with Number of Events and Number of Resolved Events (Cohort B – Japan) -Safety Population | New AE Table request. Table number adjusted to align with Part 2 SAP. |
| Table | 14.3.1.10.1.2.10 | Treatment-Emergent Adverse Events that Occurred in at Least 10% of Subjects in Any Treatment Group During the Part 1 Titration + Maintenance Period by Preferred Term with Mean Onset and Mean Duration (Cohort B – Japan) - Safety Population | New AE Table request. Table number adjusted to align with Part 2 SAP. |
| | 14.3.2 | Listings of Deaths, Other Serious and Significant<br>Adverse Events | |
| Table | 14.3.2.1.1 | Listing of Deaths (Cohort A – North America, Europe, Australia) | |
| Table | 14.3.2.1.2 | Listing of Deaths (Cohort B – Japan) | |
| Table | 14.3.2.2.1 | Listing of SAEs (Cohort A – North America, Europe, Australia) | |
| Table | 14.3.2.2.2 | Listing of SAEs (Cohort B – Japan) | |
| Table | 14.3.2.3.1 | Listing of Discontinuations Due to AE (Cohort A – North America, Europe, Australia) | |
| Table | 14.3.2.3.2 | Listing of Discontinuations Due to AE (Cohort B – Japan) | |
| | 14.3.4 | Summary of Laboratory Data | |

|---|---|---|---|
| Table | 14.3.4.1.1.1 | Laboratory Parameters in Part 1 – Hematology: Summary Statistics (Cohort A – North America, Europe, Australia) - Safety Population | ingles |
| Table | 14.3.4.1.1.2 | Laboratory Parameters in Part 1 – Hematology: Summary Statistics (Cohort B – Japan) – Safety Population | 15 |
| Table | 14.3.4.1.2.1 | Shift Tables for Laboratory Parameters in Part 1 – Hematology (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.4.1.2.2 | Shift Tables for Laboratory Parameters in Part 1 – Hematology (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.2.1.1 | Laboratory Parameters in Part 1 – Biochemistry: Summary Statistics (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.4.2.1.2 | Laboratory Parameters in Part 1 – Biochemistry: Summary Statistics (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.2.2.1 | Shift Tables for Laboratory Parameters in Part 1 – Biochemistry (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.4.2.2.2 | Shift Tables for Laboratory Parameters in Part 1 – Biochemistry (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.3.1.1 | Laboratory Parameters in Part 1 – Urinalysis (Quantitative Parameters): Summary Statistics (Cohort A – North America, Europe, Australia) – Safety Population | |

|---|---|---|---|
| Table | 14.3.4.3.1.2 | Laboratory Parameters in Part 1 – Urinalysis (Quantitative Parameters): Summary Statistics (Cohort B – Japan) – Safety Population | illo |
| Table | 14.3.4.3.2.1 | Laboratory Parameters in Part 1 – Urinalysis (Categorical Parameters): Summary Statistics (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.4.3.2.2 | Laboratory Parameters in Part 1 – Urinalysis (Categorical Parameters): Summary Statistics (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.3.3.1 | Shift Tables for Laboratory Parameters in Part 1 – Urinalysis (Quantitative Parameters) (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.4.3.3.2 | Shift Tables for Laboratory Parameters in Part 1 – Urinalysis (Quantitative Parameters) (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.3.4.1 | Shift Tables for Laboratory Parameters in Part 1 – Urinalysis (Categorical Parameters) (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.3.4.3.4.2 | Shift Tables for Laboratory Parameters in Part 1 – Urinalysis (Categorical Parameters) (Cohort B – Japan) – Safety Population | |

|---|---|---|
| Table | 14.3.4.4.1.1 | Laboratory Parameters in Part 1 – Tests of Precocious<br>Puberty and Thyroid Function: Summary Statistics (Cohort<br>A – North America, Europe, Australia) – Safety Population |
| Table | 14.3.4.4.1.2 | Laboratory Parameters in Part 1 – Tests of Precocious<br>Puberty and Thyroid Function: Summary Statistics (Cohort<br>B – Japan) – Safety Population |
| Table | 14.3.4.4.2.1 | Shift Tables for Laboratory Parameters in Part 1 – Tests of Precocious Puberty and Thyroid Function (Cohort A – North America, Europe, Australia) – Safety Population |
| Table | 14.3.4.4.2.2 | Shift Tables for Laboratory Parameters in Part 1 – Tests of Precocious Puberty and Thyroid Function (Cohort B – Japan) – Safety Population |
| Table | 14.3.4.5.1 | Laboratory Parameters in Part 1: Epilepsy Genotype Panel (Cohort A – North America, Europe, Australia) – Safety Population |
| Table | 14.3.4.5.2 | Laboratory Parameters in Part 1 : Epilepsy Genotype Panel (Cohort B – Japan) – Safety Population |
| Table | 14.3.4.6.1.1 | Number of Subjects with Decrease in Platelets Count During Part 1 with Normal Platelet Count at Baseline (Cohort A - North America, Europe, Australia) – Safety Population |

|---|---|---|---|
| Table | 14.3.4.6.1.2 | Number of Subjects with Decrease in Platelets Count<br>During Part 1 with Normal Platelet Count at Baseline<br>(Cohort B – Japan) – Safety Population | ing ere |
| Table | 14.3.4.6.2.1 | Number of Subjects with Decrease in Platelets Count<br>During Part 1 Relative to Baseline (whether Normal or<br>Abnormal) Platelet Count (Cohort A – North America,<br>Europe, Australia) – Safety Population | |
| Table | 14.3.4.6.2.2 | Number of Subjects with Decrease in Platelets Count During Part 1 Relative to Baseline (whether Normal or Abnormal) Platelet Count (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.6.3.1 | Number of Subjects with Decrease in Platelets Count During Part 1 with Normal Platelet Count at Baseline by Valproate Use (Cohort A – North America, Europe, Australia)– Safety Population | |
| Table | 14.3.4.6.3.2 | Number of Subjects with Decrease in Platelets Count<br>During Part 1 with Normal Platelet Count at Baseline by<br>Valproate Use (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.6.4.1 | Number of Subjects with Decrease in Platelets Count<br>During Part 1 with Normal Platelet Count at Baseline by<br>Presence/Absence of Infection Event (Cohort A – North<br>America, Europe, Australia) – Safety Population | |
| Table | 14.3.4.6.4.2 | Number of Subjects with Decrease in Platelets Count<br>During Part 1 with Normal Platelet Count at Baseline by | |

|---|---|---|---|
| | | Presence/Absence of Infection Event (Cohort B – Japan) – Safety Population | ins is |
| Table | 14.3.4.7.1.1 | Number of Subjects with Normal Prolactin at Baseline who had a Prolactin Increase during Part 1 at each Visit Week (Cohort A – North America, Europe, Australia) – Safety Population | 6 |
| Table | 14.3.4.7.1.2 | Number of Subjects with Normal Prolactin at Baseline who had a Prolactin Increase during Part 1 at each Visit Week (Cohort B – Japan) – Safety Population | |
| Table | 14.3.4.7.2.1 | Number of Subjects with Normal Prolactin at Baseline who had a Prolactin Increase during Part 1 with Seizure Event within 48 hours prior to Prolactin Increase at each Visit Week (Cohort A – North America, Europe, Australia) - Safety Population | |
| Table | 14.3.4.7.2.2 | Number of Subjects with Normal Prolactin at Baseline who had a Prolactin Increase during Part 1 with Seizure Event within 48 hours prior to Prolactin Increase at each Visit Week (Cohort B – Japan) -Safety Population | |
| | 14.4.1 | Vital Signs, Weight and BMI | |
| Table | 14.4.1.1.1.1 | Vital Sign Parameters in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.4.1.1.1.2 | Vital Sign Parameters in Part 1 (Cohort B – Japan) – Safety Population | |

|---|---|---|---|
| Table | 14.4.1.2.1.1 | Body Weight and BMI in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | ing her |
| Table | 14.4.1.2.1.2 | Body Weight, Height, and BMI in Part 1 (Cohort B – Japan) – Safety Population | Minor Title Update |
| Table | 14.4.1.2.2.1 | Weight Summary (Lost/Gain >=7% or >=10%) during Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.4.1.2.2.2 | Weight Summary (Lost/Gain >=7% or >=10%) during Part 1 (Cohort B – Japan) – Safety Population | |
| Table | 14.4.1.2.2.3 | Weight Summary (Lost/Gain >=7% or >=10%) during Part<br>1 by Age Group and Treatment Group (Cohort B – Japan) –<br>Safety Population | |
| Figure | 14.4.1.3.1.1 | Spaghetti Plot of Weight by Study Day during Part 1 for Subjects who had a >= 7% Decrease from Baseline in Body Weight (Cohort A – North America, Europe, Australia) - Safety Population | |
| Figure | 14.4.1.3.1.2 | Spaghetti Plot of Weight by Study Day during Part 1 for Subjects who had a >= 7% Decrease from Baseline in Body Weight by Age Group and Treatment Group (Cohort B – Japan) - Safety Population | |
| | 14.4.4 | Tanner Staging | |
| Table | 14.4.4.1.1.1 | Tanner Staging in Part 1 by Age Group for Boys (Cohort A North America, Europe, Australia) – Safety Population | |

|---|---|---|---|
| Table | 14.4.4.1.1.2 | Tanner Staging in Part 1 by Age Group for Boys (Cohort B – Japan) – Safety Population | illosie |
| Table | 14.4.4.2.1.1 | Tanner Staging in Part 1 by Age Group for Girls (Cohort A – North America, Europe, Australia) – Safety Population | Silver |
| Table | 14.4.4.2.1.2 | Tanner Staging in Part 1 by Age Group for Girls (Cohort B – Japan) – Safety Population | |
| | 14.4.5 | Columbia-Suicide Severity Rating Scale (C-SSRS) | |
| Table | 14.4.5.1.1 | Number of Subjects with Based on the C-SSRS during Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.4.5.1.2 | Number of Subjects with Based on the C-SSRS during Part 1 (Cohort B – Japan) – Safety Population | |
| Table | 14.4.5.2.1 | Columbia Suicide Severity-Rating Scale (C-SSRS)- Shift Table of Changes in C-SSRS Categories During Part 1 (Cohort A – North America, Europe, Australia) - Safety Population | |
| Table | 14.4.5.2.2 | Columbia Suicide Severity-Rating Scale (C-SSRS)- Shift Table of Changes in C-SSRS Categories During Part 1 (Cohort B – Japan) - Safety Population | |
| | 14.4.6 | Brief Rating Inventory of Executive Function- (BRIEF) | |

|---|---|---|---|
| Table | 14.4.6.1.1 | Brief Rating Inventory of Executive Function Preschool<br>Version (BRIEF-P) in Part 1: Scoring Summary Table by<br>Treatment Group (Cohort A – North America, Europe,<br>Australia)— Safety Population | ingered |
| Table | 14.4.6.1.2 | Brief Rating Inventory of Executive Function Preschool<br>Version (BRIEF-P) in Part 1: Scoring Summary Table by<br>Treatment Group (Cohort B – Japan) – Safety Population | |
| Figure | 14.4.6.1.3 | Brief Rating Inventory of Executive Function Preschool<br>Version (BRIEF-P) in Part 1: Mean Change from Baseline<br>by Treatment Group (Cohort B – Japan) – Safety<br>Population | New Figure added for Cohort B |
| Table | 14.4.6.2.1 | Brief Rating Inventory of Executive Function (BRIEF) in Part 1: Scoring Summary Table by Treatment Group (Cohort A—North America, Europe, Australia) – Safety Population | |
| Table | 14.4.6.2.2 | Brief Rating Inventory of Executive Function (BRIEF) in Part 1: Scoring Summary Table by Treatment Group (Cohort B – Japan) – Safety Population | |
| Figure | 14.4.6.2.3 | Brief Rating Inventory of Executive Function (BRIEF) in Part 1: Mean Change from Baseline by Treatment Group (Cohort B – Japan) – Safety Population | New Figure added for Cohort B |
| Table | 14.4.6.3.1 | Brief Rating Inventory of Executive Function (BRIEF-A) in Part 1: Scoring Summary Table by Treatment Group | |

|---|---|---|---|
| | | (Cohort A – North America, Europe, Australia) – Safety<br>Population | ill sie |
| Table | 14.4.6.3.2 | Brief Rating Inventory of Executive Function (BRIEF-A) in Part 1: Scoring Summary Table by Treatment Group (Cohort B – Japan) - Safety Population | Silli |
| Figure | 14.4.6.3.3 | Brief Rating Inventory of Executive Function (BRIEF-A) in Part 1: Mean Change from Baseline by Treatment Group (Cohort B – Japan) – Safety Population | New Figure added for Cohort B |
| | 14.4.7 | Clinically Relevant Physical Examination | |
| Table | 14.4.7.1.1 | Clinically Relevant Physical Examination Findings in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.4.7.1.2 | Clinically Relevant Physical Examination Findings in Part 1 (Cohort B – Japan) - Safety Population | |
| | 14.4.8 | Clinically Relevant Neurologic Examination | |
| Table | 14.4.8.1.1 | Clinically Relevant Neurologic Examination Findings in Part 1 (Cohort A – North America, Europe, Australia) – Safety Population | |
| Table | 14.4.8.1.2 | Clinically Relevant Neurologic Examination Findings in Part 1 (Cohort B – Japan) - Safety Population | |
| | 16.2 | Subject data listing | |
| | 16.2.1 | Subject disposition and discontinuation | |

|---|---|---|---|
| Listing | 16.2.1.1.1 | Subject Completion/Discontinuation in Part 1 (Cohort A - North America, Europe, Australia) | The second |
| Listing | 16.2.1.1.2 | Subject Completion/Discontinuation in Part 1 (Cohort B-Japan) | S |
| | 16.2.2 | Protocol deviations | |
| Listing | 16.2.2.1.1 | Major Protocol Deviations in Part I (Cohort A - North<br>America, Europe, Australia) | |
| Listing | 16.2.2.1.2 | Major Protocol Deviations in Part 1 (Cohort B - Japan) | |
| | 16.2.3 | Subjects excluded from analysis | |
| Listing | 16.2.3.1.1 | Subjects Excluded from the Per Protocol Population (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.3.1.2 | Subjects Excluded from the Per Protocol Population (Cohort B - Japan) | |
| Listing | 16.2.3.2.1 | Subject Allocation to Trial Populations (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.3.2.2 | Subject Allocation to Trial Populations (Cohort B - Japan) | |
| | 16.2.4 | Demographic data and other baseline characteristics | |
| Listing | 16.2.4.1.1.1 | Demographic data (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.4.1.1.2 | Demographic data (Cohort B - Japan) | |
|---|---|---|---|
| Listing | 16.2.4.1.2.1 | Informed Consent / Informed Assent in Part 1 (Cohort A - North America, Europe, Australia) | ill voice |
| Listing | 16.2.4.1.2.2 | Informed Consent / Informed Assent in Part 1 (Cohort B Japan) | S |
| Listing | 16.2.4.1.4.1 | % Change from Baseline in Weight and BMI (Cohort A. North America, Europe, Australia) | |
| Listing | 16.2.4.1.4.2 | % Change from Baseline in Weight and BMI (Cohort B - Japan) | |
| Listing | 16.2.4.2.1.1 | Medical History and Neurologic History (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.4.2.1.2 | Medical History and Neurologic History (Cohort B - Japan) | |
| Listing | 16.2.4.2.3.1 | Seizure history (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.4.2.3.2 | Seizure history (Cohort B - Japan) | |
| Listing | 16.2.4.3.1.1 | Medications and Therapies/Treatments Stopped during or up to 30 days prior to Screening (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.4.3.1.2 | Medications and Therapies/Treatments Stopped During or Up to 30 Days Prior to Screening (Cohort B - Japan) | Title Adjustment |
| Listing | 16.2.4.3.2.1 | Concomitant Medications and Therapies/Treatments (Cohort A - North America, Europe, Australia) | |

|---|---|---|---|
| Listing | 16.2.4.3.2.2 | Concomitant Medications and Therapies/Treatments (Cohort B - Japan) | ins is |
| Listing | 16.2.4.4.1.1 | Prior Antiepileptic Drugs (AEDs)(Cohort A - North<br>America, Europe, Australia) | S |
| Listing | 16.2.4.4.1.2 | Prior Antiepileptic Drugs (AEDs)(Cohort B - Japan) | |
| Listing | 16.2.4.4.2.1 | Concomitant Antiepileptic Drugs (AEDs) (Cohort A North America, Europe, Australia) | |
| Listing | 16.2.4.4.2.2 | Concomitant Antiepileptic Drugs (AEDs) (Cohort B - Japan) | |
| Listing | 16.2.4.5.1.1 | Rescue Medications (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.4.5.1.2 | Rescue Medications (Cohort B - Japan) | |
| | 16.2.5 | Treatment exposure and compliance | |
| Listing | 16.2.5.1.1 | IMP Intake per Day during Treatment (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.5.1.2 | IMP Intake per Day during Treatment (Cohort B - Japan) | |
| Listing | 16.2.5.2.1 | IMP Intake - Self Reported % Compliance (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.5.2.2 | IMP Intake – Self Reported % Compliance (Cohort B - Japan) | |

|---|---|---|---|
| Listing | 16.2.5.3.1 | Drug Accountability (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.5.3.2 | Drug Accountability (Cohort B - Japan) | 6 |
| Listing | 16.2.5.4.1 | Background Antiepileptic Drugs (AEDs) Pharmacokinetic<br>Concentrations (Cohort A - North America, Europe,<br>Australia) | |
| Listing | 16.2.5.4.2 | Background Antiepileptic Drugs (AEDs) Pharmacokinetic<br>Concentrations (Cohort B - Japan) | |
| | 16.2.6 | Efficacy data | |
| Listing | 16.2.6.1.1.1 | Recorded Seizures – Duration and Number of Occurrences per Subject (Diary data) (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.1.1.2 | Recorded Seizures - Duration and Number of Occurrences per Subject (Diary data) (Cohort B - Japan) | |
| Listing | 16.2.6.1.2.1 | Change in Seizure Frequency Resulting in Drops (ESC Confirmed) from Baseline during Part 1 (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.1.2.1s | Sensitivity Analysis of Change in Seizure Frequency<br>Resulting in Drops (ESC Confirmed) from Baseline during<br>Part 1 (Cohort A - North America, Europe, Australia) | New Listing using Supplemental Seizure<br>File updated post-Part 1 Database Lock |

|---|---|---|---|
| Listing | 16.2.6.1.2.1c | Change in Seizure Frequency Resulting in Drops (ESC Confirmed) from Baseline during Part 1 (Cluster Sensitivity) (Cohort A - North America, Europe, Australia) | New Listing due to request for Cluster<br>Sensitivity |
| Listing | 16.2.6.1.2.1cs | Sensitivity Analysis of Change in Seizure Frequency<br>Resulting in Drops (ESC Confirmed) from Baseline during<br>Part 1 (Cluster Sensitivity) (Cohort A - North America,<br>Europe, Australia) | New Listing using Supplemental Seizure<br>File updated post-Part 1 Database Lock |
| Listing | 16.2.6.1.2.1b | Change in Seizure Frequency Resulting in Drops (ESC Confirmed) from Baseline during Part 1 (Cohort A - North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 2) | New Listing using Pre-DCR dataset Version 2 |
| Listing | 16.2.6.1.2.1c3 | Change in Seizure Frequency Resulting in Drops (ESC Confirmed) from Baseline during Part 1 (Cohort A - North America, Europe, Australia) (Pre-DCR Seizure Event Dataset Version 3) | New Listing using Pre-DCR dataset Version 3 |
| Listing | 16.2.6.1.2.2 | Change in Seizure Frequency Resulting in Drops (ESC Confirmed) from Baseline during Part 1 (Cohort B - Japan) | |
| Listing | 16.2.6.2.1.1 | Clinical Global Impression – Improvement Rating as<br>Assessed by the Investigator (Cohort A - North America,<br>Europe, Australia) | Subject – Parent/Caregiver values separated from Investigator listing. |
| Listing | 16.2.6.2.1.2 | Clinical Global Impression – Improvement Rating as<br>Assessed by the Investigator (Cohort B - Japan) | Subject – Parent/Caregiver values separated from Investigator listing. |

|---|---|---|---|
| Listing | 16.2.6.2.2.1 | Clinical Global Impression – Improvement Rating as Assessed by the Subject or Parent/Caregiver (Cohort A - North America, Europe, Australia) | Subject – Parent/Caregiver values separated from Investigator listing. |
| Listing | 16.2.6.2.2.2 | Clinical Global Impression – Improvement Rating as Assessed by the Subject or Parent/Caregiver (Cohort B - Japan) | Subject – Parent/Caregiver values separated from Investigator listing. |
| Listing | 16.2.6.3.1 | Change in Countable Motor Seizures from Baseline during Part 1 (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.3.2 | Change in Countable Motor Seizures from Baseline during Part 1 (Cohort B - Japan) | |
| Listing | 16.2.6.4.1 | Duration of Longest Interval between Seizures during Titration and Maintenance Resulting in Drops (ESC Confirmed) in Part 1 (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.4.1s | Sensitivity Analysis of Duration of Longest Interval<br>between Seizures during Titration and Maintenance<br>Resulting in Drops (ESC Confirmed) in Part 1 (Cohort A -<br>North America, Europe, Australia) | New Listing using Supplemental Seizure<br>File updated post-Part 1 Database Lock |
| Listing | 16.2.6.4.2 | Duration of Longest Interval between Seizures during<br>Titration and Maintenance Resulting in Drops (ESC<br>Confirmed) in Part 1 (Cohort B – Japan) | |

|---|---|---|---|
| Listing | 16.2.6.5.1 | Change in Seizures that Typically Result in Drops from Baseline during Part 1 (Cohort A - North America, Europe, Australia) | ingleten |
| Listing | 16.2.6.5.1b | Change in Seizures that Typically Result in Drops from<br>Baseline during Part 1 (Cohort A - North America,<br>Europe, Australia) (Pre-DCR Version 2) | |
| Listing | 16.2.6.5.1c | Change in Seizures that Typically Result in Drops from Baseline during Part 1 (Cohort A - North America, Europe, Australia) (Pre-DCR Version 3) | |
| Listing | 16.2.6.5.2 | Change in Seizures that Typically Result in Drops from Baseline during Part 1 (Cohort B - Japan) | |
| Listing | 16.2.6.6.1 | Change in Countable Non-Motor Seizures from Baseline during Part I (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.6.2 | Change in Countable Non-Motor Seizures from Baseline during Part 1 (Cohort B. Japan) | |
| Listing | 16.2.6.7.1 | Change in All Countable Seizures (Motor + Non-Motor) from Baseline during Part 1 (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.7.2 | Change in All Countable Seizures (Motor + Non-Motor) from Baseline during Part 1 (Cohort B - Japan) | |
| Listing | 16.2.6.13.1 | Change in Rescue Medication Usage from Baseline during<br>Part 1 (Cohort A - North America, Europe, Australia) | |

|---|---|---|---|
| Listing | 16.2.6.13.2 | Change in Rescue Medication Usage from Baseline during<br>Part 1 (Cohort B - Japan) | illogic |
| Listing | 16.2.6.14.1 | Seizure Free Days during Part 1 (Cohort A - North<br>America, Europe, Australia) | S |
| Listing | 16.2.6.14.2 | Countable Motor Seizure Free Days during Part 1 (Cohort B - Japan) | Modification of Title. |
| Listing | 16.2.6.14.3 | Drop Seizure Free Days (ESC Confirmed) during Part 1 (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.14.3s | Sensitivity Analysis of Drop Seizure Free Days (ESC Confirmed) during Part 1 (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.14.4 | Drop Seizure Free Days (ESC Confirmed) during Part 1 (Cohort B - Japan) | |
| Listing | 16.2.6.15.1 | Hospitalizations and Medical Services (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.6.15.2 | Hospitalizations and Medical Services (Cohort B - Japan) | |
| Listing | 16.2.6.16.1 | Vineland Adaptive Behavior Scale (VABS) (Cohort A -<br>North America, Europe, Australia) | |
| Listing | 16.2.6.16.2 | Vineland Adaptive Behavior Scale (VABS) (Cohort B - Japan) | |
| Listing | 16.2.6.17.1 | Quality of Life in Childhood Epilepsy (QOLCE) Scale<br>(Cohort A - North America, Europe, Australia) | |

|---|---|---|---|
| Listing | 16.2.6.17.2 | Quality of Life in Childhood Epilepsy (QOLCE) Scale (Cohort B - Japan) | illogie |
| Listing | 16.2.6.18.1 | Zarit Caregiver Burden Inventory (Cohort A - North<br>America, Europe, Australia) | S |
| Listing | 16.2.6.18.2 | Zarit Caregiver Burden Inventory (Cohort B - Japan) | |
| Listing | 16.2.6.19.1 | Parent/Caregiver Ratings using HADS Scale (Cohort A) North America, Europe, Australia) | |
| Listing | 16.2.6.19.2 | Parent/Caregiver Ratings Using HADS Scale (Cohort B - Japan) | Title Adjustment |
| Listing | 16.2.6.20.1 | Change in All Countable Seizures that did not Result in Drops (ESC Confirmed) from Baseline during Part 1 (Cohort A - North America, Europe, Australia) | New post-hoc defined endpoint |
| Listing | 16.2.6.20.2 | Change in All Countable Seizures that did not Result in Drops (ESC Confirmed) from Baseline during Part 1 (Cohort B - Japan) | New post-hoc defined endpoint |
| Listing | 16.2.6.21.1 | Change in Seizure Frequency Resulting in Drops<br>(Caregiver Determination) from Baseline during Part 1<br>(Cohort A - North America, Europe, Australia) | New post-hoc defined endpoint |
| | 16.2.7 | Adverse events | |
| Listing | 16.2.7.1.1 | Adverse Events (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.7.1.2 | Adverse Events (Cohort B - Japan) | |

|---|---|---|---|
| Listing | 16.2.7.2.1 | Adverse Events of Special Interest (AESI) (Cohort A - North America, Europe, Australia) | ins ie |
| Listing | 16.2.7.2.2 | Adverse Events of Special Interest (AESI) (Cohort B - Japan) | S |
| | 16.2.8 | Laboratory data | |
| Listing | 16.2.8.1.1.1 | Laboratory Data Hematology Parameters (Cohort A - North<br>America, Europe, Australia) | |
| Listing | 16.2.8.1.1.2 | Laboratory Data Hematology Parameters (Cohort B - Japan) | |
| Listing | 16.2.8.1.2.1 | Extreme Value Laboratory Parameters – Hematology (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.8.1.2.2 | Critical or Notable Value Laboratory Parameters –<br>Hematology (Cohort B - Japan) | Title Adjustment |
| Listing | 16.2.8.2.1.1 | Laboratory Data Biochemistry Parameters (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.8.2.1.2 | Laboratory Data Biochemistry Parameters (Cohort B - Japan) | |
| Listing | 16.2.8.2.2.1 | Extreme Value Laboratory Parameters – Biochemistry (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.8.2.2.2 | Critical or Notable Value Laboratory Parameters – Biochemistry (Cohort B - Japan) | Title Adjustment |

|---|---|---|---|
| Listing | 16.2.8.3.1.1 | Laboratory Data Coagulation Parameters (Cohort A - North<br>America, Europe, Australia) | insele |
| Listing | 16.2.8.3.1.2 | Laboratory Data Coagulation Parameters (Cohort B - Japan) | Sili |
| Listing | 16.2.8.4.1.1 | Laboratory Data Urinalysis Parameters (Cohort A - North<br>America, Europe, Australia) | |
| Listing | 16.2.8.4.1.2 | Laboratory Data Urinalysis Parameters (Cohort B - Japan) | |
| Listing | 16.2.8.4.2.1 | Extreme Value Urinalysis Data (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.8.4.2.2 | Critical or Notable Value Urinalysis Data (Cohort B - Japan) | Title Adjustment |
| Listing | 16.2.8.5.1 | Tests of Growth, Precocious Puberty and Thyroid Function (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.8.5.2 | Tests of Growth, Precocious Puberty and Thyroid Function (Cohort B - Japan) | |
| Listing | 16.2.8.6.1 | Urine and Serum Pregnancy tests (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.8.6.2 | Urine and Serum Pregnancy tests (Cohort B - Japan) | |
| Listing | 16.2.8.7.1 | Urine and Serum THC panel (Cohort A - North America,<br>Europe, Australia) | |
| Listing | 16.2.8.7.2 | Urine and Serum THC panel (Cohort B - Japan) | |

|---|---|---|---|
| Listing | 16.2.8.8.1 | Laboratory Data: Listing of Test Comments from Lab<br>Vendor for All Laboratory Parameters (Cohort A - North<br>America, Europe, Australia) | New Listing added. |
| Listing | 16.2.8.8.2 | Laboratory Data: Listing of Test Comments from<br>Laboratory Vendor for All Laboratory Parameters (Cohort<br>B – Japan) | New Listing added. Title Adjustment. |
| | 16.2.9 | Other Safety Data | |
| Listing | 16.2.9.1.1.1 | Vital Signs (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.9.1.1.2 | Vital Signs (Cohort B - Japan) | |
| Listing | 16.2.9.1.2.1 | Abnormal Vital Signs Data (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.9.1.2.2 | Abnormal Vital Signs Data (Cohort B - Japan) | |
| Listing | 16.2.9.2.1 | Columbia-Suicide Severity Rating Scale (C-SSRS) (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.9.2.2 | Columbia-Suicide Severity Rating Scale (C-SSRS) (Cohort B - Japan) | |
| Listing | 16.2.9.3.1.1 | Behavior Rating Inventory of Executive Function – Preschool Version (BRIEF-P) – Individual Questions (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.9.3.1.2 | Behavior Rating Inventory of Executive Function – Preschool Version (BRIEF-P) – Individual Questions (Cohort B - Japan) | |

| Table/<br>Figure/ | | | Description of Modification from Version |
|---|---|---|---|
| Listing | Number | Table Header | 2.0 SAP |
| Listing | 16.2.9.3.2.1 | Behavior Rating Inventory of Executive Function – Preschool Version (BRIEF-P) – Summary Scales and Indexes (Cohort A - North America, Europe, Australia) | in the le |
| Listing | 16.2.9.3.2.2 | Behavior Rating Inventory of Executive Function –<br>Preschool Version (BRIEF-P) – Summary Scales and<br>Indexes (Cohort B - Japan) | |
| Listing | 16.2.9.3.3.1 | Behavior Rating Inventory of Executive Function (BRIEF) – Individual Questions (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.9.3.3.2 | Behavior Rating Inventory of Executive Function (BRIEF) – Individual Questions (Cohort B - Japan) | |
| Listing | 16.2.9.3.4.1 | Behavior Rating Inventory of Executive Function (BRIEF) – Summary Scales and Indexes (Cohort A - North America, Europe, Australia) | |
| Listing | 16.2.9.3.4.2 | Behavior Rating Inventory of Executive Function (BRIEF) – Summary Scales and Indexes (Cohort B - Japan) | |
| Listing | 16.2.9.3.5.1 | Behavior Rating Inventory of Executive Function Adult<br>Version (BRIEF-A) – Individual Questions (Cohort A -<br>North America, Europe, Australia) | |
| Listing | 16.2.9.3.5.2 | Behavior Rating Inventory of Executive Function Adult<br>Version (BRIEF-A) – Individual Questions (Cohort B -<br>Japan) | |

| Table/<br>Figure/<br>Listing | Number | Description of Modification from Version 2.0 SAP |
|---|---|---|
| Listing | 16.2.9.3.6.1 | Behavior Rating Inventory of Executive Function Adult Version (BRIEF-A) – Summary Scales and Indexes (Cohort A - North America, Europe, Australia) |
| Listing | 16.2.9.3.6.2 | Behavior Rating Inventory of Executive Function Adult Version (BRIEF-A) – Summary Scales and Indexes (Cohort B - Japan) |
| Listing | 16.2.9.4.1 | Tanner Staging (Cohort A - North America, Europe, Australia) |
| Listing | 16.2.9.4.2 | Tanner Staging (Cohort B - Japan) |
| Listing | 16.2.9.5.1 | Physical Examination and Neurologic Examination (Cohort A - North America, Europe, Australia) |
| Listing | 16.2.9.5.2 | Physical Examination and Neurologic Examination (Cohort B - Japan) |
| Listing | 16.2.9.7.1 | Epilepsy Genotype panel (Cohort A - North America, Europe, Australia) |
| Listing | 16.2.9.7.2 | Epilepsy Genotype panel (Cohort B - Japan) |

### 15. REFERENCES

ICH Topic E2F: Development Safety Update Report, 2011.

Devinsky O, Patel AD, Cross JH, et al. Effect of cannabidiol on drop seizures in the Lennox-Gastaut syndrome. *N Engl J Med*. 2018;378:1888-97.

Kim KR, Lee E, Namkoong K, Lee YM, Lee JS, and Kim HD, "Caregiver's burden and quality of life in mitochondrial disease," Pediatric Neurology, vol. 42, no. 4, pp. 271-276, 2010.

Ng Y, Conry J, Drummond R, Stolle J, Weinberg M for the OV-1012 Study Investigators. Randomized, phase III study results of clobazam in Lennox-Gastaut syndrome. Neurology 2011; 77:1473-1481.

Rabbit, P. (Ed.). (1997). /react-text Methodology of frontal and executive function react-text: 2931. East Sussex, UK: Psychology Press.

Sabaz, M., Cairns, D. R., Lawson, J. A., Nheu, N., Bleasel, A. F., & Bye, A. M. (2000). Validation of a new quality of life measure for children with epilepsy. Epilepsia, 41(6), 765-774.

Sparrow, S. S., & Cicchetti, D. V. (1989). The Vineland Adaptive Behavior Scales. In C. S. Newmark (Ed.), Major psychological assessment instruments, Vol. 2, pp. 199-231). Needham Heights, MA, US: Allyn & Bacon.

Talarska, D. (2007). The usefulness of Quality of Life Childhood Epilepsy (QOLCE) questionnaire in evaluating the quality of life of children with epilepsy. Advances in Medical Sciences, 52 Suppl 1, 191-193.

Thiele EA, Marsh ED, French JA, et al. Cannabidiol in patients with seizures associated with Lennox-Gastaut syndrome (GWPCARE4): a randomised, double-blind, placebo-controlled phase 3 trial. *Lancet*. 2018;391:1085-96.

Tukey, JW (1977). Exploratory Data Analysis. Addison-Wesley.

Westphal-Guitti C, Alonso NB, Migliorini RCVP et al., "Quality of life and burden in caregivers of patients with epilepsy," The Journal of Neuroscience Nursing, vol. 39, no. 6, pp. 354-360, 2007.

#### **APPENDICES** 16.

#### 16.1. **APPENDIX 1 - SEIZURE TYPES**

| 16. APPENDICES | | | |
|---|---|---|---|
| 16.1. APPENDIX 1 - SEIZURE TYPES | | | |
| 1. All Seizures | 2. Countable<br>Motor Seizures | 3. Countable Non-<br>Motor Seizures | 4. Drop Seizures<br>(ESC confirmed or<br>Typical) |
| Generalized Tonic-Clonic | Generalized<br>Tonic-Clonic | | Generalized<br>Tonic-Clonic |
| Secondarily Generalized<br>Tonic-Clonic | Secondarily<br>Generalized<br>Tonic-Clonic | | Secondarily<br>Generalized<br>Tonic-Clonic |
| Tonic | Tonic | | Tonic |
| Atonic | Atonic | | Atonic |
| Tonic/Atonic | Tonic/Atonic Tonic/Atonic | | |
| Clonic | Tonic/Atonic Clonic Hemiclonic Focal with clear | | |
| Hemiclonic | Hemiclonic | | |
| Focal with clear observable signs | Focal with clear observable signs | UPPINS | |
| Focal without clear observable signs | 01/2/10 | Focal without clear observable signs | |
| Myoclonic | | Myoclonic | |
| Absence/atypical absence | oe use et | Absence/atypical absence | |
| Infantile Spasms | 00 00 | Infantile Spasms | |
| Epileptic Spasms | . 6 | Epileptic Spasms | |
| Other | all | Other | |

## SEIZURE CLASSIFICATION - PRIMARY ENDPOINT

The primary endpoint for Study 1601 is defined as the change from baseline in seizures that result in drops. Seizures that result in drops include those of type: atonic, tonic, tonic/atonic, and tonic clonic (ie, generalized tonic clonic, and secondarily generalized tonic clonic). The seizures that result in drops are similar to those as defined in the Epidiolex Phase 3 clinical studies GWPCARE3 and GWPCARE4, which were atonic, tonic, or tonic clonic (Devinsky 2018, Thiele 2018).

In the Statistical Analysis Plan (SAP) version 1.0 dated 5 August 2019, seizures resulting in drops were defined as those of the five types listed above and specified in the DSD as seizures that result in a fall based on a "Yes" response to Question 9 in the DSD. During study conduct a large number of data clarifications were raised for Question 9 leading to the conclusion that there was uncertainty amongst caregivers in how to properly answer the question. Based on this uncertainty, the definition of seizures that result in drops was changed to those of the five pre-specified types that have been reviewed and approved for each subject as a "drop seizure" by the Epilepsy Study Consortium (ESC). Approval is based on the seizures for each subject submitted to the ESC on the Seizure Identification Form during the Baseline Visit and logged in the eCRF on the Seizure History Form.

Thus, in version 1.1 of the SAP, drop seizures for the primary analysis will be those of the pre-specified type that have been approved for an individual subject as Drop by the ESC as indicated on the Seizure History eCRF under variable DROP\_ and captured in the DSD.

Under this definition, classifying a particular seizure in the diary as a drop seizure requires determining whether the type of seizure in question has been identified in the Seizure History eCRF as a drop seizure for that subject. This can typically be done by matching a seizure type identifier in the diary to its counterpart in the Seizure History eCRF. Specifically, each seizure type entered into the Seizure History eCRF is identified by a "Record Position" number. These seizure types are then referred to by subjects or caregivers when recording seizures into the electronic Seizure Diary where they are labeled with a "Seizure Unique ID". For most subjects, there is a direct correspondence between the Seizure Unique ID in the DSD and the Record Position number on the Seizure History eCRF. However, for some subjects the correspondence is imperfect and aligning seizure types between the diary and the Seizure History eCRF requires an examination of text fields. In order to ensure that drop seizures are properly classified. a manual reconciliation between the Record Position number and the Seizure Unique ID was performed. The reconciliation resulted in a list of ESC-approved drop seizures for each subject from which the seizures entered in the DSD would be compared against in order to identify seizures for the primary endpoint. In order to facilitate seizure selection the list generated from the reconciliation was entered into a separate database and transferred to the study database via data transfer specifications.

The procedures for the reconciliation are described in an addendum to the Data Management Plan.

## ZX1601-Part1CohortB\_SAP\_V3.0\_04FEB2022\_ CLEAN\_ZX\_Signed

Final Audit Report 2022-02-09

Created: 2022-02-09 By: Status: Signed Transaction ID:

# "ZX1601-Part1CohortB\_SAP\_V3.0\_04FEB2022\_CLEAN ned" History ned" History

- Document digitally presigned by DocuSign\, Inc. (enterprisesupport@docusign.com)

  2022-02-08 8:58:31 PM GMT- IP address:

  Document created by
- 2022-02-09 7:08:29 PM GMT- IP address:
- verified identity with Adobe Sign authentication 2022-02-09 - 7:11:19 PM GMT
- Document e-signed by Signature Date: 2022-02-09 - 7:11:19 PM GMT - Time Source: server- IP address:
- Document emailed to for signature 2022-02-09 - 7:11:21 PM GMT
- Email viewed by 2022-02-09 - 7:12:26 PM GMT- IP address
- verified identity with Adobe Sign authentication 2022-02-09 - 7:27:35 PM GMT
- Document e-signed by Signature Date: 2022-02-09 - 7:27:35 PM GMT - Time Source: server- IP address:
- Agreement completed. 2022-02-09 - 7:27:35 PM GMT

